| Study<br>Number: | ARQ-151-201 |
|---|---|
| <b>NCT #:</b> | NCT03638258 |
| Official<br>Title: | A Phase 2b 12-Week Parallel Group, Double Blind, Vehicle- Controlled Study of the Safety, Efficacy and Pharmacokinetics of ARQ-151 Cream 0.3% and ARQ-151 Cream 0.15% Administered QD in Subjects with Chronic Plaque Psoriasis |
| <b>SAP Date:</b> | 24-May-2019 |



Arcutis ARQ-151-201

Version: 1 Date: 24 MAY 2019

## STATISTICAL ANALYSIS PLAN

Protocol Number: ARQ-151-201

Study Title: A Phase 2b 12-Week Parallel Group, Double Blind,

Vehicle-Controlled Study of the Safety, Efficacy, and Pharmacokinetics of ARQ-151 Cream 0.3% and ARQ-151 Cream 0.15% Administered QD in

Subjects with Chronic Plaque Psoriasis

Development Phase of Study: Phase 2b

Sponsor: Arcutis, Inc.

2945 Townsgate Road, Suite 110 Westlake Village, CA 91361

Sponsor Contact: David Berk, MD

Vice President, Clinical Development

Statistical Analysis Plan based on

Protocol Version:

Amendment 1, 12 November 2018

Statistical Analysis Plan Date: 24MAY2019 Statistical Analysis Plan Version: Version 1



Arcutis ARQ-151-201

Version: 1 Date: 24 MAY 2019

# Authored by:

| | <br>DATE: 30MAY2019 |
|---|---|
| Associate Statistical Programmer QST Consultations, Ltd. | ** |
| Reviewed by: | |
| Director of Biostatistical Consulting QST Consultations, Ltd. | <br>DATE: SOM ay 2019 |
| Approved by: | |
| SIGNATURE: David Berk, MD Vice President, Clinical Development Arcutis, Inc. | DATE: May 29, 2019 |

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.



Arcutis ARQ-151-201 Version: 1 Date: 24 MAY 2019

# SAP Change History

Only final versions will be documented in the Change History.

| Version | Date | Summary of Changes | Author |
|---------|-----------|--------------------|--------|
| 1 | 24MAY2019 | Original document | |




# **TABLE OF CONTENTS**

| 1. | LIS | T OF A | BBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
|---|---|---|---|---|
| 2. | INT | RODU | CTION | 7 |
| 3. | | | JECTIVES | |
| <b>J.</b> | | | | |
| 4. | STU | STUDY DESIGN | | |
| | 4.1 | Overall | Study Design | |
| | | 4.1.1 | Schedule of Visits and Assessments | |
| | | 4.1.2 | Method of Assigning Subjects to Treatment Groups | |
| | | 4.1.3 | Blinding | 9 |
| <b>5.</b> | EFI | FICACY | AND SAFETY ENDPOINTS | 9 |
| | 5.1 | Efficac | y Endpoints | 9 |
| | | 5.1.1 | Primary Efficacy Endpoint | 10 |
| | | 5.1.2 | Secondary Efficacy Endpoints | 10 |
| | | 5.1.3 | Additional Efficacy Endpoints | 11 |
| | 5.2 | Safety | Endpoints | 11 |
| 6. | STA | ATISTIC | CAL AND ANALYTICAL PLANS | 12 |
| | 6.1 | Genera | l Methodology | 12 |
| | | 6.1.1 | Statistical Analysis | 12 |
| | | 6.1.2 | Baseline Definition | 12 |
| | | 6.1.3 | Visit Windowing | 13 |
| | | 6.1.4 | Adjustments for Covariates | 13 |
| | | 6.1.5 | Handling of Dropouts or Missing Data | 14 |
| | | 6.1.6 | Interim Analyses and Data Monitoring | 14 |
| | | 6.1.7 | Multicenter Studies | 14 |
| | | 6.1.8 | Multiple Comparisons/Multiplicity | 14 |
| | | 6.1.9 | Use of an Efficacy Subset of Subjects | 14 |
| | | 6.1.10 | Active-Control Studies Intended to Show Equivalence | 14 |
| | | 6.1.11 | Examination of Subgroups | 15 |
| | 6.2 | Dispos | ition of Subjects | |
| | 6.3 | Protoco | ol Deviations | 15 |
| | 6.4 | Data Se | ets Analyzed | 15 |
| | | 6.4.1 | Intent-to-Treat Population | 1 <i>6</i> |



# **Statistical Analysis Plan** Arcutis ARQ-151-201

Version: 1 Date: 24 MAY 2019

| | | 6.4.2 | Safety Po | pulation | 16 |
|---|---|---|---|---|---|
| | | 6.4.3 | Per-Proto | col Population | 16 |
| | | 6.4.4 | Pharmaco | kinetic Population | 16 |
| | 6.5 | Demog | graphic and | Other Baseline Characteristics | 16 |
| | 6.6 | Analys | sis of Effica | cy | 17 |
| | | 6.6.1 | Primary E | Efficacy Analysis | 17 |
| | | 6.6.2 | Secondary | y Efficacy Analysis | 17 |
| | | 6.6.3 | Explorato | ry Efficacy Analysis | 18 |
| | 6.7 | Safety | Evaluation | | 18 |
| | | 6.7.1 | Extent of | Exposure | 19 |
| | | 6.7.2 | Adverse E | Events | 19 |
| | | 6.7.3 | Clinical L | aboratory Evaluation | 20 |
| | | 6.7.4 | Other Obs | servations Related to Safety | 20 |
| | | | 6.7.4.1 | Electrocardiogram Measurements | 20 |
| | | | 6.7.4.2 | Vital Signs | 20 |
| | | | 6.7.4.3 | Physical Examination | 20 |
| | | | 6.7.4.4 | Medical History | 21 |
| | | | 6.7.4.5 | Local Tolerance Assessments | 21 |
| | | | 6.7.4.6 | Patient Health Questionnaire Depression Scale | 21 |
| | | | 6.7.4.7 | Columbia-Suicide Severity Rating Scale | 21 |
| | | | 6.7.4.8 | Prior and Concomitant Medications | 21 |
| | 6.8 | Other | Evaluations | | 21 |
| | | 6.8.1 | Pharmaco | kinetic Evaluation | 21 |
| 7. | DE | ΓERMI | NATION ( | OF SAMPLE SIZE | 22 |
| 8. | CH | ANGES | S IN THE P | PLANNED ANALYSES | 22 |
| 9. | REI | FEREN | <b>CES</b> | | 22 |
| 10. | IND | EX OF | 'PLANNE | D TABLES | 23 |
| 11. | IND | EX OF | ' PLANNE | D LISTINGS | 157 |



Arcutis ARQ-151-201

Version: 1 Date: 24 MAY 2019

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE(s) Adverse Event(s)
BSA Body Surface Area
CRF(s) Case Report Form(s)

C-SSRS Columbia-Suicide Severity Rating Scale

DLQI Dermatology Life Quality Index

ECG Electrocardiogram

IGA Investigator's Global Assessment

I-IGA Intertriginous IGA ITT Intent-to-Treat

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities mPASI Modified Psoriasis Area and Severity Index

N Sample Size

NRS Numerical Rating Score

PHQ-8 Patient Health Questionnaire Depression Scale

PK Pharmacokinetic
PP Per-Protocol

PSD Patient Symptoms Diary

QD Once a Day

SAE(s) Serious Adverse Event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

SD Standard Deviation

TEAE(s) Treatment-Emergent Adverse Event(s)

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

World Health Organization-Anatomical Therapeutic Chemical

WHO-ATC Classification System

WI-NRS Worst Itch Numerical Rating Scale

WPAI Work Productivity and Activity Impairment




#### 2. INTRODUCTION

Roflumilast is a phosphodiesterase 4 (PDE-4) inhibitor approved globally to reduce the risk of exacerbations in patients with severe chronic obstructive pulmonary disease (COPD) associated with chronic bronchitis. Roflumilast and its active metabolite, roflumilast N-oxide, are high affinity selective inhibitors of PDE-4 (a major cyclic-3′,5′-adenosine monophosphate (cyclic AMP)-metabolizing enzyme), whose activity leads to accumulation of intracellular cyclic AMP. There are four different subtypes of PDE-4: PDE-4a, PDE-4b, PDE-4c, and PDE-4d, each with several isoforms (splicing variants). IC50 values of both roflumilast and roflumilast N-oxide for the different PDE-4 isoforms and subtypes are mostly sub-nanomolar and single digit nanomolar (Hatzelmann 2010). The PDE-4 family of enzymes are the most prevalent phosphodiesterases in immune cells and inhibition of PDE-4 subtypes has been associated with anti-inflammatory effects in many biological systems.

Psoriasis is a chronic inflammatory skin disease characterized by raised, well-demarcated, erythematous oval plaques with adherent silvery scales. Numerous past reports have suggested a deficiency of cyclic AMP-dependent protein kinases in human psoriatic skin (Brion 1986). More recently, various cytokines produced by Th1 and Th17 cells have been shown to play a crucial role in the pathogenesis of psoriasis. It has been postulated that the anti-inflammatory effects of PDE-4 inhibitors may provide a beneficial therapeutic intervention in the treatment of chronic plaque psoriasis, and recently Otezla® (apremilast) a PDE-4 inhibitor has been approved for the oral treatment of chronic plaque psoriasis.

The past 15 years have witnessed a transformation in the systemic treatment of moderate to severe psoriasis with the advent of biological therapies. However, for patients with milder forms of disease, best treated with topical options, the therapeutic landscape really has not changed in several decades. Topical steroids come in all shapes and forms, but the lower potency steroids are not effective and the higher potency steroids are beset with issues of local skin atrophy and the potential for hypothalamic-pituitary axis suppression when applied over larger body surface areas and for prolonged periods of time. Vitamin D has been the other staple of topical psoriasis treatment but it is irritating, not suitable for use on the face or intertriginous areas, and its efficacy is rather modest. Hence, there is substantial medical need for additional topical approaches in the treatment of psoriasis. Arcutis, Inc is developing a topical formulation of roflumilast for the treatment of chronic plaque psoriasis.




#### 3. STUDY OBJECTIVES

To assess the safety, pharmacokinetics and efficacy of ARQ-151 cream 0.3% and ARQ-151 cream 0.15% vs. vehicle applied QD for 12 weeks to individuals treated with 2 to 20% (inclusive) Body Surface Area (BSA) of chronic plaque psoriasis.

#### 4. STUDY DESIGN

#### 4.1 Overall Study Design

This is a parallel group, double blind, vehicle-controlled study in which ARQ-151 cream 0.3%, ARQ-151 cream 0.15% or vehicle cream QD is applied for 84 days to subjects with between 2% to 20% (inclusive) BSA of chronic plaque psoriasis.

A total of up to approximately 300 subjects will be enrolled at approximately 30 study sites in the United States and Canada. Subjects will be adult (≥18 y/o) males or females with chronic plaque psoriasis. Subjects must have an Investigator's Global Assessment (IGA) of disease severity of at least Mild ('2') at Baseline. Subjects with an IGA of 'Mild' (2) will be limited to 20% of total enrollment. Subjects with an IGA of 'Severe' (4) will be limited to 15% of total enrollment. Subjects must have at least 2% and no more than 20% BSA of chronic plaque psoriasis. All psoriasis lesions on a subject will be treated including the face, trunk, genitals/skin folds, or limbs (excluding the scalp). The palms and soles will be treated but will not be counted towards any measurements of efficacy (IGA, BSA, Modified Psoriasis Area and Severity Index (mPASI)). For subjects with intertriginous area involvement, and with severity of the intertriginous area lesions at least 'mild' (IGA≥2) at Baseline, Intertriginous IGA (I-IGA) score will be recorded at weeks 4, 6, 8 and 12. The same IGA used for the primary endpoint (whole body) will also be used for I-IGA, but only intertriginous areas will be evaluated for I-IGA, not the rest of the body.

#### 4.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 5 of the protocol.

#### 4.1.2 Method of Assigning Subjects to Treatment Groups

Assignment of drug or vehicle will be made at a 1:1:1 ratio according to a computer-generated randomization list. Randomization will take place at Baseline after the patient has been found to be fully eligible for participation. Kits containing tubes of study medication will be assigned to each subject using an internet-based randomization system (IWRS). A subject may receive more than one kit for the treatment period.




The kits and tubes are blinded and each kit is numbered with a unique kit number.

## 4.1.3 Blinding

This is a double-blind study, therefore neither the subjects nor the Investigator, clinical team, and study sponsor will be aware of which treatment an individual has received.

If the situation requires emergency unblinding this will be done by investigator using the study IWRS system after discussion with Medical Monitor and the Sponsor's CMO.

The treatment assignments for all enrolled subjects will be unblinded only after the conclusion of the study. Specifically, the blind will be broken only after all data are verified, entered into the database, and validated; subject evaluability assessments are performed and entered into the database; and the database is locked.

#### 5. EFFICACY AND SAFETY ENDPOINTS

## 5.1 Efficacy Endpoints

mPASI is one of the measurements used for the severity of psoriasis. mPASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).






## 5.1.1 Primary Efficacy Endpoint

The primary efficacy endpoint is as follows:

Success in Investigator Global Assessment (IGA) of disease severity, defined as an IGA
of 'Clear' or 'Almost Clear' at Week 6.

### **5.1.2** Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- IGA score of 'clear' or 'almost clear' at weeks 2, 4, 8, and 12.
- Percent change from Baseline in mPASI at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Percent BSA affected at weeks 2, 4, 6, 8, and 12.
- IGA score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline at weeks 2, 4, 6, 8 and 12.
- For subjects with intertriginous area involvement, and with severity of the intertriginous lesions at least 'mild' (I-IGA≥2) at Baseline, 'I-IGA' score of 'clear' or 'almost clear' at weeks 2, 4, 6, 8 and 12.
- Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) pruritus score at weeks 2, 4, 6, 8, and 12.
- In subjects with WI-NRS pruritus score  $\geq 6$  at Baseline, a 4-point reduction in WI-NRS pruritus score at 2, 4, 6, 8, and 12 weeks as compared to Baseline.




- Change from Baseline in Modified Psoriasis Area Severity Index-75 (mPASI-75) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-90 (mPASI-90) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Total Patient Symptoms Diary (PSD) at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Itch-related Sleep Loss score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Dermatology Life Quality Index (DLQI) score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in responses to the questions of Total Patient Symptom Diary (PSD) at weeks 2, 4, 6, 8, and 12.

Change from Baseline will be calculating by subtracting the score at Baseline from the post-baseline score. Percent change from Baseline will be calculated by dividing change from Baseline by the Baseline score, multiplied by 100.

#### **5.1.3** Additional Efficacy Endpoints

The exploratory endpoints are as follows:

- Change from Baseline in Fatigue Numerical Rating Score (NRS) score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Work Productivity and Activity Impairment (WPAI) score at weeks 2, 4, 6, 8, and 12.

Change from Baseline will be calculating by subtracting the score at Baseline from the post-baseline score.

## 5.2 Safety Endpoints

Safety will be evaluated through examination of data collected during physical examinations, 12-lead Electrocardiograms (ECGs), local tolerability assessments, vital signs, counts and percentages of subjects who gain or lose >5% and >10% body weight, clinical laboratory parameters, Patient Health Questionnaire Depression Scale (PHQ-8), Columbia-Suicide Severity Rating Scale (C-SSRS) and adverse events (AEs) as outlined in the Schedule of Visits and Assessments. If deemed necessary, additional safety assessments will be performed at the discretion of the Principal Investigator.




## 6. STATISTICAL AND ANALYTICAL PLANS

## 6.1 General Methodology

All statistical processing will be performed using SAS® (Version 9.4 or later) unless otherwise stated. No interim analyses are planned. Except where noted, all statistical tests will be two-sided and will be performed at the 0.05 level of significance. No adjustment will be made for multiplicity.

Descriptive statistics will be used to provide an overview of the efficacy, safety, and pharmacokinetic results. For categorical parameters, the number and percentage of subjects in each category will be presented. The denominator for percentage will be based on the number of subjects appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include n (number of subjects), mean, standard deviation (SD), median, minimum and maximum. Appropriate inferential statistics will be used for the primary, secondary, and exploratory efficacy variables.

The primary method of handling missing efficacy data will be a mixture of linear interpolation and last observation carried forward (LOCF).

The efficacy analysis performed on the Intent-to-Treat (ITT) population is considered the primary analysis. The efficacy analysis performed on the Per-Protocol (PP) population is considered supportive analysis.

The number of subjects in each analysis set will be summarized. Reasons for study withdrawal during the blinded study will be summarized using frequencies and percentages by treatment group. Reported AEs, medical history terms and prior and concomitant procedures and therapies will be classified on the basis of Medical Dictionary for Regulatory Activities (MedDRA) terminology. Prior and concomitant medications will be classified on the basis of World Health Organization Drug Dictionary (WHO-DD) terminology.

## **6.1.1** Statistical Analysis

All analyses will be performed by QST using SAS® Version 9.4 or later. All summary tables and data listings will be prepared utilizing SAS® software.

The standard operating procedures (SOPs) of QST will be followed in the creation and quality control of all data displays and analyses.

#### **6.1.2** Baseline Definition

Baseline is defined as the last non-missing assessment prior to first dose of study drug.

TOOL.AN.10-01.01 Statistical Analysis Plan Template




## 6.1.3 Visit Windowing

Data will be summarized based on nominal visit indications with the exception of data captured at early termination and unscheduled visits. Data from early termination and unscheduled visits will be summarized based on mapped visit values. The analysis windows for early termination and unscheduled visits are presented in the following table.

**Analysis Windows for Efficacy and Safety Assessments** 

| Scheduled Visit | Target Study Day | Window (Days) |
|-----------------|------------------|---------------|
| Week 2 | 15 | 8 to 22 |
| Week 4 | 29 | 23 to 36 |
| Week 6 | 43 | 37 to 50 |
| Week 8 | 57 | 51 to 71 |
| Week 12 | 85 | 72 to 99 |
| Week 16 | 113 | 100 to 127 |

Data collected at early termination and unscheduled visits prior to study day 8 will not be analyzed, with the exception of those identified as baseline values. Data collected at visits after study day 127 will not be included in analyses.

The definition for the study day included in each study window is defined as below:

Study Day prior to Baseline Day 1 = Visit Date – Baseline Day 1 Date

Study Day on or after Baseline Day 1 = Visit Date – Baseline Day 1 Date + 1

If an assessment's mapped visit is a visit at which the subject has data from a scheduled visit present, or if no analyses are planned for the assessment at the mapped visit, the data collected at the early termination or unscheduled visit will not be included in analyses.

In the event of multiple values from unscheduled or early termination assessments within an analysis window, the value closest to the scheduled visit target study day will be used for analyses. If two values tie as closest to the time point (for example, one value is before and the other value is after the time point), then the later value will be selected.

Data collected at all visits will be included in the data listings with visit presented as reported by the site.

#### 6.1.4 Adjustments for Covariates

The Baseline score will be used as a covariate for each endpoint analyzed.

TOOL.AN.10-01.01 Statistical Analysis Plan Template




## 6.1.5 Handling of Dropouts or Missing Data

The primary method of handling missing efficacy data will be a mixture of linear interpolation and LOCF. Linear interpolation will be used for all instances where subjects have observed values for at least one assessment both preceding and following the missing assessment. If an unscheduled assessment occurs between the preceding or following scheduled assessment and the missing assessment, the unscheduled assessment will be used in the linear interpolation. The actual study day of assessment will be used for the preceding and following assessments, and planned study day will be used for the missing assessment. IGA and I-IGA values imputed with linear interpolation will be rounded to the nearest integer. If the missing assessment is not followed by at least one observed assessment, the method of LOCF will be used.

#### 6.1.6 Interim Analyses and Data Monitoring

No interim analysis or data monitoring is planned for this study.

#### **6.1.7** Multicenter Studies

The clinical study will be conducted under a common protocol for each investigational site. Every effort will be made to promote consistency in study execution at each investigational site. Sites will be pooled for analyses.

#### 6.1.8 Multiple Comparisons/Multiplicity

No adjustments for multiple comparisons or multiplicity will be made.

#### 6.1.9 Use of an Efficacy Subset of Subjects

Subjects randomized to study drug who were at least 80% compliant with the study drug, did not miss more than three consecutive doses, and who do not have major protocol deviations will form the Per Protocol (PP) Population. The major protocol deviations will be defined at the time of evaluability evaluation, the time between the database soft lock and hard lock before unblinding.

Excluding subjects who have major protocol deviations will decrease the variability in treatment response and will allow for a better determination of efficacy of ARQ-151 Cream 0.3% and ARQ-151 Cream 0.15%.

#### 6.1.10 Active-Control Studies Intended to Show Equivalence

Not applicable to this study.




## **6.1.11** Examination of Subgroups

Subset analyses will be conducted for the ITT population for the subgroups baseline IGA and baseline I-IGA. I-IGA will be dichotomized into presence or absence of I-IGA  $\geq 2$  at baseline. These analyses will contain only descriptive statistics of the primary efficacy endpoint.

#### 6.2 Disposition of Subjects

The number of subjects included in each analysis population (ITT, safety, PP, pharmacokinetic (PK)) will be summarized by treatment group. The number of subjects enrolled, completed, and discontinued (including the reasons for discontinuation) will be summarized for each treatment group.

Subjects who are excluded from an analysis population will be summarized by the primary reason for exclusion.

#### **6.3** Protocol Deviations

Protocol deviations leading to exclusion from the PP population will be tabulated. In addition to protocol deviations leading to exclusion from the PP population, the protocol deviations listed below will be presented in a data listing.

- Baseline PHQ-8 score greater than or equal to 15
- Received incorrect treatment
- Baseline mPASI less than 2
- Baseline IGA of Clear or Almost Clear
- Missed visit
- Missed IGA at attended visit
- Missed I-IGA at attended visit
- Missed safety labs at attended visit

#### 6.4 Data Sets Analyzed

Subjects will be presented/summarized based on the primary reason for exclusion. The primary reason for exclusion for each population is the first inclusion condition a subject fails to meet based on the order listed below.




## 6.4.1 Intent-to-Treat Population

All randomized subjects will be included in the ITT population and analyzed according to the treatment group they were randomized. All efficacy analyses will be presented using the ITT population.

#### 6.4.2 Safety Population

All subjects in the ITT population who have at least one post-baseline safety assessment will be included in the safety population and analyzed according to the treatment group they received. In the event a subject receives more than one treatment, they will be analyzed based on the treatment they received for the majority of the study. All safety analyses will be performed using the safety population.

### 6.4.3 Per-Protocol Population

All subjects in the safety population who were at least 80% compliant with study medication, did not miss more than 3 consecutive doses, and showed no other serious protocol violations will be included in the PP population and analyzed according to the treatment group they received. All efficacy analyses will be performed on the PP population.

#### 6.4.4 Pharmacokinetic Population

All subjects receiving the active drug with quantifiable plasma concentrations of roflumilast will be included in the PK population.

#### 6.5 Demographic and Other Baseline Characteristics

All summaries will be done on the ITT, PP, safety, and PK populations.

Sex, race, and ethnicity will be summarized by counts and percentages. Age (years) will be summarized with descriptive statistics.

Height, Weight, BSA, IGA, mPASI, WI-NRS, DLQI, Itch-Related Sleep Loss, and Total PSD will be summarized at baseline with descriptive statistics.

Medical histories will be coded using the MedDRA dictionary and presented in a by-subject listing.




## 6.6 Analysis of Efficacy

## 6.6.1 Primary Efficacy Analysis

The primary efficacy endpoint is success in IGA, defined as an IGA of 'Clear' or 'Almost Clear' at Week 6. The primary efficacy endpoint will be analyzed with a logistic regression with a factor of treatment group and the respective Baseline IGA score as a covariate. Statistical comparison between the active treatment arms and vehicle arms will be facilitated by using contrasts.

The primary efficacy analysis will be presented on both the ITT and PP populations.

## 6.6.2 Secondary Efficacy Analysis

The secondary efficacy endpoints will include:

- IGA score of 'clear' or 'almost clear' at weeks 2, 4, 8, and 12.
- Percent change from Baseline in mPASI at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Percent BSA affected at weeks 2, 4, 6, 8, and 12.
- IGA score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline at weeks 2, 4, 6, 8 and 12.
- For subjects with intertriginous area involvement, and with severity of the intertriginous lesions at least 'mild' (I-IGA≥2) at Baseline, 'I-IGA' score of 'clear' or 'almost clear' at weeks 2, 4, 6, 8 and 12.
- For subjects with intertriginous area involvement, and with severity of the intertriginous lesions at least 'mild' (I-IGA≥2) at Baseline, 'I-IGA' score of 'clear' or 'almost clear' and a 2-point improvement from Baseline at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in WI-NRS pruritus score at weeks 2, 4, 6, 8, and 12.
- In subjects with WI-NRS pruritus score ≥ 6 at baseline, a 4-point reduction in WI-NRS pruritus score at weeks 2, 4, 6, 8, and 12 as compared to Baseline.
- Change from Baseline in Modified Psoriasis Area Severity Index-75 (mPASI-75) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-90 (mPASI-90) improvement at weeks 2, 4, 6, 8, and 12.




- Change from Baseline in Modified Psoriasis Area Severity Index-100 (mPASI-100) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Total PSD at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Itch-related Sleep Loss score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in DLQI score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in responses to the questions of PSD at weeks 2, 4, 6, 8, and 12

Change from Baseline will be calculated by subtracting the score at Baseline from the post-baseline score. Percent change from Baseline will be calculated by dividing change from Baseline by the Baseline score, multiplied by 100.

The IGA, I-IGA, WI-NRS, and mPASI dichotomous endpoints will be analyzed with a logistic regression with a factor of treatment group and the respective Baseline score as a covariate. The remainder of the endpoints will be considered continuous and analyzed with an analysis of covariance with a factor of treatment group and the respective Baseline score as a covariate. Statistical comparisons between the active treatment arms and vehicle arm will be facilitated by using contrasts.

The secondary efficacy analysis will be presented on both the ITT and PP populations.

#### **6.6.3** Exploratory Efficacy Analysis

There are two exploratory endpoints:

- Change from Baseline in Fatigue NRS score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in WPAI score at weeks 2, 4, 6, 8, and 12.

Only descriptive statistics will be used to analyze these endpoints. Change from Baseline will be calculating by subtracting the score at Baseline from the post-baseline score.

## 6.7 Safety Evaluation

The following analyses will be performed; however, no formal inferential statistics will be done on safety assessments.

Descriptive statistics will be presented by visit and treatment group for quantitative safety data and frequency counts will be compiled for classification of qualitative safety data. Summaries of local tolerability will be presented by visit and treatment group.




## **6.7.1** Extent of Exposure

The extent of exposure to study drug in each treatment group will be summarized by total number of days of exposure, total number of applications, total amount of study drug used, number of missed applications, and number and percentage of subjects who are compliant. A subject will be considered compliant with the dosing regimen if the subject applied at least 80% of the expected number of applications while enrolled in the study and does not miss more than 3 consecutive doses.

Days of exposure = Date of last study application - Date of first study application + 1.

The total number of applications is as follows:

(Date of Last Application – Date of First Application + 1) – (Number of Days marked as missed dose on the Case Report Form (CRF)).

The expected number of applications is as follows:

Expected Date of Last Application – Date of Randomization + 1

Where the Expected Date of Last Application is the date of the Week 12 visit or the date of the discontinuation visit for subjects who discontinue prior to Week 12.

Compliance will be calculated as a percentage as 100 times the total number of applications divided by the expected number of applications.

#### 6.7.2 Adverse Events

All treatment-emergent AEs (TEAEs) occurring during the study will be recorded and classified on the basis of MedDRA terminology for the safety population. TEAEs are those AEs with an onset on or after the date of first study drug treatment. All AEs with incomplete onset date information will be considered treatment-emergent unless the available information indicates that this is not possible. All TEAEs will be summarized by treatment group, the number of subjects reporting TEAEs, system organ class, preferred term, severity, relationship, and seriousness. Each subject will be counted only once within a system organ class or a preferred term using the event with the greatest relationship and greatest severity.

Comparisons between treatment groups will be made by tabulating the frequency of subjects with one or more TEAEs (classified into MedDRA terms) during the study.

Serious AEs (SAEs) will be listed by subject. Treatment-emergent SAEs will be summarized by treatment group, severity, and relationship to study treatment.




All information pertaining to AEs noted during the study will be listed by subject, detailing the verbatim description given by the Investigator, preferred term, system organ class, start date, stop date, severity, action taken regarding study drug, corrective treatment, outcome, and drug relatedness. The event onset will also be shown relative (in number of days) to date of first application. In addition a listing of subjects who prematurely discontinue from the study due to AEs will also be provided.

## 6.7.3 Clinical Laboratory Evaluation

Laboratory test results will be summarized by treatment group and visit as observed values and changes from Baseline using descriptive statistics. Additionally, shifts from Baseline to Week 4 and Week 12 in laboratory test results based on normal ranges will be summarized with frequency counts and percentages.

Individual laboratory test results, as well as abnormal laboratory results, will be presented in a by-subject listing.

## 6.7.4 Other Observations Related to Safety

## **6.7.4.1** Electrocardiogram Measurements

Descriptive statistics of actual values and changes from baseline will be provided by treatment group and visit for the following ECG parameters: heart rate (HR), RR duration, QRS duration, PR duration, QT duration, QTc Interval, QTcB interval, QTcF interval. Investigator and cardiologist interpretation of the ECG will be summarized by counts and percentages.

Individual ECG parameters, as well as interpretations, will be presented in a by-subject listing.

#### 6.7.4.2 Vital Signs

Descriptive statistics of actual values and changes from baseline will be provided by treatment group and visit for the following parameters: temperature, systolic blood pressure, diastolic blood pressure, heart rate, and weight. Additionally, counts and percentages of subjects who gain or lose > 5% body weight will be summarized by visit in a table.

#### 6.7.4.3 Physical Examination

Abnormal physical examination findings will recorded as AEs and included in the AE summaries.




## 6.7.4.4 Medical History

Medical history for all subjects will be presented in a by-subject listing.

#### 6.7.4.5 Local Tolerance Assessments

For the investigator's assessment and subject local tolerability assessment of sensation following drug application, the numeric application site reaction scores will be summarized individually by using number and percentage of subjects by visit. In addition, a by-subject listing of investigator and subject assessments will be provided.

#### 6.7.4.6 Patient Health Questionnaire Depression Scale

The PHQ-8 will be analyzed by a shift in state of severity using the following scoring system:

- None Minimal depression (0 to 4)
- Mild depression (5 to 9)
- Moderate depression (10 to 14)
- Moderately severe depression (15 to 19)
- Severe depression (20 to 24)

In addition, a by-subject listing of results will be provided.

#### 6.7.4.7 Columbia-Suicide Severity Rating Scale

The C-SSRS will be analyzed per the C-SSRS Scoring and Data Analysis Guide (Nilsson 2013).

#### 6.7.4.8 Prior and Concomitant Medications

Prior and concomitant medication information for all randomized subjects will be presented in a by-subject listing. Summary tables will be presented by World Health Organization-Anatomical Therapeutic Chemical Classification System (WHO-ATC) therapeutic category and product.

#### 6.8 Other Evaluations

#### **6.8.1** Pharmacokinetic Evaluation

Plasma drug concentrations at pre-dose will be summarized using descriptive statistics, reporting n, mean, standard deviation, median, minimum, and maximum.




#### 7. DETERMINATION OF SAMPLE SIZE

The sample size was not powered based on data for the primary endpoint to provide statistical significance because of the absence of previous primary endpoint data. However, based on efficacy data from the Phase 1/2a study, this Phase 2b study is expected to provide reliable information regarding the efficacy and safety of the drug products.

#### 8. CHANGES IN THE PLANNED ANALYSES

The Per-Protocol population was updated to exclude subjects with more than three consecutive missed doses in order to fully capture compliant subjects.

A covariate of the respective Baseline score was added to the models used for analysis of the primary and secondary endpoints.

A secondary efficacy analysis endpoint of 'clear' or 'almost clear' plus a 2-point improvement from Baseline for Intertriginous Investigator Global Assessment (I-IGA) at weeks 2, 4, 6, 8, and 12 was added.

A secondary efficacy analysis endpoint for change from Baseline in Modified Psoriasis Area Severity Index-100 (mPASI-100) at weeks 2, 4, 6, 8, and 12 was added.

Week 2 was added to all secondary and exploratory efficacy endpoints.

#### 9. REFERENCES

Brion DE, Raynaud F, Plet A, Laurent P, Leduc B, and Anderson W. Deficiency of cyclic AMP-dependent protein kinases in human psoriasis. Proc. Natl. Acad. Sci. 1986; 83:5272-5276.

Hatzelmann A, Morcillo EJ, Lungarella G, Adnot S, Sanjar S, Beume R, et al. The preclinical pharmacology of roflumilast – a selective, oral phosphodiesterase 4 inhibitor in development for chronic obstructive pulmonary disease. Pulm Pharmacol Ther. 2010; 23:235–256.

Nilsson M, Suryawanshi S, Gassmann-Mayer C, Dubrava S, McSorley P, and Jiang K. Columbia–Suicide Severity Rating Scale Scoring and Data Analysis Guide. Version 2. 2013



Version: 1

Date: 24 MAY 2019

## 10. INDEX OF PLANNED TABLES

| Table 14.0.1: Summary of Subject Enrollment and Evaluability 29 | 9 |
|---|---|
| Table 14.0.2: Summary of Subject Completion/Discontinuation (Randomized Subjects)30 | 0 |
| Table 14.1.1.1: Summary of Subject Demographics (Intent-to-Treat Population)3 | 1 |
| Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population)3 | 1 |
| Table 14.1.1.3: Summary of Subject Demographics (Safety Population) 3 | 1 |
| Table 14.1.1.4: Summary of Subject Demographics (PK Population) | 1 |
| Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population)32 | 2 |
| Table 14.1.2.2: Summary of Subject Baseline Characteristics (Per-Protocol Population)34 | 4 |
| Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population)34 | 4 |
| Table 14.1.2.4: Summary of Subject Baseline Characteristics (PK Population)34 | 4 |
| Table 14.1.3: Summary of Medical History by MedDRA System Organ Class and Preferred Term (Safety Population) | 5 |
| Table 14.1.4.1: Summary of Prior Medications by WHO-DD ATC Level 2 Term and Preferred Name (Safety Population) | 6 |
| Table 14.1.4.2: Summary of Concomitant Medications by WHO-DD ATC Level 2 Term and Preferred Name (Safety Population) | 7 |
| Table 14.2.1.1: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Intent-to-Treat Population) | 8 |
| Table 14.2.1.2: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Per-Protocol Population) | 8 |
| Figure 14.2.1.1: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Intent-to-Treat Population) | 9 |
| Figure 14.2.1.2: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Per-Protocol Population) | 9 |
| Table 14.2.2.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population)4 | _ |
| Table 14.2.2.2: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Per-Protocol Population) | • |
| Table 14.2.3.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline (Intent-to- | |
| Treat Population)4 | 1 |



Version: 1 Date: 24 MAY 2019

| Table 14.2.3.2: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline (Per- Protocol Population) |
|---|
| Figure 14.2.3.1: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline by Visit (Intent-to-Treat Population) |
| Figure 14.2.3.2: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline by Visit (Per-Protocol Population) |
| Table 14.2.3.3: Summary of Proportion of Subjects Achieving an Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline by Investigational Site (Intent-to-Treat Population) |
| Table 14.2.4.1.1: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
| Table 14.2.4.1.2: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
| Figure 14.2.4.1.1: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
| Figure 14.2.4.1.2: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
| Table 14.2.4.2.1: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
| Table 14.2.4.2.2: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
| Figure 14.2.4.2.1: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
| Figure 14.2.4.2.2: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a |



Arcutis ARQ-151-201 Version: 1

Date: 24 MAY 2019

| 2 Grade Improvement from Baseline (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
|---|
| Table 14.2.5.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Intent-to-Treat Population) |
| Table 14.2.5.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Per-Protocol Population) |
| Figure 14.2.5.1: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Intent-to-Treat Population) |
| Table 14.2.6.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.6.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.6.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.6.2 Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population) |
| Table 14.2.7.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.7.2: Dichotomized Percent Reduction(s) in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population) |
| Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population) |
| Table 14.2.8.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Per-Protocol Population) |
| Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population) |
| Table 14.2.9.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Per-Protocol Population) |
| Table 14.2.10.1.1: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Intent-to-Treat Population: Subjects with WI-NRS Score ≥ 6 at Baseline) |




Date: 24 MAY 2019

| Table 14.2.10.1.2: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score ≥ 6 at Baseline) |
|---|
| Table 14.2.10.2.1: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score $\geq 6$ at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Intent-to-Treat Population: Subjects with WI-NRS Score $\geq 6$ at Baseline) |
| Table 14.2.10.2.2: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score $\geq 6$ at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score $\geq 6$ at Baseline) |
| Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.11.2: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Per-Protocol Population) |
| Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)85 |
| Table 14.2.12.2: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Per-Protocol Population)90 |
| Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population) |
| Table 14.2.13.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Per-Protocol Population) |
| Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)96 |
| Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)97 |
| Table 14.2.14.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Per-Protocol Population)100 |
| Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population) |
| Table 14.2.15.2: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Per-Protocol Population) |
| Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population) |
| Table 14.2.16.2: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Per-Protocol Population) |




Date: 24 MAY 2019

| Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA) (Intent-to-Treat Population) |
|---|
| Table 14.2.17.2: Summary of Whole Body Investigator Global Assessment (IGA) (Per-Protocol Population) |
| Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA) (Intent-to-Treat Population) |
| Table 14.2.18.2: Summary of Intertriginous Area Investigator Global Assessment (I-IGA) (Per-Protocol Population) |
| Table 14.3.0.1.1: Summary of Extent of Exposure (Safety Population) |
| Table 14.3.0.2.1: Summary of Pre-Dose Pharmacokinetic Concentrations (PK Population)122 |
| Table 14.3.0.2.2: Summary of Additional Pharmacokinetic Concentrations (PK Population)124 |
| Table 14.3.1.1: Summary of Local Tolerability (Safety Population) |
| Figure 14.3.1.1: Subject Local Tolerability Sensation Following Drug Application (Safety Population) |
| Table 14.3.1.2.1: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Injurious Behavior without Suicidal Intent Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population) |
| Table 14.3.1.2.2: Number of Patients with Suicide-Related Treatment-Emergent Events Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population) 131 |
| Table 14.3.1.3.1: Summary of PHQ-8 Assessments by Treatment Group (Safety Population)132 |
| Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population) |
| Table 14.3.1.4.1: Overall Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) |
| Table 14.3.1.4.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.4.3: Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug by MedDRA System Organ Class and Preferred Term (Safety Population)138 |
| Table 14.3.1.4.4: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population) |
| Table 14.3.1.4.5: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.4.6: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) |



Version: 1 Date: 24 MAY 2019

| Date: 24 MAY 2019 |
|---|
| Table 14.3.1.4.7: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.4.8: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population). 143 |
| Table 14.3.1.4.9: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results (Safety Population)145 |
| Table 14.3.1.5.1.2: Summary of Hematology Laboratory Results (Safety Population)146 |
| Table 14.3.1.5.1.3: Summary of Quantitative Urinalysis Laboratory Results (Safety Population)146 |
| Table 14.3.1.5.2.1: Shift Summary of Chemistry Laboratory Results (Safety Population)147 |
| Table 14.3.1.5.2.2: Shift Summary of Hematology Laboratory Results (Safety Population)147 |
| Table 14.3.1.5.2.3: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population) |
| Table 14.3.1.6.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population)148 |
| Table 14.3.1.6.2: Shift Summary of Overall Electrocardiogram (ECG) Assessments (Safety Population) |
| Table 14.3.1.7.1: Summary of Vital Signs (Safety Population) |
| Table 14.3.1.7.2: Summary of Change in Body Weight Compared to Baseline (Safety Population) |



Table 14.0.1: Summary of Subject Enrollment and Evaluability

| | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| Number of Subjects in the ITT Population | XX | XX | XX |
| Number of Subjects Included from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded in the Safety Population<br>Reason for Exclusion from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Post-Baseline Safety Assessment | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included from the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded in the PP Population<br>Reason for Exclusion from the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Less than 80% Compliant | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missed 3 or More Consecutive Doses | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other Serious Protocol Violations | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included from the PK Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded in the PK Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Evidence of Dosing with Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Insufficient Plasma Concentrations | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: ITT population includes all randomized subjects.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.0.2: Summary of Subject Completion/Discontinuation (Randomized Subjects)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Completed Study | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation | | | |
| Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Lost to Follow-Up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pregnancy | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Protocol Deviation | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Withdrawal by Subject | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Study Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Physician Decision | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Lack of Efficacy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.1.1.1: Summary of Subject Demographics (Intent-to-Treat Population)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Age (years) | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| N | XX | XX | XX |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Female | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Ethnicity | | | |
| N | XX | XX | XX |
| Hispanic or Latino | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Race | | | |
| N | XX | XX | XX |
| American Indian or Alaska Native | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Black or African American | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| White | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Multiple/Other | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.1.1.1 for the following:

Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population)

Table 14.1.1.3: Summary of Subject Demographics (Safety Population)

Table 14.1.1.4: Summary of Subject Demographics (PK Population)

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| TT 1 D 1 I | (N=xx) | (N=xx) | (N=xx) |
| Whole Body Investigator Global Assessment Score | | | |
| N | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Intertriginous Area Investigator Global Assessment Score <sup>a</sup> | | | |
| N | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Itch-Related Sleep Loss Score | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>a</sup> Collected for subjects with intertriginous involvement.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Body Surface Area (%) Affected by Psoriasis | (1V-AA) | (11-AA) | (11-AA) |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| mPASI | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| WI-NRS Score | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Total Psoriasis Symptom Diary (PSD) Score | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>a</sup> Collected for subjects with intertriginous involvement.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Dermatology Life Quality Index (DLQI) Score | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Height (cm) | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Weight (kg) | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

#### Repeat Table 14.1.2.1 for the following:

Table 14.1.2.2: Summary of Subject Baseline Characteristics (Per-Protocol Population)

Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population)

Table 14.1.2.4: Summary of Subject Baseline Characteristics (PK Population)



Table 14.1.3: Summary of Medical History by MedDRA System Organ Class and Preferred Term (Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | ARQ-151 Cream 0.3% (N=xxx) | ARQ-151 Cream 0.15%<br>(N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more medical histories that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)


Table 14.1.4.1: Summary of Prior Medications by WHO-DD ATC Level 2 Term and Preferred Name (Safety Population)

| ATC Level 2 Term <sup>a</sup> Preferred Name | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |

Note: Table includes all medications used prior to date of first dose of study drug.

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more prior medications that map to the WHO-DD (Version March 1, 2018). At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once.



Table 14.1.4.2: Summary of Concomitant Medications by WHO-DD ATC Level 2 Term and Preferred Name (Safety Population)

| ATC Level 2 Term <sup>a</sup> Preferred Name | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Table includes all medications used on or after date of first dose of study drug.

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more concomitant medications that map to the WHO-DD (Version March 1, 2018). At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once.



Table 14.2.1.1: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Intent-to-Treat Population)

| IGA Score of Clear or Almost Clear at Week 6 | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline IGA score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.1.1 for the following:

Table 14.2.1.2: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Per-Protocol Population)



Figure 14.2.1.1: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Intent-to-Treat Population)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

Repeat Figure 14.2.1.1 for the following:

Figure 14.2.1.2: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Per-Protocol Population)



Table 14.2.2.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population)

| GA Score of Clear or Almost Clear<br>Week 2 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 8 | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | $XX.X^{0}/_{0}$ | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 12 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline IGA score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## Repeat Table 14.2.2.1 for the following:

Table 14.2.2.2: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Per-Protocol Population)



Table 14.2.3.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA)
Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline
(Intent-to-Treat Population)

| IGA Score of Clear or Almost Clear<br>Plus a 2-Grade Improvement from Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 2 | (N-xx) | (IN-XX) | (IN-XX) |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | MMM/0 |
| Week 4 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 6 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 8 | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 12 | | | |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline IGA score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

 $SOURCE: USERNAME \verb|\SPONSOR| PROJECT \verb|\JOBNAME| (DATE, TIME)$ 

Repeat Table 14.2.3.1 for the following:

Table 14.2.3.2: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline (Per-Protocol Population)



Figure 14.2.3.1: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline by Visit (Intent-to-Treat Population)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Figure 14.2.3.1 for the following:

Figure 14.2.3.2: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline by Visit (Per-Protocol Population)



Table 14.2.3.3: Summary of Proportion of Subjects Achieving an Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear'
Plus a 2-Grade Improvement from Baseline by Investigational Site
(Intent-to-Treat Population)

| Investigational Site | ARQ-151 Cream 0.3% (N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxx | xx/xx ( xx.x%) | xx/xx ( xx.x%) | xx/xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxx | $xx/xx$ ( $xx.x^{0}$ %) | xx/xx (xx.x%) | xx/xx ( $xx.x%$ ) |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx/xx ( $xx.x%$ ) | xx/xx (xx.x%) | xx/xx ( $xx.x%$ ) |
| xxxxxxxxxxxxxxxxxxxxxx | $xx/xx$ ( $xx.x^{0}$ %) | xx/xx (xx.x%) | xx/xx ( $xx.x%$ ) |
| xxxxxxxxxxxxxxxxxxxxxx | xx/xx ( $xx.x%$ ) | xx/xx ( xx.x%) | xx/xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxx | xx/xx ( xx.x%) | xx/xx ( $xx.x%$ ) | xx/xx ( $xx.x%$ ) |

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.4.1.1: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)

| I-IGA Score of Clear or Almost Clear Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2 | (IV IIII) | (IV III) | (III) |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| Success | XX.X% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 6 | | | |
| Success | XX.X% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| Success | XX.X% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | XX.X% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 12 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline I-IGA score.

Restricted to subjects with an I-IGA severity score of at least "Mild" at baseline.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.



Repeat Table 14.2.4.1.1 for the following:

Table 14.2.4.1.2: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Figure 14.2.4.1.1: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear'

(Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Figure 14.2.4.1.1 for the following:

Figure 14.2.4.1.2: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Table 14.2.4.2.1: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)

| I-IGA Score of Clear or Almost Clear Plus a 2 Grade<br>Improvement from Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 2 | (2 \ 122) | (1 · 1112) | (1, 1111) |
| Success | xx.x% | $XX.X^{0}/_{0}$ | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 6 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 12 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | $XX.X^{0}/_{0}$ | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline I-IGA score.

Restricted to subjects with an I-IGA severity score of at least "Mild" at baseline.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.



Repeat Table 14.2.4.2.1 for the following:

Table 14.2.4.2.2: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Figure 14.2.4.2.1: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Figure 14.2.4.2.1 for the following:

Figure 14.2.4.2.2: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Table 14.2.5.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| ASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | , , |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 16 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.5.1 for the following:

Table 14.2.5.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Per-Protocol Population)



Figure 14.2.5.1: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Intent-to-Treat Population)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.6.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline
(Intent-to-Treat Population)


| Reduction in mPASI Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 2 | (IV MI) | (IV III) | (1) III) |
| 75% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 90% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 100% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| 75% Reduction | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| 100% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline mPASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.6.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| Reduction in mPASI Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | | (IV III) | (III) |
| 75% Reduction | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 90% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 100% Reduction | | | |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| 75% Reduction | | | |
| Success | xx.x% | xx.x% | XX.X <sup>0</sup> /0 |
| Failure | $XX.X^{0}\!\!/_{\!0}$ | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | $XX.X^{0}\!\!/_{\!0}$ | XX.X% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 100% Reduction | | | |
| Success | $XX.X^{0}\!\!/_{\!0}$ | XX.X% | xx.x% |
| Failure | $XX.X^{0}\!\!/_{\!0}$ | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline mPASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.6.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| Reduction in mPASI Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Veek 12 | · · · · · · | | |
| 75% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 100% Reduction | | | |
| Success | xx.x% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline mPASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## Repeat Table 14.2.6.1 for the following:

Table 14.2.6.2 Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population)



Table 14.2.7.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2 | | | |
| 75% Reduction in mPASI Compared to Baseline | ( 0() | ( 0() | ( 0() |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | , | , | , |
| Week 4 | | | |
| 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1000/P 1 di PAGE | | | |
| 100% Reduction in mPASI Compared to Baseline | ( 0/) | ( 0/) | 0/) |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.7.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | | | |
| 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | $xx(x_0^{1/2})$ | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | | |
| 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.7.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| W. 1.10 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 12 | | | |
| 75% Reduction in mPASI Compared to Baseline Success | vv ( vv v0/) | vv ( vv v0/) | vv ( vv v0/) |
| Failure | xx ( xx.x%) | XX ( XX.X%) | XX ( XX.X%) |
| ranure | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | , | , | , |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 16 | | | |
| 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 000/ P. 1 | | | |
| 90% Reduction in mPASI Compared to Baseline | ( 0() | ( 0/) | ( 0() |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ranuic | AA ( AA.A /0) | AA ( AA.A /0) | AA ( AA.A/0) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.7.1 for the following:

Table 14.2.7.2: Dichotomized Percent Reduction(s) in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population)



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| N | XX | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data at Week 16 was not imputed.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| BSA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | xx.x | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | xx.xx |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | xx.x | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | xx.x | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data at Week 16 was not imputed.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data at Week 16 was not imputed.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data at Week 16 was not imputed.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| BSA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 16 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.8.1 for the following:

Table 14.2.8.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Per-Protocol Population)



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| /I-NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)


Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| -NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| I-NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup>P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| I-NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup>P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| I-NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup>P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.9.1 for the following:

Table 14.2.9.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Per-Protocol Population)



Table 14.2.10.1.1: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline

(Intent-to-Treat Population: Subjects with WI-NRS Score ≥ 6 at Baseline)

| 4 Point Reduction in WI-NRS Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2 | (IN-XX) | (IN-XX) | (IN-XX) |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 6 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 12 | | | |
| Success | xx.x% | xx.x% | XX.X% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score.

Restricted to subjects with a baseline WI-NRS Score of 6 or greater.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.



Repeat Table 14.2.10.1.1 for the following:

Table 14.2.10.1.2: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score ≥ 6 at Baseline)



Table 14.2.10.2.1: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline

(Intent-to-Treat Population: Subjects with WI-NRS Score ≥ 6 at Baseline)

| 4 Point Reduction in WI-NRS Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | $xx(x_0^{1/2})$ | XX (XX.X%) | xx ( xx.x%) |
| Week 6 | | | |
| Success | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| Week 8 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| Week 12 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

Restricted to subjects with a baseline WI-NRS Score of 6 or greater.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## Repeat Table 14.2.10.2.1 for the following:

Table 14.2.10.2.2: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score  $\geq 6$  at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score  $\geq 6$  at Baseline)



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| otal PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| al PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| al PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| otal PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| al PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | xx.xx |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| otal PSD Score<br>Week 16 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.11.1 for the following:

Table 14.2.11.2: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Per-Protocol Population)



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| PSD Responses to Individual Questions <question></question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions Question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Question | | | |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions Question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Question | | | |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions<br>Question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions Question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Question | | | |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions<br>Question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.12.1 for the following:

Table 14.2.12.2: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Per-Protocol Population)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| tch-Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| -Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| -Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| -Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | xx.x | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| h-Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.13.1 for the following:

Table 14.2.13.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Per-Protocol Population)



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| DLQI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| QI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| QI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| Į | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| LQI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.

Repeat Table 14.2.14.1 for the following:

Table 14.2.14.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Per-Protocol Population)



Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population)


| VRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population)


| NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 4 | (2: 122) | (1. 122) | (1, 1111) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population)


| NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 8 | | | (= : ====) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Repeat Table 14.2.15.1 for the following: Table 14.2.15.2: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Per-Protocol Population)



Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population)


| Score Type> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population)

| Score Type> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population)


| Score Type> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |


Repeat Table 14.2.16.1 for the following:

Table 14.2.16.2: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Per-Protocol Population)



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.17.1 for the following:

Table 14.2.17.2: Summary of Whole Body Investigator Global Assessment (IGA) (Per-Protocol Population)



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | | |
| 0-Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| 0-Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | $xx(x_0\%)$ | XX (XX.X%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.18.1 for the following:

Table 14.2.18.2: Summary of Intertriginous Area Investigator Global Assessment (I-IGA) (Per-Protocol Population)

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.



Table 14.3.0.1.1: Summary of Extent of Exposure (Safety Population)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Number of Doses | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Amount of Drug Applied (g) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Compliant <sup>a</sup> | | | |
| n | XX | XX | XX |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> A subject is considered compliant with the dosing regimen if the subject applied at least 80% of the expected doses during the dosing period and did not miss more than 3 consecutive doses.



Table 14.3.0.2.1: Summary of Pre-Dose Pharmacokinetic Concentrations (PK Population) (Page 1 of xx)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.0.2.1: Summary of Pre-Dose Pharmacokinetic Concentrations (PK Population) (Page 2 of xx)

| <parameter> (<units>) Week 12</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.0.2.2: Summary of Additional Pharmacokinetic Concentrations
(PK Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| 72 hr (3 days) | (IN-XX) | (IN-XX) | (IV-XX) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| 120 hr (5 days) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| 168 hr (7 days) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| 216 hr (9 days) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | , | , | , |
| Minimal edema or minimal papular response | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Subject Local Tolerability Sensation Following Drug Application Baseline | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | xx ( xx.x%) | XX (XX.X%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | AA ( AA.A/0) | AA ( AA.A.70) | AA ( AA.A70) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Week 4 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | AA ( AA.A/0) | AA ( AAAA70) | AA ( AAAA70) |
| Minimal edema or minimal papular response | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Subject Local Tolerability Sensation Following<br>Drug Application<br>Week 4 | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Week 8 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | Mr ( Min, v) | Mr ( MM/70) | mi (min, v) |
| Minimal edema or minimal papular response | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Subject Local Tolerability Sensation Following<br>Drug Application<br>Week 8 | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Week 12 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | m (mm/o) | Mr ( MM/70) | mi (min, v) |
| Minimal edema or minimal papular response | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Subject Local Tolerability Sensation Following<br>Drug Application | | | |
| Week 12 | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Figure 14.3.1.1: Subject Local Tolerability Sensation Following Drug Application (Safety Population)



Note: 0 (No sensation), 1 (Slight warm, tingling sensation; not really bothersome), 2 (Definite warm, tingling sensation that is somewhat bothersome),

3 (Hot, tingling/stinging sensation that has caused definite discomfort)



Table 14.3.1.2.1: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Injurious Behavior without Suicidal Intent Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population)

| Events during treatment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Suicidal Ideation (1-5) | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| 1) Wish to be dead | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2) Non-specific active suicidal thoughts | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3) Active suicidal ideation with any methods (not plan) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| without intent to act | AA ( AA.A/0) | AA ( AA.A/0) | AA ( AA.A/0) |
| 4) Active suicidal ideation with some intent to act, without | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| specific plan | AA ( AA.A/0) | AA ( AA.A/0) | AA ( AA.A/0) |
| 5) Active suicidal ideation with specific plan and intent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3) Active suicidal ideation with specific plan and intent | AA ( AA.A/0) | AA ( AA.A/0) | AA ( AA.A/0) |
| Suicidal Behavior (6-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6) Preparatory acts or behavior | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7) Aborted attempt | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 8) Interrupted attempt | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| 9) Non-fatal suicide attempt | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| 10) Completed suicide | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| , 1 | , | , | , |
| Suicidal Ideation or Behavior (1-10) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| | ` , | , | ` / |
| Self-injurious behavior without suicidal intent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| | ` , | . , | . , |



Table 14.3.1.2.2: Number of Patients with Suicide-Related Treatment-Emergent Events Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During
Treatment
(Safety Population)

| Treatment-emergent (TE) Events TE suicidal ideation (1-5) compared to recent history <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx)<br>xx ( xx.x%) | ARQ-151 Cream 0.15%<br>(N=xx)<br>xx ( xx.x%) | Vehicle Cream (N=xx) xx ( xx.x%) |
|---|---|---|---|
| TE serious suicidal ideation (0-3 to 4-5) compared to recent history <sup>b</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Emergence of serious suicidal ideation (0 to 4-5) compared to recent history <sup>c</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Improvement in suicidal ideation at endpoint compared with baseline <sup>d</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Emergence of suicidal behavior (6-10) compared to all prior history <sup>e</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> N=Number of enrolled patients with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the comparison period is non-missing and <5.

<sup>&</sup>lt;sup>b</sup> N=Number of enrolled patients with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the comparison period is 0-3.

<sup>&</sup>lt;sup>c</sup> N=Number of enrolled patients with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the comparison period is 0.

<sup>&</sup>lt;sup>d</sup> N=Number of enrolled patients whose suicidal ideation score is non-missing and >0 just prior to treatment.

<sup>&</sup>lt;sup>e</sup>N=number of enrolled patients with with at least one post-baseline C-SSRS assessment and who did not have suicidal behavior (6-10) prior to treatment.



Table 14.3.1.3.1: Summary of PHQ-8 Assessments by Treatment Group (Safety Population)

| DHO 8 Aggagament | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| PHQ-8 Assessment<br>Baseline | (N-XX) | (IN-XX) | (N-XX) |
| n | XX | | |
| None – Minimal Depression (0 to 4) | ( 0() | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | ` , | 200 | |
| Moderate Depression (10 to 14) | xx ( xx.x%) | . , | XX ( XX.X%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | | |
| n<br>N N N N N N N N N N N N N N N N N N N | XX | XX | XX |
| None – Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | | |
| n | XX | XX | XX |
| None – Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | | |
| n | XX | XX | XX |
| None – Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population)


| PHQ-8 for (ARQ-151 Cream 0.3%) | | | Week 4 | | |
|---|---|---|---|---|---|
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 8 | | |
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | $xx \overline{(xx.x\%)}$ |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 12 | | |
| <u>Baseline</u> | <u>None</u> | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).



Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population)


| PHQ-8 for (ARQ-151 Cream 0.15%) | | | Week 4 | | |
|---|---|---|---|---|---|
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | xx (xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 8 | | |
| <u>Baseline</u> | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | xx (xx.x%) |
| Mild | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 12 | | |
| <u>Baseline</u> | <u>None</u> | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).



Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population)


| PHQ-8 for (Vehicle Cream) | | | Week 4 | | |
|---|---|---|---|---|---|
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | $xx \frac{30+315}{(xx.x\%)}$ |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 8 | | |
| <u>Baseline</u> | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | $xx \overline{(xx.x}\%)$ |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 12 | | |
| Baseline | None | <u>Mild</u> | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).



Table 14.3.1.4.1: Overall Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Subjects with any TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of TEAEs | XX | XX | XX |
| subjects with any Related TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related TEAEs | XX | XX | XX |
| subjects with any Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX |
| subjects with any Related Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Serious TEAEs | XX | XX | XX |
| ubjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ubjects who Discontinued Study Drug due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ubjects who Discontinued Study due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity By Subject | | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | |
| Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unrelated | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.4.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Table 14.3.1.4.3: Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug by MedDRA System Organ Class and Preferred Term

(Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | XX (XX.X%) | xx (xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Table 14.3.1.4.4: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | Severity <sup>b</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|---|
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.



Table 14.3.1.4.5: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)


| System Organ Class <sup>a</sup><br>Preferred Term | Relationship | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|---|
| Total | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| | Possibly | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.



Table 14.3.1.4.6: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Subjects with any Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX |
| Subjects with any Related Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Serious TEAEs | XX | XX | XX |
| Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Subjects who Discontinued Study Drug due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Subjects who Discontinued Study due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity By Subject | | | |
| Grade 5 | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 4 | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | |
| Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unlikely | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unrelated | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset after first dose of study drug. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.3.1.4.7: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Table 14.3.1.4.8: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | Severity <sup>b</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|---|
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| , | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.


Table 14.3.1.4.9: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)

| System Organ Class <sup>a</sup> | | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|---|
| Preferred Term | <u>Relationship</u> | (N=xx) | (N=xx) | (N=xx) |
| Total | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: Treatment-emergent adverse events are those with an onset after first dose of study drug.



Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results
(Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results (Safety Population)

| Parameter> ( <units>)<br/>Week 12</units> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

Repeat Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results

For the following tables:

Table 14.3.1.5.1.2: Summary of Hematology Laboratory Results (Safety Population)

Table 14.3.1.5.1.3: Summary of Quantitative Urinalysis Laboratory Results (Safety Population)



# Table 14.3.1.5.2.1: Shift Summary of Chemistry Laboratory Results (Safety Population) (Page 1 of x)

| <test name=""> (<units>)</units></test> | AF | Q-151 Cream (<br>(N=xx) | 0.3% | ARG | Q-151 Cream 0<br>(N=xx) | .15% | | Vehicle Cream<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|
| | | Week 4 | | | Week 4 | | | Week 4 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) xx | x ( xx.x%) |
| WNL | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx ( xx.x%) xx | x ( xx.x%) |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) xx | x ( xx.x%) |
| | | Week 12 | | | Week 12 | | | Week 12 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | $\overline{xx(xx.x\%)}$ | xx( xx.x%) | xx ( xx.x%) | xx( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx( xx.x%) | xx ( xx.x%) xx | x ( xx.x%) |
| WNL | xx ( xx.x%) | xx(xx.x%) | xx(xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx ( xx.x%) xx | x ( xx.x%) |
| ANL | xx ( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) xx | x ( xx.x%) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.3.1.5.2.1: Shift Summary of Chemistry Laboratory Results

For the following tables:

Table 14.3.1.5.2.2: Shift Summary of Hematology Laboratory Results (Safety Population)

Table 14.3.1.5.2.3: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population)



Table 14.3.1.6.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.6.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population)

| Parameter> ( <units>)<br/>Week 12</units> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.6.2: Shift Summary of Overall Electrocardiogram (ECG) Assessments (Safety Population)
(Page 1 of x)

| Overall ECG Assessment | | | Cream 0.3% | | Cream 0.15%<br>=xx) | | le Cream<br>=xx) |
|---|---|---|---|---|---|---|---|
| | | W | eek 4 | W | eek 4 | W | eek 4 |
| | <u>Baseline</u> | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal |
| | Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Abnormal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | We | eek 12 | We | eek 12 | We | eek 12 |
| | <b>Baseline</b> | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal |
| | Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Abnormal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 8 | (IV AA) | (IV AA) | (IV AA) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | xx.x |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| <parameter> (<units>) Week 16</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.2: Summary of Change in Body Weight Compared to Baseline (Safety Population)


| Change in Body Weight Compared to Baseline <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | (11-AA) | (IV-AX) | (IV-AA) |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx (xx.x%) | xx ( xx.x%) | XX (XX.X%) |
| Week 6 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |

<sup>&</sup>lt;sup>a</sup> Percentages may sum to over 100% due to the possibility of being included in more than one category. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.3.1.7.2: Summary of Change in Body Weight Compared to Baseline (Safety Population)


| Change in Body Weight Compared to Baseline <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Percentages may sum to over 100% due to the possibility of being included in more than one category. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



#### 11. INDEX OF PLANNED LISTINGS

| Listing 16.2.1.1: End of Study Information | 159 |
|---|---|
| Listing 16.2.1.2: Discontinued Subjects | 160 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations | 161 |
| Listing 16.2.2.2: Protocol Deviations | 162 |
| Listing 16.2.3: Analysis Populations | 163 |
| Listing 16.2.4.1: Subject Demographic Information | 164 |
| Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Cla<br>and Preferred Terms | |
| Listing 16.2.4.2.2: Medical/Surgical History | 166 |
| Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DD ATC Level 2 Terms and Preferred Names | |
| Listing 16.2.4.3.2: Prior and Concomitant Medications | 168 |
| Listing 16.2.4.4.1: Unique Therapies and Procedures Coded to MedDRA System Organ Cl and Preferred Terms | |
| Listing 16.2.4.4.2: Prior and Concomitant Therapies and Procedures | 170 |
| Listing 16.2.4.5: Physical Examination | 171 |
| Listing 16.2.5.1: Study Visit Compliance | 172 |
| Listing 16.2.5.2: Drug Accountability | 173 |
| Listing 16.2.5.3: Study Drug Application | 174 |
| Listing 16.2.5.4: Dosing Compliance | 175 |
| Listing 16.2.5.5: Dosing Deviations | 176 |
| Listing 16.2.6.1: Investigator Global Assessment (IGA) | 177 |
| Listing 16.2.6.2: Body Surface Area (BSA) Involved with Psoriasis | 178 |
| Listing 16.2.6.3: Modified Psoriasis Area and Severity Index (mPASI) | 179 |
| Listing 16.2.6.4: Numeric Rating Scale (NRS) Assessments/Sleep Loss | 180 |
| Listing 16.2.6.5.1: Dermatology Life Quality Index (DLQI) Questionnaire Descriptions | 181 |
| Listing 16.2.6.5.2: Dermatology Life Quality Index (DLQI) Questionnaire | 182 |
| Listing 16.2.6.6.1: Work Productivity and Activity Impairment (WPAI) Questionnaire Descriptions | 183 |
| Listing 16.2.6.6.2: Work Productivity and Activity Impairment (WPAI) Questionnaire | 184 |
| Listing 16.2.6.7: Columbia-Suicide Severity Rating Scale (C-SSRS) | 185 |



| Listing 16.2.6.8.1: Patient Health Questionnaire Depression Scale (PHQ-8) Question Descriptions | 186 |
|---|---|
| Listing 16.2.6.8.2: Patient Health Questionnaire Depression Scale (PHQ-8) | 187 |
| Listing 16.2.6.9.1: Psoriasis Symptom Diary (PSD) Questionnaire Descriptions | 188 |
| Listing 16.2.6.9.2: Psoriasis Symptom Diary (PSD) Questionnaire | 189 |
| Listing 16.2.6.10: Photography Information | 190 |
| Listing 16.2.7.1.1: Investigator Local Tolerability Assessment | 191 |
| Listing 16.2.7.1.2: Subject Local Tolerability Assessment | 192 |
| Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes an Preferred Terms | |
| Listing 16.2.7.2.2: Treatment-Emergent Adverse Events | 194 |
| Listing 16.2.7.2.3: Serious Adverse Events | 195 |
| Listing 16.2.7.2.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse | Events 196 |
| Listing 16.2.8.1: Urine Pregnancy Test Results | 197 |
| Listing 16.2.8.2.1: Laboratory Test Results | 198 |
| Listing 16.2.8.2.2: Abnormal Laboratory Results | 199 |
| Listing 16.2.8.3: 12-lead Electrocardiogram Test Results | 200 |
| Listing 16.2.8.4: Vital Signs | 201 |
| Listing 16.2.8.5: Pharmacokinetics Blood Sample Collections | 202 |



## Listing 16.2.1.1: End of Study Information Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | F: Date of First Dose of Dru<br>L: Date of Last Dose of Drug | | Date of Completion/Discontinuation |
|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxxxxxxxx<br>L: xxxxxxxxxx | xxxxxxxxx xx xxxxxxxxxxxxx | xxxxxxxxx xxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxx | ********** | xxxxxxxxx xxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxx | xxxxxxxx xxxx xxxxxxx xxxx | xxxxxxxx xxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Note to programmer: concatenate 'Describe' text onto Primary Reason where applicable.



## Listing 16.2.1.2: Discontinued Subjects Treatment Group (Page xx of yy)

| S: Subject | | | |
|---|---|---|---|
| A: Age/Sex | F: Date of First Dose of Dr | | |
| E: Eval | L: Date of Last Dose of Dru | g Completion/Discontinuation | Date of Completion/Discontinuation |
| S: xxxxxx | F: xxxxxxxxx | ********* ** ********** | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxxx | | |
| E: xxxxxxxxx | | | |
| S: xxxxxx | F: xxxxxxxxx | xxxxxxxxx xx xxxxxxxxxxxxx | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxx | | |
| E: xxxxxxxxx | | | |
| S: xxxxxx | F: xxxxxxxxx | xxxxxxxx xxxx xxxxxxx xxxxx | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxx | | |
| E: xxxxxxxxx | | | |

\_\_\_\_\_



## Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Criterion<br>Category | Criterion<br>Identifier | Description |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | Х | ******* **** **** * ***** ** * ******* ** * |
| | | | xxxxxxxx | х | ******* **** **** * ***** ** * ******** |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxx | х | ******* **** **** * ***** ** * ******** |
| | | | xxxxxxxx | xx | ******** **** ***** **** **** ****** **** |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | х | ******* **** **** * ***** ** * ******** |
| | | | xxxxxxxx | xx | ******* **** **** * **** ** * ******* ** * |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Criterion Category, and Criterion Identifier.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



## Listing 16.2.2.2: Protocol Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Protocol Deviation |
|---------|---------|----------|----------------------------------------------|
| xxxxxx | xxxx | xxxxxxxx | XXXXXXXXX XXXX X XXXXXXX XX X XXXXXXXX |
| xxxxxx | xxxx | xxxxxxxx | XXXXXXXX X XXXXXX XXXXXXXXX XX XXX<br>XXXXXX |
| xxxxxx | xxxx | xxxxxxxx | ********* **** * **** * * ******* |
| xxxxxx | xxxx | xxxxxxxx | XXXXXXXX X XXXXXX XXXXXXXX XXXXXXXX XX |



## Listing 16.2.3: Analysis Populations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Population | Included | Reason(s) Excluded |
|---|---|---|---|---|
| xxxxxx | xxxx | Safety | XX | xxxxxx x xxxxxx xxxxxxxx |
| 212121212121 | 21212121 | Intent-to-Treat | XXX | |
| | | Per-Protocol | XXX | |
| | | Pharmacokinetic | XXX | |
| xxxxx | xxxx | Safety | xxx | |
| | | Intent-to-Treat | XXX | |
| | | Per-Protocol | XXX | |
| | | Pharmacokinetic | XXX | |
| xxxxx | XXXX | Safety | xxx | |
| | | Intent-to-Treat | XXX | |
| | | Per-Protocol | XX | xxxxxx xxxxxx xxxx |
| | | Pharmacokinetic | XX | ******* ******* ******** *** ******* ** **** |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, and Population.



#### Listing 16.2.4.1: Subject Demographic Information (Page xx of yy)

| Subject | Eval | B: Date of Birth<br>S: Sex | D: Date/Time of Informed Consent A: Age at Consent | R: Race<br>E: Ethnicity | C: Childbearing Potential B: Birth Control Method | P: Did the Subject<br>Consent to Photography?<br>D: Date of<br>Photography Consent |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxx | B: xxxxxxxxxx<br>S: xxxx | D: xxxx-xx-xxTxx:xx:xx<br>A: xx | R: xxxxx xx xxxxxxx<br>E: xxx xxxxxxx xx | C: xx<br>B: | P: xxx<br>D: xxxxxxxxx |
| xxxxx | xxxxxxx | B: xxxxxxxxxx<br>S: xxxxxx | D: xxxx-xx-xxTxx:xx<br>A: xx | R: xxxxx<br>E: xxx xxxxxxx xx | C: xxx<br>B: xxxxxxxxx xxxxxxx | P: xx<br>D: |
| xxxxxx | xxxxxxxx | B: xxxxxxxxxx<br>S: xxxxxx | D: xxxx-xx-xxTxx:xx:xx<br>A: xx | R: xxxxx<br>E: xxx xxxxxxx xx | C: xxx<br>B: xxxx xxxxxxxxxxxxx | P: xxx<br>D: xxxxxxxxx |



#### Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Condition/Surgery Verbatim Term |
|---|---|---|
| x xxx xxxxx | xxxx xxx xxxxx | xxxx xxxxxxxxx xx xxxxxx |
| | | xxxxx xxx xxxxxx xx |
| xxxx x xxxxxxxxx | xxxxxx xxxxxxxxxx | xxxx xxxxxx xxxxxxxx xx xxxxxx |
| xxxx xxx xxxxx | xxxx xxx xxxxx | xxxx xxxxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, and Verbatim Term.



### Listing 16.2.4.2.2: Medical/Surgical History Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Condition/Surgery<br>Verbatim Term | P: MedDRA Preferred Term S: MedDRA System Organ Class | S: Onset Date E: End Date |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxx xxxxxxx (xxxxxxxx xxxxx) | P: xxxxxx xxxxxxxxx<br>S: xxxxxxxxxx xxxxxxx | S: xxxxxxxxxx<br>E: xxxxxxxxxx |
| | | | xxxxxxx xxxxxxxxx | P: xxxxxx xxxxxxx<br>S: xxxxx xxxxxxxxxx | S: xxxxxxxxxx<br>E: xxxxxxxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Medical Condition/Surgery, Start Date, and End Date.



#### Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DD ATC Level 2 Terms and Preferred Names (Page xx of yy)

| ATC Level 2 Term | Preferred Name | Medication Name | I: Indication<br>R: Route |
|---|---|---|---|
| ****** ****** ** *** | xxxxxxxxx | xxxxxxxxx | I: xxxxxx xxxxxxx<br>R: xxxx |
| | xxxxxxx x | xxxxxx | I: xxxxxxx xxxxxxx<br>xxxxxxxxxxx<br>R: xxxx |
| | xxxxxxxxx | xxxxxxxx | I: xxxxxx xxxxxxx xxxx<br>xxxx xxxxxxx<br>R: xxxx |

Note: Preferred Name and ATC Level 2 Term map to the WHO-DD (Version March 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Preferred Name, Medication Name, Indication, and Route.



#### Listing 16.2.4.3.2: Prior and Concomitant Medications Treatment Group (Page xx of yy)

M: Medication Name D: Dose P: Preferred Name F: Date of First Dose U: Units A: ATC Level 2 Term S: Start Date (Day) 1 F: Frequency Subject Age/Sex I: Indication E: End Date (Day) 1 Eval R: Route XXXXXX XXXX XXXXXXXXX M: xxxxxxxxxxxx F: xxxxxxxxxx D: xx U: xx P: xxxxxxxxxxxx S: xxxxxxxxxx A: xxxxxxxxxxxx E: xxxxxxxxxx F: xxxx I: xxxxxxxx R:xxxx M: xxxxxxxxxxx F: xxxxxxxxxx D: xxxxx P: xxxxxxxxxxxx S: xxxxxxxxxx U: xx E: xxxxxxxxxx F: xx A: xxxxxxxxxxxx I: xxxxxxxx R:xxxx M: xxxxxxxxxxxx F: xxxxxxxxxx D: xxx XXXXXX XXXX XXXXXXXXX P: xxxxxxxxxxxx S: xxxxxxxxxx U: xx F: xx A: xxxxxxxxxxxx E: xxxxxxxxxx I: xxxxxxxx R:xxxx

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route. If ongoing, include 'Ongoing' in place of End Date. Concatenate Topical Area Treated onto route where applicable.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose. Note: Preferred Name and ATC Level 2 Term map to the WHO-DD (Version March 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



#### Listing 16.2.4.4.1: Unique Therapies and Procedures Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Procedure/Therapy Verbatim Term |
|---|---|---|
| xxxx xxx xxxxx | xxxx xxx xxxxx | xxxx |
| | | xxxxxx xxxxxxxx xx xxxxxx |
| | | ****** ******** ** ***** |
| xxxx xxx xxxxx | xxxx xxx xxxxx | xxxx |
| Anna Anna Anna | Ann Ann Anna | ****** ******** ** ***** |
| | | XXXXXX XXXXXXXXX XX XXXXX |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, MedDRA Preferred Term, and Procedure/Therapy Verbatim Term.



#### Listing 16.2.4.4.2: Prior and Concomitant Therapies and Procedures (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | Procedure/Therapy Verbatim Term | I: Indication A: Anatomical Area | P: MedDRA Preferred Term S: MedDRA System Organ Class | S: Start Date<br>E: End Date |
|---|---|---|---|---|
| S: xxxxxx | xxxxx xxxxxxx (xxxxxxx xxxxx) | I: xxxxxxxxx | P: xxxxxx xxxxxxxxx | S: xxxxxxxxxx |
| A: XXXX | | A: xxxx | S: xxxxxxxxxx xxxxxx | E: xxxxxxxxxx |
| : xxxxxxxx | | | | |
| | xxxxxx xxxxxxx xxxxxxx | I: xxxxxxxxx xxxxx | P: xxxxxx xxxxxxxxx | S: xxxxxxxxxxx |
| | | A: | S: xxxxxxxxxx xxxxxxx | E: xxxxxxxxxx |
| S: xxxxxx | xxxxxx xxxxxxxxxxxxx | I: xxxxxxxxx xxxxx | P: xxxxxx xxxxxxxxxx | S: xxxxxxxxxx |
| A: XXXX | | A: xxxx xxx xxxxx | S: xxxxxxxxxx xxxxxx | E: xxxxxxxxxx |
| E: xxxxxxxx | | | | |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Procedure/Therapy, Indication. If ongoing, include 'Ongoing' in place of End Date.



## Listing 16.2.4.5: Physical Examination Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | Visit | Date | Body System Assessed | Finding | Abnormal Finding<br>Specification |
|---|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | xxxxxxxxx | xxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis)<br><other, specify=""></other,> | XXXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | ****** |
| | xxxxxxxxxx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxx<br>xxxxx xxxxxxx<br>xxxxxxxx | |
| | xxxx xx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxx<br>xxxxx xxxxxxx | |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | xxxxxxxxxx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxxx<br>xxxxxxxxx xx<br>xxxx xxxxxxxx | xxxxxx |
| | xxxxxxxxx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxx xxxxx<br>xxxxxxxx | |
| | xxxx xx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxx<br>xxxxxxxxx | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, Body System Assessed.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



## Listing 16.2.5.1: Study Visit Compliance Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Visit Date | Study<br>Day¹ | Within Visit<br>Window | Days Out of<br>Window <sup>2</sup> |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | Х | xxx | |
| | | | xxxxxxxx | xxxxxxxxx | Х | xxx | |
| | | | XXXX X | xxxxxxxxx | xx | XXX | xxxx |
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx to xxxxxxxxx | x | XXX | |
| | | | xxxxxxxx | xxxxxxxxx | Х | XXX | |
| | | | xxxx x | xxxxxxxxx | XX | XXX | |
| | | | XXXX X | xxxxxxxxx | XX | XXX | |
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | XX | XXX | |
| | | | xxxxxxxx | xxxxxxxxx | Х | XXX | |
| | | | xxxx x | xxxxxxxxx | XX | XXX | |

Listing sorted by Subject, Visit, Visit Date.

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - baseline date for dates prior to baseline visit. Otherwise, day is calculated as date - baseline date + 1 for dates on or after baseline visit.

 $<sup>^{2}</sup>$  Populated only for post baseline visits that are planned and out of window. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



## Listing 16.2.5.2: Drug Accountability Treatment Group (Page xx of yy)

| ubject | Age/Sex | Evaluable | Kit Number | Date<br>Dispensed | Date<br>Returned | Tube ID | Dispensed<br>Weight (g) | Returned<br>Weight (g) |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | Х | XX.X | XX.X |
| | | | | | | Х | XX.X | XX.X |
| | | | | | | Х | xx.x | XX.X |
| | | | | | | Х | xx.x | XX.X |
| | | | xxxxx | xxxxxxxx | xxxxxxxxx | Х | xx.x | XX.X |
| | | | | | | X | xx.x | XX.X |
| | | | | | | Х | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | XXXXX | XXXXXXXXX | XXXXXXXXX | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | Х | XX.X | XX.X |
| xxxx | XXXX | xxxxxxx | xxxxx | xxxxxxxxx | xxxxxxxx | х | xx.x | xx.x |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | XXXXX | XXXXXXXXX | XXXXXXXXX | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Kit Number, Date Dispensed, Date Returned, and Tube ID.



## Listing 16.2.5.3: Study Drug Application Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date/Time of Study<br>Drug Application | Study Drug<br>Applied in Clinic? | Pre-Dose<br>Weight (g) | Post-Dose<br>Weight (g) | Reason<br>Not Done |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | XXXXX | xxxxxTxxxx | xxx | XX.X | XX.X | |
| | | | XXXXX | XXXXTXXXX | XXX | XX.X | XX.X | |
| | | | XXXXX | XXXXXTXXXX | XXX | XX.X | XX.X | |
| xxxxx | xxxx | xxxxxxx | xxxxx<br>xxxxx | xxxxxTxxxx<br>xxxxxTxxxx<br>xxxxxTxxxx | xx<br>xxx<br>xxx | xx.x<br>xx.x | xx.x<br>xx.x | xxx xxx xxxxx |
| xxxxxx | xxxx | xxxxxxx | xxxxx<br>xxxxx | xxxxxTxxxx<br>xxxxxTxxxx<br>xxxxxTxxxx | xxx<br>xxx<br>xxx | xx.x<br>xx.x<br>xx.x | xx.x<br>xx.x<br>xx.x | |
| xxxxx | xxxx | xxxxxxx | xxxxx<br>xxxxx | xxxxxTxxxx<br>xxxxxTxxxx<br>xxxxxTxxxx | xx<br>xxx<br>xxx | xx.x<br>xx.x | xx.x<br>xx.x | xxx xxx xxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Date/Time of Study Drug Application, Visit.



### Listing 16.2.5.4: Dosing Compliance Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | D: Date of First Dose<br>R: Date of Last Dose | Number of<br>Days of<br>Exposure | Calculated¹<br>Number of<br>Doses | Amount of<br>Study Drug<br>Used (g) | Maximum Number<br>of Missed<br>Consecutive Doses | Percent<br>Compliant | Compliant? <sup>2</sup> |
|---|---|---|---|---|---|---|---|
| S: xxxxx<br>A: xxxx<br>E: xxxxxxxx | D: xxxxxxxxxxx<br>R: xxxxxxxxxxx | xx | xx | xxxx | х | xxx | xxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | D: xxxxxxxxxxxx<br>R: xxxxxxxxxxxx | xx | xx | xxxx | х | xxx | xx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | D: xxxxxxxxxxx<br>R: xxxxxxxxxxx | xx | xx | xxxx | | xxxx | xxx |

<sup>&</sup>lt;sup>1</sup> The total number of doses was calculated from the date of first dose and the date of last known dose minus the missed doses plus additional dose deviations.

<sup>&</sup>lt;sup>2</sup> A subject was considered compliant with the dosing regimen if the subject applied at least 80% of the expected doses during the study drug application period and did not miss more than 3 consecutive doses.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



## Listing 16.2.5.5: Dosing Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Date of First Dose | Date of Dosing Deviation | Number of Doses Applied |
|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | ************************************** | х<br>х<br>х |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | x<br>x |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx<br>xxxxxxxxx | x<br>x |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, and Date of Dosing Deviation.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Listing 16.2.6.1: Investigator Global Assessment (IGA)

Treatment Group

(Page xx of yy)

| S: Subject<br>A: Age/Sex<br>B: Eval | Visit | Date of<br>Assessment | Whole Body<br>Investigator Global<br>Assessment Score | Does the Subject have Intertriginous Area involvement? | Intertriginous<br>Investigator Global<br>Assessment Score | Evaluator<br>Initials |
|---|---|---|---|---|---|---|
| : xxxxx<br>: xxxx | SCREENING | xxxxxxxxx | x x xxxxxxx | xxx | x x xxxxxxxx | xxx |
| • AAAAAAA | BASELINE | xxxxxxxxx | x x xxxxxxxx | xxx | x x xxxxxxxx | xxx |
| | WEEK 2 | XXXXXXXXX | x x xxxxxxx | XXX | x x xxxxxxx | XXX |
| | WEEK 4 | XXXXXXXXX | x x xxxxxxx | XXX | x x xxxxxxx | XXX |
| | WEEK 6 | xxxxxxxxx | x x xxxxxxxx | XXX | x x xxxxxxxx | XXX |
| | WEEK 8 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |
| | WEEK 12 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |
| | WEEK 16 | xxxxxxxxx | x x xxxxxxxx | XX | | xxx |
| 5: xxxxxx<br>4: xxxx | SCREENING | xxxxxxxxx | x x xxxxxxxx | xx | | x-x |
| | BASELINE | XXXXXXXXX | x x xxxxxxxx | XX | | x-x |
| | WEEK 2 | XXXXXXXXX | x x xxxxxxx | XX | | x-x |
| | WEEK 4 | xxxxxxxxx | x x xxxxxxxx | XX | | x-x |
| | WEEK 6 | xxxxxxxxx | x x xxxxxxxx | XX | | xxx |
| | WEEK 8 | xxxxxxxxx | x x xxxxxxxx | XX | | xxx |
| | WEEK 12 | XXXXXXXXX | x x xxxxxxxx | XX | | XXX |
| | WEEK 16 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |

Listing sorted by Subject, Visit, and Date of Assessment.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



## Listing 16.2.6.2: Body Surface Area (BSA) Involved with Psoriasis Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of Assessment | BSA¹ (%) | Evaluator Initials |
|---|---|---|---|---|---|---|
| XXXXXXX | XXXX | XXXXXXXX | XXXXXXX | XXXXXXXX | XX.X | XXX |
| | | | XXXXXXXX | XXXXXXXXX | XX.X | XXX |
| | | | xxxx x | XXXXXXXXX | XX.X | XXX |
| | | | XXXX X | XXXXXXXXX | XX.X | XXX |
| | | | XXXX X | XXXXXXXXX | XX.X | XXX |
| | | | XXXX X | XXXXXXXXX | XX.X | XXX |
| | | | XXXX XX | XXXXXXXXX | XX.X | XXX |
| xxxxxxx | xxxx | xxxxxxxx | XXXXXXX | xxxxxxxxx | xx.x | xxx |
| 21212121212121 | 21212121 | 2121212121212121 | XXXXXXXXX | XXXXXXXXX | XX.X | XXX |
| | | | XXXX X | XXXXXXXX | XX.X | XXX |
| | | | xxxx x | XXXXXXXXX | XX.X | XXX |
| | | | XXXX X | XXXXXXXXX | XX.X | XXX |
| | | | XXXX X | XXXXXXXXX | XX.X | XXX |
| | | | XXXX XX | XXXXXXXXX | XX.X | XXX |

Listing sorted by Subject, Visit, Date of Assessment.

<sup>1</sup> Body Surface Area (BSA) involved with psoriasis (excluding the scalp, palms and soles).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Listing 16.2.6.3: Modified Psoriasis Area and Severity Index (mPASI)

Treatment Group

(Page xx of yy)

| S: Subject | V: Visit<br>D: Date | | | | | |
|---|---|---|---|---|---|---|
| A: Age/Sex | E: Evaluator | Affected | Percent of | | Parameter Score | |
| E: Eval | Initials | Area | Skin Involved | Erythema (redness) | Induration (thickness) | Desquamation (scaling |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | V: SCREENING D: xxxxxxxxx E: xxx | Arms | xx-xx | x - xxxxxx xxxxxxx | x - xxxxxx xxxxxxx | x - xxxxxx xxxxxxx |
| | | Head | XX-XX | x - xxxxxxx xxxxxxx | x - xxxxxxx xxxxxxxx | x - xxxxxxx xxxxxxx |
| | | Legs | XX-XX | x - xxxx | x - xxxx | х |
| | | Trunk | X.X | x - xxxx | x - xxxx | Х |
| | V: BASELINE<br>D: xxxxxxxxx<br>E: xxx | Arms | х.х | х | х | х |
| | | Head | X.X | x - xxxxxxx xxxxxxx | x - xxxxxxx xxxxxxx | x - xxxxxxx xxxxxxx |
| | | Legs | XX-XX | x - xxxx | x - xxxx | X |
| | | Trunk | XX-XX | x - xxxx | x - xxxx | Х |
| | V: WEEK 2<br>D: xxxxxxxxxx<br>E: xxx | Arms | xx-xx | х | х | х |
| | | Head | XX-XX | x | x | х |
| | | Legs | XX-XX | x - xxxx | x - xxxx | x - xxxx |
| | | Trunk | XX-XX | x - xxxx | x - xxxx | x - xxxx |
| | V: WEEK 6 D: xxxxxxxxx E: xxx | Arms | xx-xx | x - xxxx | x - xxxx | х |
| | | Head | XX-XX | x - xxxx | X | x - xxxx |
| | | Legs | X.X | x - xxxx | x - xxxx | x - xxxx |
| | | Trunk | xx-xx | x - xxxx | x - xxxx | x - xxxx |

Listing sorted by Subject, Visit, Date, and Affected Area. If < 10% of skin involved, present actual percent involved.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Page 179 of 202


Listing 16.2.6.4: Numeric Rating Scale (NRS) Assessments/Sleep Loss
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Assessment | Patient Reported<br>Severity Score |
|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | SCREENING | xxxxxxxxx | xxxxxxxxx | x - xx xxxxxxx |
| | | | | | xxxxxxxxx xx | xx - xxxxx xxxxxxxxx xxxx |
| | | | | | xxxxxxxxxxxxxxxxxxxx | х |
| | | | BASELINE | xxxxxxxxx | xxxxxxxxxx | х |
| | | | | | xxxxxxxxx xx | X |
| | | | | | xxxxxxxxxxxxxxxxxxxx | x - xx xxxx-xxxxxxx xxxxx xxxx |
| | | | WEEK 2 | xxxxxxxxx | xxxxxxxxxx | х |
| | | | | | xxxxxxxxxx xx | Х |
| | | | | | xxxxxxxxxxxxxxxxxxxx | x - xx xxxx-xxxxxxx xxxxx xxxx |
| | | | WEEK 4 | xxxxxxxxx | xxxxxxxxxx | x - xx xxxx |
| | | | | | xxxxxxxxx xx | X |
| | | | | | xxxxxxxxxxxxxxxxxxx | x - xx xxxx-xxxxxxx xxxxx xxxx |
| | | | WEEK 6 | xxxxxxxxx | xxxxxxxxxx | x - xx xxxx |
| | | | | | XXXXXXXXXX XX | X |
| | | | | | xxxxxxxxxxxxxxxxxxx | x - xx xxxx-xxxxxx xxxxx xxxx |
| | | | WEEK 8 | XXXXXXXXX | xxxxxxxxxx | x - xx xxxx |
| | | | | | XXXXXXXXXX XX | X |
| | | | | | xxxxxxxxxxxxxxxxxxxx | x - xx xxxx-xxxxxx xxxxx xxxx |
| | | | WEEK 12 | xxxxxxxx | xxxxxxxxxx | x - xx xxxx |
| | | | | | xxxxxxxxx xx | Х |
| | | | | | XXXXXXXXXXXXXXXXXXXXXXX | x - xx xxxx-xxxxxxx xxxxx xxxx |

Note: Score is the patient-reported severity of this symptom at its highest intensity during the previous 24-hour period. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, and Assessment.



Listing 16.2.6.5.1: Dermatology Life Quality Index (DLQI) Questionnaire Descriptions

| Number | DLQI Question |
|---|---|
| 1 | Over the last week, how itchy, sore, painful or stinging has your skin been? |
| 2 | Over the last week, how embarrassed or self conscious have you been because of your skin? |
| 3 | Over the last week, how much has your skin interfered with you going shopping or looking after your home or garden? |
| 4 | Over the last week, how much has your skin influenced the clothes you wear? |
| 5 | Over the last week, how much has your skin affected any social or leisure activities? |
| 6 | Over the last week, how much has your skin made it difficult for you to do any sport? |
| 7a | Over the last week, has your skin prevented you from working or studying? |
| 7b | If "No", over the last week how much has your skin been a problem at work or studying? |
| 8 | Over the last week, how much has your skin created problems with your partner or any of your close friends or relatives? |
| 9 | Over the last week, how much has your skin caused any sexual difficulties? |
| 10 | Over the last week, how much of a problem has the treatment for your skin been, for example by making your home messy, or by taking up time? |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Question Number.



Listing 16.2.6.5.2: Dermatology Life Quality Index (DLQI) Questionnaire Treatment Group (Page xx of yy)

| | | | | Data af | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 0.1.1.1 | 3 /0 | D 1 | **! - ! b | Date of | 1 | 0 | 2 | 4 | _ | _ | 7 - | 71. | 0 | 0 | 1.0 |
| Subject | Age/Sex | Eval | Visit | Assessment | 1 | 2 | 3 | 4 | 5 | 6 | 7a | 7b | 8 | 9 | 10 |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | x | × | x | x | х | Х | × | X | х | х | x |
| | 21212121 | 777777777777 | XXXXXXXX | XXXXXXXXXX | X | х | х | X | X | X | X | X | Х | X | X |
| | | | XXXX X | XXXXXXXXXX | X | Х | Х | X | X | X | X | X | X | X | X |
| | | | XXXX X | XXXXXXXXXX | X | Х | Х | X | X | X | X | X | X | X | X |
| | | | XXXX X | XXXXXXXXXX | X | X | X | X | | X | | X | | X | |
| | | | | | | | | | X | | х | | Х | | X |
| | | | XXXX XX | XXXXXXXXX | X | X | X | X | Х | Х | Х | Х | Х | Х | Х |
| XXXXX | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| | | | XXXXXXXX | XXXXXXXXX | X | X | X | X | X | X | X | X | X | X | X |
| | | | XXXX X | xxxxxxxxx | X | Х | Х | X | X | X | X | X | Х | Х | X |
| | | | XXXX X | XXXXXXXXX | Х | Х | Х | X | X | X | Х | X | Х | Х | X |
| | | | XXXX X | xxxxxxxxx | X | X | X | Х | Х | X | X | Х | Х | Х | X |
| | | | XXXX XX | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| XXXXX | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | х | Х | Х | х | Х | х | Х | Х | Х | Х | Х |
| | | | XXXXXXX | XXXXXXXXX | X | Х | Х | Х | Х | X | Х | Х | Х | Х | X |
| | | | xxxx x | XXXXXXXXX | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | Х |
| | | | xxxx x | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | Х | х | х | Х |
| | | | xxxx x | xxxxxxxxx | Х | х | х | х | х | х | Х | х | х | х | X |
| | | | xxxx xx | xxxxxxxxx | х | х | х | х | х | х | х | х | х | х | X |

Note: Questions 1-6, 7b-10: 1 = Very much, 2 = A lot, 3 = A little, 4 = Not at all. Question 7a: 1 = Yes, 0 = No. NR = Not relevant.

ND = Not done.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Date of assessment



Listing 16.2.6.6.1: Work Productivity and Activity Impairment (WPAI) Questionnaire Descriptions

| Number | WPAI Question |
|---|---|
| 1 | Are you currently employed (working for pay)? |
| 2 | During the past seven days, how many hours did you miss from work because of problems associated with your psoriasis? Include hours you missed on sick days, times you went in late, left early, etc., because of your psoriasis. Do not include time you missed to participate in this study. |
| 3 | During the past seven days, how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study? |
| 4 | During the past seven days, how many hours did you actually work? |
| 5 | During the past seven days, how much did your psoriasis affect your productivity while you were working? |
| 6 | During the past seven days, how much did your psoriasis affect your ability to do your regular daily activities, other than work at a job? |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Question Number.



# Listing 16.2.6.6.2: Work Productivity and Activity Impairment (WPAI) Questionnaire Treatment Group (Page xx of yy)

| S: Subject A: Age/Sex E: Eval | V: Visit<br>D: Date of Assessment | 1. Employed | 2. Psoriasis<br>Hours Missed | 3. Other<br>Hours Missed | | 5. Productivity<br>Affected | 6. Regular Activities<br>Affected |
|---|---|---|---|---|---|---|---|
| S: xxxxxx<br>A: xx xxxx<br>E: xx xx | V: xxxx<br>D: xxxxxxx | xxx | xxx.x | xxx.x | xxx.x | х | х |
| | V: xxxx<br>D: xxxxxxx | xxx | xxx.x | xxx.x | xxx.x | х | х |
| S: xxxxxx<br>A: xx xxxx<br>E: xx xx | V: xxxx<br>D: xxxxxxx | xxx | xxx.x | xxx.x | xxx.x | х | х |
| D. AA AA | V: xxxx<br>D: xxxxxxx | xxx | XXX.X | xxx.x | xxx.x | x | х |

```
Note: Questions 2 - 5 are answered conditionally based on the response to Question 1.

Questions 2 - 4 are reported in hours.

Question 5: Scaled (0 - Psoriasis had no effect on my) to (10 - Psoriasis completely prevented me from working).

Question 6: Scaled (0 - Psoriasis had no effect on my daily activities) to (10 - Psoriasis completely prevented me from doing my daily activities).
```

ND = Not done.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Date of assessment



# Listing 16.2.6.7: Columbia-Suicide Severity Rating Scale (C-SSRS) Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex | V: Visit | | | _ |
|---|---|---|---|---|
| : Eval | D: Date | Question | Time Period | Response |
| : xxxxxx | V: SCREENING | xxxx xx xx xxxx | xxxxxxx | XX |
| : xxxx | D: xxxxxxxxxx | | XXXX X XXXXXX | xxx xxxx |
| | | *** ****** ***** ****** | xxxxxxx | xxx |
| | | | xxxx x xxxxxx | xx |
| | | XXX XXXXXXX XXXXX XXXXXXX | XXXXXXX | XX |
| | | XXX XXXX XXXXXXX XXXXX XX XXX | XXXX X XXXXXX | XX |
| | | XXXXXX XXXXXXX XXXXXX XXXX | XXXXXXX | XX |
| | | XX XXX XXXXXXX XXXXXX XXXX | xxxx x xxxxxx | XX |
| | | XXXXXX XXXXXXX XXXXXXX XXXX | XXXXXXX | XXX |
| | | XXXX XXX XXXXXX | xxxx x xxxxxx | XX |
| | | xxxx xxxxxx xxxxxxx | XXXXXXX | х |
| | | | xxxx x xxxxxx | xxx xxxx |
| | | XXX XXXX XXXXX XXXX XXXX XXXX | XXXXXXX | X XXX XXXX |
| | | | XXXX X XXXXXX | XXX XXXX |
| | | XXXX XX XXX XXXX XXXXXX | XXXXXXX | X X XXX XX XX |
| | | XXX XXX XXXX XX XXXX | XXXX X XXXXXX | XXX XXXX |
| | | XXXXXXX XXXXXXX | XXXXXXX | XX |
| | | | XXXX X XXXXXX | XXX XXXX |
| | | XXX XXXXXX XXXXXX XX XXX XXXXX | XXXXXXX | XX |
| | | XXXXXXXXX XXXXXXX | xxxx x xxxxxx | XX |
| | | XXXXXXXX XXXXXXX | XXXXXXX | XXX XXXXX |
| | | | XXXX X XXXXXX | xxx xxxx |
| | V: BASELINE<br>D: xxxxxxxxxx | XXXX XX XX XXXX | xxxxx xxxx xxxxx | xx |
| | | xxx xxxxxxx xxxxx xxxxxxxx xxxxxxx | xxxxx xxxx xxxxx | xx |
| | | XXX XXXXXXX XXXXX XXXXXXX | XXXXX XXXX XXXXX | XX |
| | | XXX XXXX XXXXXXX XXXXX XX XXX | | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, Question (in order in CRF), and Time Period (in order in CRF). All additional information (such as description, number of attempts) will be concatenated onto the response for the main question.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Listing 16.2.6.8.1: Patient Health Questionnaire Depression Scale (PHQ-8) Question Descriptions

| Number | PHQ-8 Question |
|---|---|
| 1 | How often during the past 2 weeks were you bothered by: Little interest or pleasure in doing things? |
| 2 | How often during the past 2 weeks were you bothered by: Feeling down, depressed, or hopeless? |
| 3 | How often during the past 2 weeks were you bothered by: Trouble falling or staying asleep, or sleeping too much? |
| 4 | How often during the past 2 weeks were you bothered by: Feeling tired or having little energy? |
| 5 | How often during the past 2 weeks were you bothered by: Poor appetite or overeating? |
| 6 | How often during the past 2 weeks were you bothered by: Feeling bad about yourself, or that you are a failure, or have let yourself or your family down? |
| 7 | How often during the past 2 weeks were you bothered by: Trouble concentrating on things, such as reading the newspaper or watching television? |
| 8 | How often during the past 2 weeks were you bothered by: Moving or speaking so slowly that other people could have noticed. Or the opposite - being so fidgety or restless that you have been moving around a lot more than usual? |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Question Number.



# Listing 16.2.6.8.2: Patient Health Questionnaire Depression Scale (PHQ-8) Treatment Group (Page xx of yy)

| | | | | Date of | | - | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Age/Sex | Eval | Visit | Assessment | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| XXXXXX | XXXX | XXXXXXXX | XXXXXXXX | XXXXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXXXXXX | XXXXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXX X | XXXXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXX X | XXXXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXX XX | XXXXXXXXX | X | Х | Х | Х | X | X | X | X |
| xxxxx | xxxx | xxxxxxxx | XXXXXXXXX | xxxxxxxxx | х | х | х | х | Х | Х | х | Х |
| | | | XXXXXXX | XXXXXXXXX | х | Х | Х | Х | Х | Х | Х | Х |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | Х | Х | Х | Х | Х |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | Х | Х | Х | Х | X |
| | | | XXXX XX | XXXXXXXXX | Х | X | Х | Х | X | Х | Х | X |
| xxxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | X | X | Х | Х | X | X | X | X |
| | | *************************************** | XXXXXXXX | XXXXXXXXX | X | X | Х | Х | X | X | X | x |
| | | | XXXX X | XXXXXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXX X | XXXXXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXX XX | XXXXXXXXXX | X | X | X | X | X | X | X | X |
| | | | 222222 22 | MANAMANA A | Λ | Λ | Λ | Λ | Λ | Δ. | Λ | 23 |

Note: For all Questions: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day, ND = Not Done. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Date of Assessment.



Listing 16.2.6.9.1: Psoriasis Symptom Diary (PSD) Questionnaire Descriptions

| Number | PSD Question |
|---|---|
| 1 | Overall, how severe was your psoriasis-related itching over the past 24 hours? |
| 2 | Overall, how bothered were you by your psoriasis-related itching over the past 24 hours? |
| 3 | Overall, how severe was your psoriasis-related stinging over the past 24 hours? |
| 4 | Overall, how bothered were you by your psoriasis-related stinging over the past 24 hours? |
| 5 | Overall, how severe was your psoriasis-related burning over the past 24 hours? |
| 6 | Overall, how bothered were you by your psoriasis-related burning over the past 24 hours? |
| 7 | Overall, how severe was your psoriasis-affected skin cracking over the past 24 hours? |
| 8 | Overall, how bothered were you by your psoriasis-affected skin cracking over the past 24 hours? |
| 9 | Overall, how severe was your psoriasis-related pain over the past 24 hours? |
| 10 | Overall, how bothered were you by your psoriasis-related pain over the past 24 hours? |
| 11 | Overall, how severe was your psoriasis scaling over the past 24 hours? |
| 12 | Overall, how bothered were you by your psoriasis scaling over the past 24 hours? |
| 13 | Overall, how noticeable did you think the colour of your psoriasis-affected skin was over the past 24 hours? |
| 14 | Overall, how much did you try to hide your psoriasis-affected skin over the past 24 hours? |
| 15 | Overall, how much did your psoriasis cause you to avoid activities with other people over the past 24 hours? |
| 16 | Overall, how embarrassed were you because of your psoriasis over the past 24 hours? |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Question Number.



# Listing 16.2.6.9.2: Psoriasis Symptom Diary (PSD) Questionnaire Treatment Group (Page xx of yy)

| | | | | Date of | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cubicat | 700/001 | Erro 1 | Visit | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| Subject | Age/Sex | Eval | VISIC | Assessment | | | | 4 | | | | 0 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 10 |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | Х | х | Х | х | х | х | х | Х | х | х | Х | Х | Х | Х | Х | Х |
| | | | xxxxxxx | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | | | XXXX X | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| | | | XXXX X | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | | | XXXX X | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | | | xxxx xx | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| | | | XXXXXXXX | XXXXXXXXX | X | Х | Х | X | Х | Х | X | X | Х | X | Х | Х | Х | X | Х | X |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | X | Х | Х | X | X | Х | X | Х | Х | Х | X | Х | X |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | X | Х | Х | X | X | Х | X | Х | Х | X | X | Х | X |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х |
| | | | XXXX XX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | Х | Х | Х | X | X | X | X | х | Х | Х | X | Х | X | Х | X | Х |
| | | | XXXXXXXX | XXXXXXXXX | X | X | X | X | Х | Х | X | X | X | X | Х | X | X | X | Х | X |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х |
| | | | XXXX X | XXXXXXXXX | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х |
| | | | XXXX XX | XXXXXXXXX | X | Х | Х | X | Х | Х | X | X | Х | X | Х | Х | X | X | Х | X |

```
Note: Questions 1, 3, 5, 7, 9, 11: Scaled (0 - None) to (10 - As bad as you can imagine)
Questions 2, 4, 6, 8, 10, 12: Scaled (0 - Not bothered at all) to (10 - As bothered as you can imagine)
Question 13: Scaled (0 - Not at all noticeable) to (10 - As noticeable as you can imagine)
Question 14: Scaled (0 - Did not try to hide at all) to (10 - Totally avoided being seen by others)
Question 15: Scaled (0 - You did not avoid other people) to (10 - Avoided other people as much as you ever have)
Question 16: Scaled (0 - No embarrassment) to (10 - As embarrassed as you can imagine)
ND = Not done.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)
```

#### Listing sorted by Subject, Visit, and Date of assessment



# Listing 16.2.6.10: Photography Information Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Were Photographs Taken? | Date of Photograph |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxx | xxx | xxxxxxxxx |
| ΛΛΛΛΛ | AAAA | ΑΛΛΛΛΛΛ | XXXX X | XXX | XXXXXXXXX |
| | | | XXXX X | XXX | XXXXXXXXX |
| | | | XXXX X | XXX | XXXXXXXXX |
| | | | XXXX XX | | XXXXXXXXX |
| | | | **** | XXX | ******* |
| xxxxxx | XXXX | XXXXXXXXX | xxxxxxxx | xxx | xxxxxxxxx |
| | | | XXXX X | XXX | xxxxxxxxx |
| | | | XXXX X | XX | |
| | | | XXXX X | XXX | xxxxxxxxx |
| | | | xxxx xx | XXX | xxxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxx | xxxxxxxxx |
| | ******** | *************************************** | XXXX X | XX | *************************************** |
| | | | XXXX X | XXX | xxxxxxxxx |
| | | | XXXX X | XXX | XXXXXXXXX |
| | | | XXXX XX | XXX | XXXXXXXXX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Date of Photograph.



# Listing 16.2.7.1.1: Investigator Local Tolerability Assessment Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | V: Visit<br>D: Date<br>E: Evaluator Initials | Dermal Response | Other Effects<br>Assessed? | Other Effects<br>Present | Locations where Other<br>Effects are Present |
|---|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxx<br>D: xxxxxxxxx xxxx<br>E: xxx | **** ******* ******* | xxx | xxxxxx xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXX XXXXX<br>XXXX XXXXX XXXX XXXX |
| | V: xxxxxxxx<br>D: xxxxxxxxx xxxx<br>E: xxx | xxxx xxxxxxx xxxxxxx<br>xxxxxxxx xxxxxx | xxx | xxxxxx xxx xxxxxxxx | xxxx xxxxx xxxxxxx |
| | V: xxxxxxxx<br>D: xxxxxxxxx xxxx<br>E: xxx | xxxx xxxxxxx xxxxxxx<br>xxxxxxxx xxxxxx | xxx | xxxxxx xxx xxxxxxxx | xxxx |
| | V: xxxxxxxx<br>D: xxxxxxxxxx xxxx<br>E: xxx | xxxx xxxxxxx xxxxxxx<br>xxxxxxxx xxxxxx | xxx | xxxxxx xxx xxxxxxx | XXXX |
| S: xxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxx<br>D: xxxxxxxxx xxxx<br>E: xxx | **** ******* ******* | xxx | ****** ******************************* | XXXX XXXXX<br>XXXX<br>XXXX |
| | V: xxxxxxxx<br>D: xxxxxxxxx xxxx<br>E: xxx | xxxx xxxxxxx xxxxxxxx | xxx | xxxxxx xxx xxxxxxx | xxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Date.



# Listing 16.2.7.1.2: Subject Local Tolerability Assessment Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of Assessment | Subject Reported Tolerability |
|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXX | XXXXXXX | XXXXXXXXX | X XXXXXXXX |
| | | | XXXX X | XXXXXXXXX | X XXXXXXXXX |
| | | | XXXX X | XXXXXXXXX | X XXXX |
| | | | XXXX XX | XXXXXXXXX | X XXXX |
| XXXXXX | XXXX | XXXXXXXX | XXXXXXX | xxxxxxxxx | x xxxx |
| | | | xxxx x | xxxxxxxxx | X XXXX |
| | | | xxxx x | xxxxxxxxx | X XXXX |
| | | | xxxx xx | xxxxxxxxx | x xxxx |
| XXXXXX | XXXX | XXXXXXXX | XXXXXXX | xxxxxxxxx | x xxxx |
| | | | xxxx x | xxxxxxxxx | x xxxxxxx |
| | | | xxxx x | xxxxxxxxx | x xxxx |
| | | | xxxx xx | XXXXXXXXX | X XXXX |
| XXXXXX | XXXX | XXXXXXXX | xxxxxxxx | xxxxxxxxx | x xxxx |
| | | | xxxx x | xxxxxxxxx | x xxxx |
| | | | xxxx x | xxxxxxxxx | x xxxx |
| | | | XXXX XX | XXXXXXXXX | X XXXX |
| | | | AAAA AA | ΛΛΛΛΛΛΛΛΛ | A AAAA |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Date of Assessment.



# Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Adverse Event |
|---|---|---|
| ****** *** ******* ****** | xxxxxxx | xxxxxx |
| | | xxxxxx |
| | xxxxxxxxxx | xxxxxxxxxx |
| xxx xxx xxxxxxxx xxxxxxxx | xxxxxxx | xxxxxxx |
| xxx xxxxxxxx | xxxxxx xxxxxx xxxxxxx | xxxxxxxx xxxxx xxxxxx |
| xxxxxxxxxxxx xxxxxxx | xxxxxxxx xxxx | xxxxxxxx xxxx |
| | xxxxxxxx xxxxxxxxxxx | xxxxx xxxxxxxx xxxxxxxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, MedDRA Preferred Term, and Adverse Event.



# Listing 16.2.7.2.2: Treatment-Emergent Adverse Events Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | F: Date of First Dose S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> | G: Grade <sup>2</sup> R: Relationship to Study Drug O: Outcome | S: Serious Event? A: In Treatment Area? T: Action Taken with Study Drug E: Action Taken to Treat Event |
|---|---|---|---|---|
| S: xxxxxx | A: xxxxxxxxxxxx | F: xxxxxxxxx | G: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxx | S: xxxxxxxxx xxxx | R: xxxxxxxxx | A: xxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx xxxx | O: xxxxxxxxx | T: xxx |
| | | | | E: xxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxxxxxxx | G: xxxx | S: xx |
| A: XXXX | C: xxxxxxxxxxxxxx | S: xxxxxxxxx xxxx | R: xxxxxxxxxx | A: xxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx xxxx | O: xxxxxxxxx | T: xxx |
| | | | | E: xxxxxx |
| : xxxxxx | A: xxxxxxxxxxxxx | F: xxxxxxxxx | G: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxxxxxxx xxxx | R: xxxxxxxxxx | A: xx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx xxxx | O: xxxxxxxxx | T: xxx |
| | | | | E: xxxxxxx |

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.
Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.7.2.3: Serious Adverse Events Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | F: Date of First Dose S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> | G: Grade <sup>2</sup> R: Relationship to Study Drug O: Outcome | S: Serious Evemt? A: In Treatment Area? T: Action Taken with Study Drug E: Action Taken to Treat Event |
|---|---|---|---|---|
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxxxxxxx | G: xxxx | S: xxx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxxxxxxx xxxx | R: xxxxxxxxxx | A: xxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx xxxx | O: xxxxxxxxx | T: xxx |
| | | | | E: xxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxxxxxxx | G: xxxx | S: xxx |
| A: XXXX | C: xxxxxxxxxxxxxx | S: xxxxxxxxx xxxx | R: xxxxxxxxxx | A: xxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx xxxx | O: xxxxxxxxx | T: xxx |
| | | | | E: xxxxxx |
| : xxxxxx | A: xxxxxxxxxxxxx | F: xxxxxxxxx | G: xxxx | S: xxx |
| A: XXXX | C: xxxxxxxxxxxxxx | S: xxxxxxxxx xxxx | R: xxxxxxxxxx | A: xx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx xxxx | O: xxxxxxxxx | T: xxx |
| | | | | E: xxxxxxx |

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.
Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.7.2.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events Treatment Group (Page xx of yy)

| S: Subject | R: Pr | rimary Reason for Study | | | A | dverse Events | | |
|---|---|---|---|---|---|---|---|---|
| A: Age/Sex | Co | ompletion/Discontinuation | | | G: | Grade <sup>2</sup> | | |
| E: Eval | S: Da | ate of Study | A: | Adverse Event Description | R: | Relationship to | | |
| F: Date of First Do | se Co | ompletion/Discontinuation ( | Day) 1 C: | System Organ Class | | Study Drug | S: | Start Date (Day) 1 |
| L: Date of Last Dos | e V: La | ast Visit Attended | P: | Preferred Term | A: | Action Taken | E: | End Date (Day) 1 |
| S: xxxxx | R: xx | XXXXX XXXX | A: | xxxxxxx xxx | G: | xxxxx x | s: | xxxxxxxxx xxxx |
| A: xxxx | S: xx | XXXXXXXX XXXX | C: | XXXXXXXX XXXX | R: | XXXXXXXX | E: | XXXXXXXXX XXXX |
| E: xxxxxxxx | V: xx | XXX X | P: | XXXXXXXX XXXXXXX XXXX | A: | XXXXXXX XXXXXXXX | | |
| F: xxxxxxxxx | | | | XXXXXXXX | | XXXXXX | | |
| L: xxxxxxxxxx | | | | | | | | |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death. Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.8.1: Urine Pregnancy Test Results Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date | Result |
|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXX | XXXXXXXX | XXXXXXXXX | XXXXXXX |
| | | | XXXXXXX | XXXXXXXXX | XXXXXXX |
| | | | XXXX X | XXXXXXXXX | XXXXXXX |
| | | | XXXX X | XXXXXXXXX | XXXXXXX |
| | | | XXXX XX | XXXXXXXXX | XXXXXXX |
| XXXXXX | XXXX | XXXXXXX | xxxxxxxx | xxxxxxxxx | XXXXXXX |
| | | | xxxxxxxx | XXXXXXXXX | XXXXXXX |
| | | | XXXX X | xxxxxxxxx | XXXXXXX |
| | | | XXXX X | xxxxxxxxx | XXXXXXX |
| | | | XXXX X | xxxxxxxxx | XXXXXXX |
| | | | xxxx xx | xxxxxxxxx | XXXXXXX |
| XXXXXX | xxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | XXXXXXX |
| | | | XXXXXXXX | xxxxxxxxx | XXXXXXX |
| | | | xxxx x | xxxxxxxxx | XXXXXXX |
| | | | xxxx x | xxxxxxxxx | xxxxxxx |
| | | | XXXXXXXX XX | xxxxxxxxx | XXXXXXX |
| | | | XXXX XX | xxxxxxxxx | XXXXXXX |
| | | | 1111111 1111 | 111111111111111111111111111111111111111 | *************************************** |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Date.



# Listing 16.2.8.2.1: Laboratory Test Results Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex | <pre>V: Visit D: Date/Time</pre> | | Results | Refere | ence Range |
|---|---|---|---|---|---|
| E: Eval | C: Category | Laboratory Test | (Units) | Normal Range | Indicator (CS1) |
| S: xxxxxx<br>A: xxxx<br>S: xxxxxxxx | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:<br>C: xxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx (xx) | x to xx | xxxxxx xxxx |
| | | xxxxxxxxxxxxxxxx | xx (x) | xx to xx<br>xx to xx | xxxxxx xxxx<br>xxxxxx xxxx |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx (xx)<br>xx xx (xx) | xx to xx<br>xx to xx<br>xxxxx xxxx xxxx | XXXXXX XXXX<br>XXXXXX XXXX |
| | | xxxxxxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxx xxxxx |
| | | xxxxxxxxxxxxxx | xx (xx) | x to xx | xxxxxx xxxx |

Listing sorted by Subject, Visit, Date/Time, Category, and Lab Test.

¹ Clinically Significant per Investigator.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.8.2.2: Abnormal Laboratory Results Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex | V: Visit D: Date/Time | | Results | Refere | ence Range |
|---|---|---|---|---|---|
| : Eval | C: Category | Laboratory Test | (Units) | Normal Range | Indicator (CS1) |
| : xxxxx<br>: xxxx | V: xxxxxxxxx<br>D: xxxx-xx-xxTxx:xx | xxxxxxxxxxxxxx | xx (xx) | x to xx | xxxxxx xxxx |
| : xxxxxxxxx | C: xxxxxxxxx | | | | |
| | | xxxxxxxxxxxxxx | xx (x) | xx to xx | XXXXXX XXXX |
| | | xxxxxxxxxxxxxx | xx (x) | xx to xx | xxxxxx xxxx |
| | | xxxxxxxxxxxxxx | xx (xx) | xx to xx | xxxxxx xxxx |
| | | xxxxxxxxxxxxxx | xx xx (xx) | xx to xx | XXXXXX XXXX |
| | | xxxxxxxxxxxxxx | XXX XXXXXX | XXXXX XXXX XXXX | XXXXXX XXXX |
| | | xxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxx xxxxx |
| | | ****** | xx (xx) | x to xx | |

Listing sorted by Subject, Visit, Date/Time, Category, and Lab Test.

¹ Clinically Significant per Investigator.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



#### Listing 16.2.8.3: 12-lead Electrocardiogram Test Results Treatment Group (Page x of xx)

| Subject | Age/Sex | Eval | V: Visit D: Date/Time of ECG | Category | Evaluator | ECG Parameter | Result (Units) |
|---|---|---|---|---|---|---|---|
| | | | | | | | · · · |
| xxxxxxx | xxxx | xxxxxxxx | V: xxxxxxxx | xxxxxxxxx | xxxxxxxxxxx | xxxxxxxxx | xxxx xxxxx xx |
| 2121212121212121 | 21212121 | 71717171717171 | D: xxxx-xx-xxTxx:xx | 217171717171717171 | XXXXXXXXXXXX | XXXXXXXXXX | XXXX XXXXX XX |
| | | | D. MANA AN ANIAM. | | *************************************** | XXXXXXXXXX | XXXX XXXXX XX |
| | | | | | | XXXXXXXXXX | XXXX XXXXX XX |
| | | | | | | XXXXXXXXX | XXXX XXXXX XX |
| | | | | | | XXXXXXXXX | XXXX XXXXX XX |
| | | | | | | XXXXXXXXX | XXXX XXXXX XX |
| | | | | | | xxxxxxxxx | xxxx xxxxx xx |
| XXXXXXX | XXXX | xxxxxxx | V: xxxxxxxx | xxxxxxxxx | XXXXXXXXXXX | XXXXXXXXX | xxxx xxxxx xx |
| | | | D: xxxx-xx-xxTxx:xx | | XXXXXXXXXX | XXXXXXXXX | xxxx xxxxx xx |
| | | | | | | XXXXXXXXX | xxxx xxxxx xx |
| | | | | | | XXXXXXXXX | xxxx xxxxx xx |
| | | | | | | XXXXXXXXX | xxxx xxxxx xx |
| | | | | | | XXXXXXXXX | xxxx xxxxx xx |
| | | | | | | XXXXXXXXX | xxxx xxxxx xx |
| | | | | | | xxxxxxxxx | xxxx xxxxx xx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date/Time, Category, and ECG Parameter.



# Listing 16.2.8.4: Vital Signs Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date | Vital Sign | Result | Units |
|---|---|---|---|---|---|---|---|
| XXXXX | xxxx | xxxxxxx | SCREENING | xxxxxxxxx | Temperature | xxxx | Х |
| | | | | | Heart Rate | XX | xxxxxxxx |
| | | | | | Systolic Blood Pressure | XXX | xxxx |
| | | | | | Diastolic Blood Pressure | XX | XXXX |
| | | | BASELINE | xxxxxxxxx | Temperature | xxxx | X |
| | | | | | Heart Rate | XX | xxxxxxxx |
| | | | | | Systolic Blood Pressure | XXX | xxxx |
| | | | | | Diastolic Blood Pressure | XX | xxxx |
| | | | | | Height | XX | xx |
| | | | | | Weight | XXX | XX |
| | | | xxxx x | xxxxxxxxx | Temperature | xxxx | Х |
| | | | | | Heart Rate | XX | xxxxxxxx |
| | | | | | Systolic Blood Pressure | XXX | XXXX |
| | | | | | Diastolic Blood Pressure | XX | XXXX |
| | | | | | Weight | XXX | XX |
| | | | xxxx x | xxxxxxxxx | Temperature | xxxx | Х |
| | | | | | Heart Rate | XX | xxxxxxxx |
| | | | | | Systolic Blood Pressure | XXX | XXXX |
| | | | | | Diastolic Blood Pressure | XX | XXXX |
| | | | | | Weight | XXX | XX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, and Vital Sign (in the order displayed in the CRF).



# Listing 16.2.8.5: Pharmacokinetics Blood Sample Collections Treatment Group (Page x of xx)

Date/Time S: Subject A: Age/Sex of Pre-Dose Percent BSA Additional PK Date/Time PK E: Eval Visit Being Treated Sample Collections 1 Sample Obtained PK Sample S: xxxxxx XXXXXXXXX xxxx-xx-xxTxx:xx:xx XX.X% 72-Hour PK Sample xxxx-xx-xxTxx:xx:xx A: xxxx E: xxxxx 120-Hour PK Sample xxxx-xx-xxTxx:xx:xx 168-Hour PK Sample xxxx-xx-xxTxx:xx:xx 216-Hour PK Sample xxxx-xx-xxTxx:xx:xx S: xxxxxx xxxx-xx-xxTxx:xx:xx XX.X% XXXXXXXXX A: xxxx E: xxxxx 72-Hour PK Sample xxxx-xx-xxTxx:xx:xx S: xxxxxx XXXXXXXXX xxxx-xx-xxTxx:xx:xx XX.X% A: xxxx E: xxxxx 120-Hour PK Sample xxxx-xx-xxTxx:xx:xx 168-Hour PK Sample xxxx-xx-xxTxx:xx:xx 216-Hour PK Sample xxxx-xx-xxTxx:xx:xx

Listing sorted by Subject, Visit, Date/Time of Pre-Dose PK Sample, and Date/Time PK Sample Obtained.

<sup>1</sup> Additional PK samples are collected on a conditional basis, date and time the PK sample was obtained is included in the listing. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Arcutis ARQ-151-201

Version: 2

Date: 11 JUN 2019
STATISTICAL ANALYSIS PLAN

Protocol Number: ARQ-151-201

Study Title: A Phase 2b 12-Week Parallel Group, Double Blind,

Vehicle-Controlled Study of the Safety, Efficacy, and Pharmacokinetics of ARQ-151 Cream 0.3% and ARQ-151 Cream 0.15% Administered QD in

Subjects with Chronic Plaque Psoriasis

Development Phase of Study: Phase 2b

Sponsor: Arcutis, Inc.

2945 Townsgate Road, Suite 110 Westlake Village, CA 91361

Sponsor Contact: David Berk, MD

Vice President, Clinical Development

Statistical Analysis Plan based on

Protocol Version:

Amendment 1, 12 November 2018

Statistical Analysis Plan Date: 11JUN2019 Statistical Analysis Plan Version: Version 2



Arcutis ARQ-151-201 Version: 2

Date: 11 JUN 2019

## Authored by:

| SIGNATURE: Associate Statistical Programmer QST Consultations, Ltd. | DATE: _/2 <i>JUN 2019</i> |
|---|---|
| Reviewed by: | |
| SIGNATURE: Director of Biostatistical Consulting QST Consultations, Ltd. | DATE: 19 Jun 2019 |
| Approved by: | |
| SIGNATURE: David Serk (Jun 11, 2019) David Berk, MD Vice President, Clinical Development Arcutis, Inc. | Jun 11, 2019 DATE: |

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.



# Statistical Analysis Plan Arcutis ARQ-151-201

Arcutis ARQ-151-201 Version: 2 Date: 11 JUN 2019

# SAP Change History

Only final versions will be documented in the Change History.

| Version | Date | Summary of Changes | Author |
|---------|-----------|---------------------------------|--------|
| 1 | 24MAY2019 | Original document | |
| 2 | 11JUN2019 | Added PASI to efficacy analysis | |



# **Statistical Analysis Plan** Arcutis ARQ-151-201


Date: 11 JUN 2019

# **TABLE OF CONTENTS**

| 1. | LIS | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS6 | | |
|---|---|---|---|---|
| 2. | INT | RODU | CTION | 7 |
| 3. | | | JECTIVES | |
| J. | | | | |
| 4. | STUDY DESIGN | | | |
| | 4.1 | Overall | l Study Design | |
| | | 4.1.1 | Schedule of Visits and Assessments | |
| | | 4.1.2 | Method of Assigning Subjects to Treatment Groups | |
| | | 4.1.3 | Blinding | 9 |
| 5. | EFI | FICACY | AND SAFETY ENDPOINTS | 9 |
| | 5.1 | Efficac | y Endpoints | 9 |
| | | 5.1.1 | Primary Efficacy Endpoint | 10 |
| | | 5.1.2 | Secondary Efficacy Endpoints | 10 |
| | | 5.1.3 | Additional Efficacy Endpoints | 11 |
| | 5.2 | Safety | Endpoints | 12 |
| 6. | STA | ATISTIC | CAL AND ANALYTICAL PLANS | 12 |
| | 6.1 | Genera | l Methodology | 12 |
| | | 6.1.1 | Statistical Analysis | 13 |
| | | 6.1.2 | Baseline Definition | 13 |
| | | 6.1.3 | Visit Windowing | 13 |
| | | 6.1.4 | Adjustments for Covariates | 14 |
| | | 6.1.5 | Handling of Dropouts or Missing Data | 14 |
| | | 6.1.6 | Interim Analyses and Data Monitoring | 14 |
| | | 6.1.7 | Multicenter Studies | 14 |
| | | 6.1.8 | Multiple Comparisons/Multiplicity | 14 |
| | | 6.1.9 | Use of an Efficacy Subset of Subjects | 15 |
| | | 6.1.10 | Active-Control Studies Intended to Show Equivalence | 15 |
| | | 6.1.11 | Examination of Subgroups | 15 |
| | 6.2 | 2 Disposition of Subjects | | |
| | 6.3 | Protoco | ol Deviations | 15 |
| | 6.4 | Data Sets Analyzed | | |
| | | | Intent-to-Treat Population | |



# Statistical Analysis Plan Arcutis ARQ-151-201


Date: 11 JUN 2019

| | | 6.4.2 | Safety Po | pulation | 16 |
|---|---|---|---|---|---|
| | | 6.4.3 | Per-Proto | ocol Population | 16 |
| | | 6.4.4 | Pharmaco | okinetic Population | 16 |
| | 6.5 | Demog | graphic and | Other Baseline Characteristics | 17 |
| | 6.6 | Analys | sis of Effica | ncy | 17 |
| | | 6.6.1 | Primary I | Efficacy Analysis | 17 |
| | | 6.6.2 | Secondar | y Efficacy Analysis | 17 |
| | | 6.6.3 | Explorato | ory Efficacy Analysis | 19 |
| | 6.7 | Safety | Evaluation | | 19 |
| | | 6.7.1 | Extent of | Exposure | 19 |
| | | 6.7.2 | Adverse l | Events | 20 |
| | | 6.7.3 | Clinical I | Laboratory Evaluation | 20 |
| | | 6.7.4 | Other Ob | servations Related to Safety | 21 |
| | | | 6.7.4.1 | Electrocardiogram Measurements | 21 |
| | | | 6.7.4.2 | Vital Signs | |
| | | | 6.7.4.3 | Physical Examination | 21 |
| | | | 6.7.4.4 | Medical History | 21 |
| | | | 6.7.4.5 | Local Tolerance Assessments | 21 |
| | | | 6.7.4.6 | Patient Health Questionnaire Depression Scale | |
| | | | 6.7.4.7 | Columbia-Suicide Severity Rating Scale | 22 |
| | | | 6.7.4.8 | Prior and Concomitant Medications | |
| | 6.8 | Other | Evaluations | 3 | 22 |
| | | 6.8.1 | Pharmaco | okinetic Evaluation | 22 |
| 7. | DE | ΓERMI | NATION ( | OF SAMPLE SIZE | 22 |
| 8. | CH | ANGES | S IN THE I | PLANNED ANALYSES | 22 |
| 9. | REFERENCES | | | | |
| 10. | IND | EX OF | PLANNE | D TABLES | 24 |
| 11. | IND | EX OF | F PLANNE | D LISTINGS | 172 |



Arcutis ARQ-151-201


Date: 11 JUN 2019

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE(s) Adverse Event(s)
BSA Body Surface Area
CRF(s) Case Report Form(s)

C-SSRS Columbia-Suicide Severity Rating Scale

DLQI Dermatology Life Quality Index

ECG Electrocardiogram

IGA Investigator's Global Assessment

I-IGA Intertriginous IGA ITT Intent-to-Treat

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities mPASI Modified Psoriasis Area and Severity Index

N Sample Size

NRS Numerical Rating Score

PASI Psoriasis Area and Severity Index

PHQ-8 Patient Health Questionnaire Depression Scale

PK Pharmacokinetic
PP Per-Protocol

PSD Patient Symptoms Diary

QD Once a Day

SAE(s) Serious Adverse Event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

SD Standard Deviation

TEAE(s) Treatment-Emergent Adverse Event(s)

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

World Health Organization-Anatomical Therapeutic Chemical

WHO-ATC Classification System

WI-NRS Worst Itch Numerical Rating Scale

WPAI Work Productivity and Activity Impairment




#### 2. INTRODUCTION

Roflumilast is a phosphodiesterase 4 (PDE-4) inhibitor approved globally to reduce the risk of exacerbations in patients with severe chronic obstructive pulmonary disease (COPD) associated with chronic bronchitis. Roflumilast and its active metabolite, roflumilast N-oxide, are high affinity selective inhibitors of PDE-4 (a major cyclic-3′,5′-adenosine monophosphate (cyclic AMP)-metabolizing enzyme), whose activity leads to accumulation of intracellular cyclic AMP. There are four different subtypes of PDE-4: PDE-4a, PDE-4b, PDE-4c, and PDE-4d, each with several isoforms (splicing variants). IC50 values of both roflumilast and roflumilast N-oxide for the different PDE-4 isoforms and subtypes are mostly sub-nanomolar and single digit nanomolar (Hatzelmann 2010). The PDE-4 family of enzymes are the most prevalent phosphodiesterases in immune cells and inhibition of PDE-4 subtypes has been associated with anti-inflammatory effects in many biological systems.

Psoriasis is a chronic inflammatory skin disease characterized by raised, well-demarcated, erythematous oval plaques with adherent silvery scales. Numerous past reports have suggested a deficiency of cyclic AMP-dependent protein kinases in human psoriatic skin (Brion 1986). More recently, various cytokines produced by Th1 and Th17 cells have been shown to play a crucial role in the pathogenesis of psoriasis. It has been postulated that the anti-inflammatory effects of PDE-4 inhibitors may provide a beneficial therapeutic intervention in the treatment of chronic plaque psoriasis, and recently Otezla® (apremilast) a PDE-4 inhibitor has been approved for the oral treatment of chronic plaque psoriasis.

The past 15 years have witnessed a transformation in the systemic treatment of moderate to severe psoriasis with the advent of biological therapies. However, for patients with milder forms of disease, best treated with topical options, the therapeutic landscape really has not changed in several decades. Topical steroids come in all shapes and forms, but the lower potency steroids are not effective and the higher potency steroids are beset with issues of local skin atrophy and the potential for hypothalamic-pituitary axis suppression when applied over larger body surface areas and for prolonged periods of time. Vitamin D has been the other staple of topical psoriasis treatment but it is irritating, not suitable for use on the face or intertriginous areas, and its efficacy is rather modest. Hence, there is substantial medical need for additional topical approaches in the treatment of psoriasis. Arcutis, Inc is developing a topical formulation of roflumilast for the treatment of chronic plaque psoriasis.




#### 3. STUDY OBJECTIVES

To assess the safety, pharmacokinetics and efficacy of ARQ-151 cream 0.3% and ARQ-151 cream 0.15% vs. vehicle applied QD for 12 weeks to individuals treated with 2 to 20% (inclusive) Body Surface Area (BSA) of chronic plaque psoriasis.

### 4. STUDY DESIGN

### 4.1 Overall Study Design

This is a parallel group, double blind, vehicle-controlled study in which ARQ-151 cream 0.3%, ARQ-151 cream 0.15% or vehicle cream QD is applied for 84 days to subjects with between 2% to 20% (inclusive) BSA of chronic plaque psoriasis.

A total of up to approximately 300 subjects will be enrolled at approximately 30 study sites in the United States and Canada. Subjects will be adult (≥18 y/o) males or females with chronic plaque psoriasis. Subjects must have an Investigator's Global Assessment (IGA) of disease severity of at least Mild ('2') at Baseline. Subjects with an IGA of 'Mild' (2) will be limited to 20% of total enrollment. Subjects with an IGA of 'Severe' (4) will be limited to 15% of total enrollment. Subjects must have at least 2% and no more than 20% BSA of chronic plaque psoriasis. All psoriasis lesions on a subject will be treated including the face, trunk, genitals/skin folds, or limbs (excluding the scalp). The palms and soles will be treated but will not be counted towards any measurements of efficacy (IGA, BSA, Psoriasis Area and Severity Index (PASI), Modified PASI (mPASI)). For subjects with intertriginous area involvement, and with severity of the intertriginous area lesions at least 'mild' (IGA≥2) at Baseline, Intertriginous IGA (I-IGA) score will be recorded at weeks 4, 6, 8 and 12. The same IGA used for the primary endpoint (whole body) will also be used for I-IGA, but only intertriginous areas will be evaluated for I-IGA, not the rest of the body.

#### 4.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 5 of the protocol.

### 4.1.2 Method of Assigning Subjects to Treatment Groups

Assignment of drug or vehicle will be made at a 1:1:1 ratio according to a computer-generated randomization list. Randomization will take place at Baseline after the patient has been found to be fully eligible for participation. Kits containing tubes of study medication will be assigned to each subject using an internet-based randomization system (IWRS). A subject may receive more than one kit for the treatment period.




The kits and tubes are blinded and each kit is numbered with a unique kit number.

### 4.1.3 Blinding

This is a double-blind study, therefore neither the subjects nor the Investigator, clinical team, and study sponsor will be aware of which treatment an individual has received.

If the situation requires emergency unblinding this will be done by investigator using the study IWRS system after discussion with Medical Monitor and the Sponsor's CMO.

The treatment assignments for all enrolled subjects will be unblinded only after the conclusion of the study. Specifically, the blind will be broken only after all data are verified, entered into the database, and validated; subject evaluability assessments are performed and entered into the database; and the database is locked.

#### 5. EFFICACY AND SAFETY ENDPOINTS

## 5.1 Efficacy Endpoints

PASI is one of the measurements used for the severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). The body is divided into four sections (head (h) (10% of a person's skin); arms (a) (20%); trunk (t) (30%); legs (l) (40%)). Each of these areas is scored by itself, and then the four scores are combined into the final PASI. For each section, the percent of area (A) of skin involved is estimated and then transformed into a grade from 0 to 6 (A):

- 0.0% of involved area
- 1. < 10% of involved area
- 2. 10–29% of involved area
- 3. 30-49% of involved area
- 4. 50-69% of involved area
- 5. 70-89% of involved area
- 6. 90-100% of involved area

Within each area, the severity is estimated by three clinical signs: erythema ('E'; redness), induration ('T'; thickness) and desquamation ('S'; scaling). Severity parameters are measured on a scale of 0 to 4, from none to maximum severity possible.

To calculate the PASI, the sum of the severity rating for the three main signs are multiplied with the numerical value of the area affected and with the various percentages of the four body areas. These values are then added to complete the formula as follows:




In addition to PASI, an mPASI will also be used for the severity of psoriasis. The mPASI will be calculated the same as the PASI except for subjects with < 10% of an involved anatomical area. For subjects with < 10% of an involved anatomical area the mPASI will be calculated using the actual percentage of the anatomical area involved (e.g. 0.1 for 1%, 0.2 for 2%, 0.3 for 3%, ... 0.9 for 9%), corresponding to the actual percentage of that particular anatomical area of involvement. The resulting values will then be rounded to the nearest tenth prior to analysis.

### 5.1.1 Primary Efficacy Endpoint

The primary efficacy endpoint is as follows:

• Success in Investigator Global Assessment (IGA) of disease severity, defined as an IGA of 'Clear' or 'Almost Clear' at Week 6.

### **5.1.2** Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- IGA score of 'clear' or 'almost clear' at weeks 2, 4, 8, and 12.
- Percent change from Baseline in PASI at weeks 2, 4, 6, 8, and 12.
- Percent change from Baseline in mPASI at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Percent BSA affected at weeks 2, 4, 6, 8, and 12.
- IGA score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline at weeks 2, 4, 6, 8 and 12.
- For subjects with intertriginous area involvement, and with severity of the intertriginous lesions at least 'mild' (I-IGA≥2) at Baseline, 'I-IGA' score of 'clear' or 'almost clear' at weeks 2, 4, 6, 8 and 12.
- Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) pruritus score at weeks 2, 4, 6, 8, and 12.
- In subjects with WI-NRS pruritus score ≥ 6 at Baseline, a 4-point reduction in WI-NRS pruritus score at 2, 4, 6, 8, and 12 weeks as compared to Baseline.




- Change from Baseline in Psoriasis Area Severity Index-75 (PASI-75) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Psoriasis Area Severity Index-90 (PASI-90) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Psoriasis Area Severity Index-100 (PASI-100) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-75 (mPASI-75) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-90 (mPASI-90) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-100 (mPASI-100) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Total Patient Symptoms Diary (PSD) at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Itch-related Sleep Loss score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Dermatology Life Quality Index (DLQI) score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in responses to the questions of Total Patient Symptom Diary (PSD) at weeks 2, 4, 6, 8, and 12.

Change from Baseline will be calculated by subtracting the score at Baseline from the post-baseline score. Percent change from Baseline will be calculated by dividing change from Baseline by the Baseline score, multiplied by 100.

### **5.1.3** Additional Efficacy Endpoints

The exploratory endpoints are as follows:

- Change from Baseline in Fatigue Numerical Rating Score (NRS) score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Work Productivity and Activity Impairment (WPAI) score at weeks 2, 4, 6, 8, and 12.




Change from Baseline will be calculating by subtracting the score at Baseline from the post-baseline score.

### 5.2 Safety Endpoints

Safety will be evaluated through examination of data collected during physical examinations, 12-lead Electrocardiograms (ECGs), local tolerability assessments, vital signs, counts and percentages of subjects who gain or lose >5% and >10% body weight, clinical laboratory parameters, Patient Health Questionnaire Depression Scale (PHQ-8), Columbia-Suicide Severity Rating Scale (C-SSRS) and adverse events (AEs) as outlined in the Schedule of Visits and Assessments. If deemed necessary, additional safety assessments will be performed at the discretion of the Principal Investigator.

#### 6. STATISTICAL AND ANALYTICAL PLANS

## 6.1 General Methodology

All statistical processing will be performed using SAS® (Version 9.4 or later) unless otherwise stated. No interim analyses are planned. Except where noted, all statistical tests will be two-sided and will be performed at the 0.05 level of significance. No adjustment will be made for multiplicity.

Descriptive statistics will be used to provide an overview of the efficacy, safety, and pharmacokinetic results. For categorical parameters, the number and percentage of subjects in each category will be presented. The denominator for percentage will be based on the number of subjects appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include n (number of subjects), mean, standard deviation (SD), median, minimum and maximum. Appropriate inferential statistics will be used for the primary, secondary, and exploratory efficacy variables.

The primary method of handling missing efficacy data will be a mixture of linear interpolation and last observation carried forward (LOCF).

The efficacy analysis performed on the Intent-to-Treat (ITT) population is considered the primary analysis. The efficacy analysis performed on the Per-Protocol (PP) population is considered supportive analysis.

The number of subjects in each analysis set will be summarized. Reasons for study withdrawal during the blinded study will be summarized using frequencies and percentages by treatment group. Reported AEs, medical history terms and prior and concomitant procedures and therapies will be classified on the basis of Medical Dictionary for Regulatory Activities (MedDRA)




Date: 11 JUN 2019

terminology. Prior and concomitant medications will be classified on the basis of World Health Organization Drug Dictionary (WHO-DD) terminology.

## 6.1.1 Statistical Analysis

All analyses will be performed by QST using SAS® Version 9.4 or later. All summary tables and data listings will be prepared utilizing SAS® software.

The standard operating procedures (SOPs) of QST will be followed in the creation and quality control of all data displays and analyses.

#### **6.1.2** Baseline Definition

Baseline is defined as the last non-missing assessment prior to first dose of study drug.

## 6.1.3 Visit Windowing

Data will be summarized based on nominal visit indications with the exception of data captured at early termination and unscheduled visits. Data from early termination and unscheduled visits will be summarized based on mapped visit values. The analysis windows for early termination and unscheduled visits are presented in the following table.

**Analysis Windows for Efficacy and Safety Assessments** 

| Scheduled Visit | Target Study Day | Window (Days) |
|-----------------|------------------|---------------|
| Week 2 | 15 | 8 to 22 |
| Week 4 | 29 | 23 to 36 |
| Week 6 | 43 | 37 to 50 |
| Week 8 | 57 | 51 to 71 |
| Week 12 | 85 | 72 to 99 |
| Week 16 | 113 | 100 to 127 |

Data collected at early termination and unscheduled visits prior to study day 8 will not be analyzed, with the exception of those identified as baseline values. Data collected at visits after study day 127 will not be included in analyses.

The definition for the study day included in each study window is defined as below:

Study Day prior to Baseline Day 1 = Visit Date – Baseline Day 1 Date

Study Day on or after Baseline Day 1 = Visit Date - Baseline Day 1 Date + 1



If an assessment's mapped visit is a visit at which the subject has data from a scheduled visit present, or if no analyses are planned for the assessment at the mapped visit, the data collected at the early termination or unscheduled visit will not be included in analyses.

In the event of multiple values from unscheduled or early termination assessments within an analysis window, the value closest to the scheduled visit target study day will be used for analyses. If two values tie as closest to the time point (for example, one value is before and the other value is after the time point), then the later value will be selected.

Data collected at all visits will be included in the data listings with visit presented as reported by the site.

#### 6.1.4 Adjustments for Covariates

The Baseline score will be used as a covariate for each endpoint analyzed.

#### 6.1.5 Handling of Dropouts or Missing Data

The primary method of handling missing efficacy data will be a mixture of linear interpolation and LOCF. Linear interpolation will be used for all instances where subjects have observed values for at least one assessment both preceding and following the missing assessment. If an unscheduled assessment occurs between the preceding or following scheduled assessment and the missing assessment, the unscheduled assessment will be used in the linear interpolation. The actual study day of assessment will be used for the preceding and following assessments, and planned study day will be used for the missing assessment. IGA and I-IGA values imputed with linear interpolation will be rounded to the nearest integer. If the missing assessment is not followed by at least one observed assessment, the method of LOCF will be used.

## 6.1.6 Interim Analyses and Data Monitoring

No interim analysis or data monitoring is planned for this study.

#### **6.1.7** Multicenter Studies

The clinical study will be conducted under a common protocol for each investigational site. Every effort will be made to promote consistency in study execution at each investigational site. Sites will be pooled for analyses.

# 6.1.8 Multiple Comparisons/Multiplicity

No adjustments for multiple comparisons or multiplicity will be made.




Date: 11 JUN 2019

# 6.1.9 Use of an Efficacy Subset of Subjects

Subjects randomized to study drug who were at least 80% compliant with the study drug, did not miss more than three consecutive doses, and who do not have major protocol deviations will form the Per Protocol (PP) Population. The major protocol deviations will be defined at the time of evaluability evaluation, the time between the database soft lock and hard lock before unblinding.

Excluding subjects who have major protocol deviations will decrease the variability in treatment response and will allow for a better determination of efficacy of ARQ-151 Cream 0.3% and ARQ-151 Cream 0.15%.

# 6.1.10 Active-Control Studies Intended to Show Equivalence

Not applicable to this study.

### **6.1.11** Examination of Subgroups

Subset analyses will be conducted for the ITT population for the subgroups baseline IGA and baseline I-IGA. I-IGA will be dichotomized into presence or absence of I-IGA  $\geq 2$  at baseline. These analyses will contain only descriptive statistics of the primary efficacy endpoint.

#### 6.2 Disposition of Subjects

The number of subjects included in each analysis population (ITT, safety, PP, pharmacokinetic (PK)) will be summarized by treatment group. The number of subjects enrolled, completed, and discontinued (including the reasons for discontinuation) will be summarized for each treatment group.

Subjects who are excluded from an analysis population will be summarized by the primary reason for exclusion.

#### **6.3** Protocol Deviations

Protocol deviations leading to exclusion from the PP population will be tabulated. In addition to protocol deviations leading to exclusion from the PP population, the protocol deviations listed below will be presented in a data listing.

- Baseline PHQ-8 score greater than or equal to 15
- Received incorrect treatment
- •




Date: 11 JUN 2019

- Baseline IGA of Clear or Almost Clear
- Missed visit
- Missed IGA at attended visit
- Missed I-IGA at attended visit
- Missed safety labs at attended visit

# 6.4 Data Sets Analyzed

Subjects will be presented/summarized based on the primary reason for exclusion. The primary reason for exclusion for each population is the first inclusion condition a subject fails to meet based on the order listed below.

#### 6.4.1 Intent-to-Treat Population

All randomized subjects will be included in the ITT population and analyzed according to the treatment group they were randomized. All efficacy analyses will be presented using the ITT population.

#### 6.4.2 Safety Population

All subjects in the ITT population who have at least one post-baseline safety assessment will be included in the safety population and analyzed according to the treatment group they received. In the event a subject receives more than one treatment, they will be analyzed based on the treatment they received for the majority of the study. All safety analyses will be performed using the safety population.

#### 6.4.3 Per-Protocol Population

All subjects in the safety population who were at least 80% compliant with study medication, did not miss more than 3 consecutive doses, and showed no other serious protocol violations will be included in the PP population and analyzed according to the treatment group they received. All efficacy analyses will be performed on the PP population.

#### 6.4.4 Pharmacokinetic Population

All subjects receiving the active drug with quantifiable plasma concentrations of roflumilast will be included in the PK population.




Date: 11 JUN 2019

# 6.5 Demographic and Other Baseline Characteristics

All summaries will be done on the ITT, PP, safety, and PK populations.

Sex, race, and ethnicity will be summarized by counts and percentages. Age (years) will be summarized with descriptive statistics.

Height, Weight, BSA, IGA, mPASI, WI-NRS, DLQI, Itch-Related Sleep Loss, and Total PSD will be summarized at baseline with descriptive statistics.

Medical histories will be coded using the MedDRA dictionary and presented in a by-subject listing.

#### 6.6 Analysis of Efficacy

#### 6.6.1 Primary Efficacy Analysis

The primary efficacy endpoint is success in IGA, defined as an IGA of 'Clear' or 'Almost Clear' at Week 6. The primary efficacy endpoint will be analyzed with a logistic regression with a factor of treatment group and the respective Baseline IGA score as a covariate. Statistical comparison between the active treatment arms and vehicle arms will be facilitated by using contrasts.

The primary efficacy analysis will be presented on both the ITT and PP populations.

# 6.6.2 Secondary Efficacy Analysis

The secondary efficacy endpoints will include:

- IGA score of 'clear' or 'almost clear' at weeks 2, 4, 8, and 12.
- Percent change from Baseline in PASI at weeks 2, 4, 6, 8, and 12.
- Percent change from Baseline in mPASI at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Percent BSA affected at weeks 2, 4, 6, 8, and 12.
- IGA score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline at weeks 2, 4, 6, 8 and 12.
- For subjects with intertriginous area involvement, and with severity of the intertriginous lesions at least 'mild' (I-IGA\ge 2) at Baseline, 'I-IGA' score of 'clear' or 'almost clear' at weeks 2, 4, 6, 8 and 12.




- For subjects with intertriginous area involvement, and with severity of the intertriginous lesions at least 'mild' (I-IGA\ge 2) at Baseline, 'I-IGA' score of 'clear' or 'almost clear' and a 2-point improvement from Baseline at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in WI-NRS pruritus score at weeks 2, 4, 6, 8, and 12.
- In subjects with WI-NRS pruritus score ≥ 6 at baseline, a 4-point reduction in WI-NRS pruritus score at weeks 2, 4, 6, 8, and 12 as compared to Baseline.
- Change from Baseline in Psoriasis Area Severity Index-75 (PASI-75) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Psoriasis Area Severity Index-90 (PASI-90) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Psoriasis Area Severity Index-100 (PASI-100) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-75 (mPASI-75) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-90 (mPASI-90) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Modified Psoriasis Area Severity Index-100 (mPASI-100) improvement at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Total PSD at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in Itch-related Sleep Loss score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in DLQI score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in responses to the questions of PSD at weeks 2, 4, 6, 8, and 12.

Change from Baseline will be calculated by subtracting the score at Baseline from the post-baseline score. Percent change from Baseline will be calculated by dividing change from Baseline by the Baseline score, multiplied by 100.

The IGA, I-IGA, WI-NRS, PASI, and mPASI dichotomous endpoints will be analyzed with a logistic regression with a factor of treatment group and the respective Baseline score as a covariate. The remainder of the endpoints will be considered continuous and analyzed with an analysis of covariance with a factor of treatment group and the respective Baseline score as a




covariate. Statistical comparisons between the active treatment arms and vehicle arm will be facilitated by using contrasts.

The secondary efficacy analysis will be presented on both the ITT and PP populations.

# **6.6.3** Exploratory Efficacy Analysis

There are two exploratory endpoints:

- Change from Baseline in Fatigue NRS score at weeks 2, 4, 6, 8, and 12.
- Change from Baseline in WPAI score at weeks 2, 4, 6, 8, and 12.

Only descriptive statistics will be used to analyze these endpoints. Change from Baseline will be calculating by subtracting the score at Baseline from the post-baseline score.

# 6.7 Safety Evaluation

The following analyses will be performed; however, no formal inferential statistics will be done on safety assessments.

Descriptive statistics will be presented by visit and treatment group for quantitative safety data and frequency counts will be compiled for classification of qualitative safety data. Summaries of local tolerability will be presented by visit and treatment group.

#### 6.7.1 Extent of Exposure

The extent of exposure to study drug in each treatment group will be summarized by total number of days of exposure, total number of applications, total amount of study drug used, number of missed applications, and number and percentage of subjects who are compliant. A subject will be considered compliant with the dosing regimen if the subject applied at least 80% of the expected number of applications while enrolled in the study and does not miss more than 3 consecutive doses.

Days of exposure = Date of last study application - Date of first study application + 1.

The total number of applications is as follows:

(Date of Last Application – Date of First Application + 1) – (Number of Days marked as missed dose on the Case Report Form (CRF)) + (Number of Additional Doses indicated on CRF).

The expected number of applications is as follows:

Expected Date of Last Application – Date of Randomization + 1

TOOL.AN.10-01.01 Statistical Analysis Plan Template




Where the Expected Date of Last Application is the date of the Week 12 visit or the date of the discontinuation visit for subjects who discontinue prior to Week 12.

Compliance will be calculated as a percentage as 100 times the total number of applications divided by the expected number of applications.

#### 6.7.2 Adverse Events

All treatment-emergent AEs (TEAEs) occurring during the study will be recorded and classified on the basis of MedDRA terminology for the safety population. TEAEs are those AEs with an onset on or after the date of first study drug treatment. All AEs with incomplete onset date information will be considered treatment-emergent unless the available information indicates that this is not possible. All TEAEs will be summarized by treatment group, the number of subjects reporting TEAEs, system organ class, preferred term, severity, relationship, and seriousness. Each subject will be counted only once within a system organ class or a preferred term using the event with the greatest relationship and greatest severity.

Comparisons between treatment groups will be made by tabulating the frequency of subjects with one or more TEAEs (classified into MedDRA terms) during the study.

Serious AEs (SAEs) will be listed by subject. Treatment-emergent SAEs will be summarized by treatment group, severity, and relationship to study treatment.

All information pertaining to AEs noted during the study will be listed by subject, detailing the verbatim description given by the Investigator, preferred term, system organ class, start date, stop date, severity, action taken regarding study drug, corrective treatment, outcome, and drug relatedness. The event onset will also be shown relative (in number of days) to date of first application. In addition a listing of subjects who prematurely discontinue from the study due to AEs will also be provided.

#### 6.7.3 Clinical Laboratory Evaluation

Laboratory test results will be summarized by treatment group and visit as observed values and changes from Baseline using descriptive statistics. Additionally, shifts from Baseline to Week 4 and Week 12 in laboratory test results based on normal ranges will be summarized with frequency counts and percentages.

Individual laboratory test results, as well as abnormal laboratory results, will be presented in a by-subject listing.




Date: 11 JUN 2019

# 6.7.4 Other Observations Related to Safety

# 6.7.4.1 Electrocardiogram Measurements

Descriptive statistics of actual values and changes from baseline will be provided by treatment group and visit for the following ECG parameters: heart rate (HR), RR duration, QRS duration, PR duration, QT duration, QTc Interval, QTcB interval, QTcF interval. Investigator and cardiologist interpretation of the ECG will be summarized by counts and percentages.

Individual ECG parameters, as well as interpretations, will be presented in a by-subject listing.

#### 6.7.4.2 Vital Signs

Descriptive statistics of actual values and changes from baseline will be provided by treatment group and visit for the following parameters: temperature, systolic blood pressure, diastolic blood pressure, heart rate, and weight. Additionally, counts and percentages of subjects who gain or lose > 5% body weight will be summarized by visit in a table.

### 6.7.4.3 Physical Examination

Abnormal physical examination findings will recorded as AEs and included in the AE summaries.

# 6.7.4.4 Medical History

Medical history for all subjects will be presented in a by-subject listing.

#### **6.7.4.5** Local Tolerance Assessments

For the investigator's assessment and subject local tolerability assessment of sensation following drug application, the numeric application site reaction scores will be summarized individually by using number and percentage of subjects by visit. In addition, a by-subject listing of investigator and subject assessments will be provided.

#### 6.7.4.6 Patient Health Questionnaire Depression Scale

The PHQ-8 will be analyzed by a shift in state of severity using the following scoring system:

- None Minimal depression (0 to 4)
- Mild depression (5 to 9)
- Moderate depression (10 to 14)

TOOL.AN.10-01.01 Statistical Analysis Plan Template




Date: 11 JUN 2019

- Moderately severe depression (15 to 19)
- Severe depression (20 to 24)

In addition, a by-subject listing of results will be provided.

#### 6.7.4.7 Columbia-Suicide Severity Rating Scale

The C-SSRS will be analyzed per the C-SSRS Scoring and Data Analysis Guide (Nilsson 2013).

#### 6.7.4.8 Prior and Concomitant Medications

Prior and concomitant medication information for all randomized subjects will be presented in a by-subject listing. Summary tables will be presented by World Health Organization-Anatomical Therapeutic Chemical Classification System (WHO-ATC) therapeutic category and product.

#### 6.8 Other Evaluations

#### **6.8.1** Pharmacokinetic Evaluation

Plasma drug concentrations at pre-dose will be summarized using descriptive statistics, reporting n, mean, standard deviation, median, minimum, and maximum.

#### 7. DETERMINATION OF SAMPLE SIZE

The sample size was not powered based on data for the primary endpoint to provide statistical significance because of the absence of previous primary endpoint data. However, based on efficacy data from the Phase 1/2a study, this Phase 2b study is expected to provide reliable information regarding the efficacy and safety of the drug products.

#### 8. CHANGES IN THE PLANNED ANALYSES

The Per-Protocol population was updated to exclude subjects with more than three consecutive missed doses in order to fully capture compliant subjects.

A covariate of the respective Baseline score was added to the models used for analysis of the primary and secondary endpoints.

A secondary efficacy analysis endpoint of 'clear' or 'almost clear' plus a 2-point improvement from Baseline for Intertriginous Investigator Global Assessment (I-IGA) at weeks 2, 4, 6, 8, and 12 was added.

A secondary efficacy analysis endpoint for change from Baseline in Modified Psoriasis Area Severity Index-100 (mPASI-100) at weeks 2, 4, 6, 8, and 12 was added.

TOOL.AN.10-01.01 Statistical Analysis Plan Template




Week 2 was added to all secondary and exploratory efficacy endpoints.

An analysis of PASI was added for all planned mPASI analyses.

#### 9. REFERENCES

Brion DE, Raynaud F, Plet A, Laurent P, Leduc B, and Anderson W. Deficiency of cyclic AMP-dependent protein kinases in human psoriasis. Proc. Natl. Acad. Sci. 1986; 83:5272-5276.

Hatzelmann A, Morcillo EJ, Lungarella G, Adnot S, Sanjar S, Beume R, et al. The preclinical pharmacology of roflumilast – a selective, oral phosphodiesterase 4 inhibitor in development for chronic obstructive pulmonary disease. Pulm Pharmacol Ther. 2010; 23:235–256.

Nilsson M, Suryawanshi S, Gassmann-Mayer C, Dubrava S, McSorley P, and Jiang K. Columbia–Suicide Severity Rating Scale Scoring and Data Analysis Guide. Version 2. 2013




Date: 11 JUN 2019

# 10. INDEX OF PLANNED TABLES

| Table 14.0.2: Summary of Subject Completion/Discontinuation (Randomized Subjects) |
|---|
| Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population) |
| Table 14.1.1.3: Summary of Subject Demographics (Safety Population) |
| Table 14.1.1.4: Summary of Subject Demographics (PK Population) |
| Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population) |
| Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population) |
| Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population) |
| Table 14.1.2.4: Summary of Subject Baseline Characteristics (PK Population) |
| Table 14.1.3: Summary of Medical History by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Term (Safety Population) |
| Name (Safety Population) |
| Table 14.1.4.2: Summary of Concomitant Medications by WHO-DD ATC Level 2 Term and |
| Preferred Name (Safety Population) |
| Table 14.2.1.1: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Intent-to-Treat Population) |
| Table 14.2.1.2: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Per-Protocol Population) |
| Figure 14.2.1.1: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Intent-to-Treat Population) |
| Figure 14.2.1.2: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Per-Protocol Population) |
| Table 14.2.2.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population) |
| Table 14.2.2.2: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Per-Protocol Population) |
| Table 14.2.3.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline (Intent-to-Treat Population) |







| Figure 14.2.4.2.2: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline) |
|---|
| Table 14.2.5.1.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI) (Intent-to-Treat Population) |
| Table 14.2.5.1.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI) (Per-Protocol Population) |
| Figure 14.2.5.1.1: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI) (Intent-to-Treat Population) |
| Table 14.2.5.2.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Intent-to-Treat Population) |
| Table 14.2.5.2.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Per-Protocol Population) |
| Figure 14.2.5.2.1: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Intent-to-Treat Population) |
| Table 14.2.6.1.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.6.1.2 Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Per-Protocol Population)70 |
| Table 14.2.6.2.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.6.2.2 Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population) |
| Table 14.2.7.1.1: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.7.1.2: Dichotomized Percent Reduction(s) in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Per-Protocol Population) |
| Table 14.2.7.2.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population) |




| Table 14.2.7.2.2: Dichotomized Percent Reduction(s) in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population) |
|---|
| Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population) |
| Table 14.2.8.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Per-Protocol Population) |
| Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population) |
| Table 14.2.9.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Per-Protocol Population)90 |
| Table 14.2.10.1.1: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score $\geq 6$ at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Intent-to-Treat Population: Subjects with WI-NRS Score $\geq 6$ at Baseline)91 |
| Table 14.2.10.1.2: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score ≥ 6 at Baseline)92 |
| Table 14.2.10.2.1: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Intent-to-Treat Population: Subjects with WI-NRS Score ≥ 6 at Baseline) |
| Table 14.2.10.2.2: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score ≥ 6 at Baseline)93 |
| Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.11.2: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Per-Protocol Population) |
| Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population) |
| Table 14.2.12.2: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Per-Protocol Population) |
| Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population) |
| Table 14.2.13.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Per-Protocol Population) |
| Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)111 |



Version: 2 Date: 11 JUN 2019

| Date: 11 JON 2019 |
|---|
| Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)112 |
| Table 14.2.14.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Per-Protocol Population) |
| Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population) |
| Table 14.2.15.2: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Per-Protocol Population) |
| Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population)120 |
| Table 14.2.16.2: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Per-Protocol Population)123 |
| Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA) (Intent-to-Treat Population) |
| Table 14.2.17.2: Summary of Whole Body Investigator Global Assessment (IGA) (Per-Protocol Population) |
| Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA) (Intent-to-Treat Population) 139 Table 14.2.18.2: Summary of Intertriginous Area Investigator Global Assessment (I-IGA) |
| Table 14.3.18.2: Summary of Intertrigingus Area Invertigator Global Assessment (I-IGA) (Per-36 |
| Table 14.3.0.2.1: Summary of Pre-Dose Pharmacokinetic Concentrations (PK Population)137 |
| Table 14.3.0.2.2: Summary of Additional Pharmacokinetic Concentrations (PK Population)139 |
| Table 14.3.1.1: Summary of Local Tolerability (Safety Population)140 |
| Figure 14.3.1.1: Subject Local Tolerability Sensation Following Drug Application (Safety Population) |
| Table 14.3.1.2.1: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Injurious Behavior without Suicidal Intent Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population) |
| Table 14.3.1.2.2: Number of Patients with Suicide-Related Treatment-Emergent Events Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population) 146 |
| Table 14.3.1.3.1: Summary of PHQ-8 Assessments by Treatment Group (Safety Population)147 |
| Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population) |




| Table 14.3.1.4.1: Overall Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) |
|---|
| Table 14.3.1.4.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.4.3: Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug by MedDRA System Organ Class and Preferred Term (Safety Population)153 |
| Table 14.3.1.4.4: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population) |
| Table 14.3.1.4.5: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.4.6: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) |
| Table 14.3.1.4.7: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.4.8: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population) |
| Table 14.3.1.4.9: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results (Safety Population)160 |
| Table 14.3.1.5.1.2: Summary of Hematology Laboratory Results (Safety Population)161 |
| Table 14.3.1.5.1.3: Summary of Quantitative Urinalysis Laboratory Results (Safety Population) |
| Table 14.3.1.5.2.1: Shift Summary of Chemistry Laboratory Results (Safety Population)162 |
| Table 14.3.1.5.2.2: Shift Summary of Hematology Laboratory Results (Safety Population)162 |
| Table 14.3.1.5.2.3: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population) |
| Table 14.3.1.6.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population)163 |
| Table 14.3.1.6.2: Shift Summary of Overall Electrocardiogram (ECG) Assessments (Safety Population) |
| Table 14.3.1.7.1: Summary of Vital Signs (Safety Population) |
| Table 14.3.1.7.2: Summary of Change in Body Weight Compared to Baseline (Safety Population) |



Table 14.0.1: Summary of Subject Enrollment and Evaluability

| | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| Number of Subjects in the ITT Population | xx | XX | xx |
| Number of Subjects Included from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded in the Safety Population<br>Reason for Exclusion from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Post-Baseline Safety Assessment | xx ( xx.x%) | XX ( XX.X%) | XX ( XX.X%) |
| Number of Subjects Included from the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded in the PP Population<br>Reason for Exclusion from the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Less than 80% Compliant | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missed 3 or More Consecutive Doses | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other Serious Protocol Violations | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included from the PK Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded in the PK Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Evidence of Dosing with Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Insufficient Plasma Concentrations | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: ITT population includes all randomized subjects.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.0.2: Summary of Subject Completion/Discontinuation (Randomized Subjects)

| | ARQ-151 Cream 0.3% (N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Completed Study | , | , | , |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation | | | |
| Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost to Follow-Up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pregnancy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Protocol Deviation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Withdrawal by Subject | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Study Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Physician Decision | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lack of Efficacy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.1.1.1: Summary of Subject Demographics (Intent-to-Treat Population)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Age (years) | (IN=XX) | (IN-XX) | (IV-XX) |
| | VV | VV | VV |
| n<br>Mean | XX | XX | XX<br>XX.X |
| SD | XX.X | XX.X | |
| Median | XX.XX | XX.XX | XX.XX |
| | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| n | XX | XX | XX |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | xx ( xx.x%) | XX ( XX.X%) | xx ( xx.x%) |
| Ethnicity | | | |
| n | XX | XX | XX |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| Race | | | |
| n | XX | XX | XX |
| American Indian or Alaska Native | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Multiple/Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.1.1.1 for the following:

Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population)

Table 14.1.1.3: Summary of Subject Demographics (Safety Population)

Table 14.1.1.4: Summary of Subject Demographics (PK Population)

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Whole Body Investigator Global Assessment Score | | (IV-AX) | (1V-AA) |
| | | VV | VV |
| n<br>O Class | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Intertriginous Area Investigator Global Assessmen | t Score <sup>a</sup> | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) |
| 1 – Almost Clear | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Itch-Related Sleep Loss Score | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>a</sup> Collected for subjects with intertriginous involvement.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Body Surface Area (%) Affected by Psoriasis | <del></del> | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| PASI | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| mPASI | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| WI-NRS Score | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>a</sup> Collected for subjects with intertriginous involvement.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.1.2.1: Summary of Subject Baseline Characteristics (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Total Psoriasis Symptom Diary (PSD) Score | | | <u>, , </u> |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Dermatology Life Quality Index (DLQI) Score | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Height (cm) | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Weight (kg) | | | |
| n | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>a</sup> Collected for subjects with intertriginous involvement.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



# Repeat Table 14.1.2.1 for the following:

Table 14.1.2.2: Summary of Subject Baseline Characteristics (Per-Protocol Population)

Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population)

Table 14.1.2.4: Summary of Subject Baseline Characteristics (PK Population)



Table 14.1.3: Summary of Medical History by MedDRA System Organ Class and Preferred Term (Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | ARQ-151 Cream 0.3% (N=xxx) | ARQ-151 Cream 0.15%<br>(N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more medical histories that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.1.4.1: Summary of Prior Medications by WHO-DD ATC Level 2 Term and Preferred Name (Safety Population)

| ATC Level 2 Term <sup>a</sup> Preferred Name | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | XX (XX.X%) | xx (xx.x%) |
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Table includes all medications used prior to date of first dose of study drug.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more prior medications that map to the WHO-DD (Version March 1, 2018). At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once.



Table 14.1.4.2: Summary of Concomitant Medications by WHO-DD ATC Level 2 Term and Preferred Name (Safety Population)

| ATC Level 2 Term <sup>a</sup> Preferred Name | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Table includes all medications used on or after date of first dose of study drug.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more concomitant medications that map to the WHO-DD (Version March 1, 2018). At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once.



Table 14.2.1.1: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Intent-to-Treat Population)

| IGA Score of Clear or Almost Clear at Week 6 | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline IGA score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.1.1 for the following:

Table 14.2.1.2: Analysis of Primary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6 (Per-Protocol Population)



Figure 14.2.1.1: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Intent-to-Treat Population)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

 $SOURCE: USERNAME \verb|\SPONSOR|| PROJECT \verb|\JOBNAME|| (DATE, TIME)$ 

Repeat Figure 14.2.1.1 for the following:

Figure 14.2.1.2: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' by Visit (Per-Protocol Population)



Table 14.2.2.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population)

| GA Score of Clear or Almost Clear<br>Week 2 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 4 | | | |
| Success | xx.x% | XX.X% | XX.X% |
| Failure | XX.X% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 8 | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Failure | $XX.X^{0}/_{0}$ | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 12 | | | |
| Success | xx.x% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | xx.x% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Contrast P-Value vs Vehicle Cream | x.xxx | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline IGA score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

### Repeat Table 14.2.2.1 for the following:

Table 14.2.2.2: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' (Per-Protocol Population)



Table 14.2.3.1: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA)
Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline
(Intent-to-Treat Population)

| IGA Score of Clear or Almost Clear<br>Plus a 2-Grade Improvement from Baseline | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2 | (N=xx) | <u>(N=xx)</u> | (IN-XX) |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | AA.A/0 |
| Week 4 | | | |
| Success | xx.x% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | xx.x% | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 6 | | | |
| Success | xx.x% | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | xx.x% | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 8 | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| Week 12 | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline IGA score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

 $SOURCE: USERNAME \verb|\SPONSOR| PROJECT \verb|\JOBNAME| (DATE, TIME)$ 

Repeat Table 14.2.3.1 for the following:

Table 14.2.3.2: Analysis of Secondary Efficacy Endpoint: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline (Per-Protocol Population)



Figure 14.2.3.1: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline by Visit (Intent-to-Treat Population)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Figure 14.2.3.1 for the following:

Figure 14.2.3.2: Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement from Baseline by Visit (Per-Protocol Population)



Table 14.2.3.3: Summary of Proportion of Subjects Achieving an Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear'
Plus a 2-Grade Improvement from Baseline by Investigational Site
(Intent-to-Treat Population)

| Investigational Site | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxx | xx/xx ( xx.x%) | xx/xx (xx.x%) | xx/xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxx | xx/xx ( $xx.x%$ ) | xx/xx ( xx.x%) | xx/xx ( $xx.x%$ ) |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx/xx ( $xx.x%$ ) | xx/xx ( $xx.x%$ ) | xx/xx ( $xx.x%$ ) |
| xxxxxxxxxxxxxxxxxxxxxx | xx/xx ( $xx.x%$ ) | xx/xx ( xx.x%) | xx/xx ( $xx.x%$ ) |
| xxxxxxxxxxxxxxxxxxxxxx | xx/xx ( xx.x%) | xx/xx ( $xx.x%$ ) | xx/xx ( $xx.x%$ ) |
| xxxxxxxxxxxxxxxxxxxxxx | xx/xx ( xx.x%) | xx/xx ( $xx.x%$ ) | xx/xx ( $xx.x%$ ) |

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.4.1.1: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)

| I-IGA Score of Clear or Almost Clear Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2<br>Success | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | XX.X <sup>7</sup> 0<br>XX.X <sup>9</sup> % | xx.x%<br>xx.x% | XX.X % |
| Contrast P-Value vs Vehicle Cream | | | XX.X / 0 |
| Contrast F-value vs venicle Cleani | X.XXX | X.XXX | |
| Week 4 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 6 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 12 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | AA.A/0 |
| Contrast 1 value vs vemere cream | A.AAA | Α.ΑΑΑ | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline I-IGA score.

Restricted to subjects with an I-IGA severity score of at least "Mild" at baseline.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Table 14.2.4.1.1 for the following:

Table 14.2.4.1.2: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Figure 14.2.4.1.1: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear'

(Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Figure 14.2.4.1.1 for the following:

Figure 14.2.4.1.2: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)


Table 14.2.4.2.1: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)

| I-IGA Score of Clear or Almost Clear Plus a 2 Grade<br>Improvement from Baseline<br>Week 2 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 6 | | | |
| Success | xx.x% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | xx.x% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| Success | XX.X% | XX.X% | XX.X% |
| Failure | XX.X% | xx.x% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 12 | | | |
| Success | $XX.X^{0}/_{0}$ | XX.X% | XX.X% |
| Failure | $XX.X^{0}/_{0}$ | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline I-IGA score.

Restricted to subjects with an I-IGA severity score of at least "Mild" at baseline.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.



Repeat Table 14.2.4.2.1 for the following:

Table 14.2.4.2.2: Analysis of Secondary Efficacy Endpoint: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Figure 14.2.4.2.1: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Intent-to-Treat Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Figure 14.2.4.2.1 for the following:

Figure 14.2.4.2.2: Subjects with an Intertriginous Area Investigator Global Assessment (I-IGA) Severity of at Least 'Mild' at Baseline who Achieved a Score of 'Clear' or 'Almost Clear' Plus a 2 Grade Improvement from Baseline (Per-Protocol Population: Subjects with I-IGA Severity of at Least 'Mild' at Baseline)



Table 14.2.5.1.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI)

(Intent-to-Treat Population)


| ASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | · · | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PASI score.



Table 14.2.5.1.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | x.xxx | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PASI score.



Table 14.2.5.1.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI)

(Intent-to-Treat Population)


| ASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PASI score.



Table 14.2.5.1.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI)

(Intent-to-Treat Population)


| ASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PASI score.



Table 14.2.5.1.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI)

(Intent-to-Treat Population)


| ASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PASI score.



Table 14.2.5.1.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PASI score.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.5.1.1 for the following:

Table 14.2.5.1.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI) (Per-Protocol Population)



Figure 14.2.5.1.1: Percent Change from Baseline in Psoriasis Area and Severity Index (PASI) (Intent-to-Treat Population)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.5.2.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| nPASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.2.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | xx.xx | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.2.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.2.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| mPASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | x.xxx | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.2.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| mPASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | x.xxx | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.



Table 14.2.5.2.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI)

(Intent-to-Treat Population)


| PASI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline mPASI score.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.5.2.1 for the following:

Table 14.2.5.2.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Per-Protocol Population)



Figure 14.2.5.2.1: Percent Change from Baseline in Modified Psoriasis Area and Severity Index (mPASI) (Intent-to-Treat Population)



Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.6.1.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline
(Intent-to-Treat Population)


| Reduction in PASI Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 2 | (IV MI) | (IV III) | (1) III) |
| 75% Reduction | | | |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | x.xxx | |
| 90% Reduction | | | |
| Success | xx.x% | XX.X% | XX.X% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| 100% Reduction | | | |
| Success | $XX.X^{0}/_{0}$ | xx.x% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| 75% Reduction | | | |
| Success | XX.X% | XX.X% | xx.x% |
| Failure | XX.X% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | XX.X% | XX.X% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 100% Reduction | | | |
| Success | XX.X% | xx.x% | XX.X% |
| Failure | XX.X% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline PASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.6.1.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline
(Intent-to-Treat Population)


| Reduction in PASI Compared to Baseline | ARQ-151 Cream 0.3% (N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | (1) (AA) | (14 AA) | (IV AA) |
| 75% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 100% Reduction | | | |
| Success | $XX.X^{0}/_{0}$ | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | $XX.X^{0}/_{0}$ | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| 75% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 100% Reduction | | | |
| Success | XX.X% | XX.X% | xx.x% |
| Failure | XX.X% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline PASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.6.1.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Intent-to-Treat Population)


| Reduction in PASI Compared to Baseline | ARQ-151 Cream 0.3% (N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Veek 12 | (1: 111) | (2 , 1112) | (1111) |
| 75% Reduction | | | |
| Success | $XX.X^{0}/_{0}$ | xx.x% | xx.x% |
| Failure | $XX.X^{0}/_{0}$ | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 100% Reduction | | | |
| Success | $XX.X^{0}/_{0}$ | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline PASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## Repeat Table 14.2.6.1.1 for the following:

Table 14.2.6.1.2 Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Per-Protocol Population)



Table 14.2.6.2.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| Reduction in mPASI Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 2 | (IV MI) | (IV III) | (1) III) |
| 75% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 90% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 100% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| 75% Reduction | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | X.XXX | |
| 100% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline mPASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.6.2.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| Reduction in mPASI Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | (IN-AA) | (1\-\A\) | (11-XX) |
| 75% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 90% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 100% Reduction | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| 75% Reduction | | | |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 90% Reduction | | | |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| 100% Reduction | | | |
| Success | XX.X% | xx.x% | xx.x% |
| Failure | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline mPASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



## Table 14.2.6.2.1: Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population) 

| Reduction in mPASI Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | (1 - 1112) | (1, 1111) |
| 75% Reduction | | | |
| Success | xx.x% | xx.x% | XX.X% |
| Failure | xx.x% | $XX.X^{0}/_{0}$ | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 90% Reduction | | | |
| Success | xx.x% | $XX.X^{0}/_{0}$ | XX.X% |
| Failure | xx.x% | $XX.X^{0}/_{0}$ | XX.X% |
| Contrast P-Value vs Vehicle Cream | X.XXX | x.xxx | |
| 100% Reduction | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline mPASI score.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## Repeat Table 14.2.6.2.1 for the following:

Table 14.2.6.2.2 Analysis of Secondary Efficacy Endpoints: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population)



Table 14.2.7.1.1: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Intent-to-Treat Population)


| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2 | | | |
| 75% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in PASI Compared to Baseline | | | |
| Success | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | | |
| 75% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.7.1.1: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Intent-to-Treat Population)


| Week 6 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| 75% Reduction in PASI Compared to Baseline Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 diluic | AA ( AA.A70) | AA ( AAA70) | AA ( AA.A/0) |
| 90% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in PASI Compared to Baseline Success Failure | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Week 8 75% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in PASI Compared to Baseline | ( 0/) | ( 0() | ( ) |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.7.1.1: Dichotomized Percent Reductions in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Intent-to-Treat Population)


| Week 12 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| 75% Reduction in PASI Compared to Baseline Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | XX (XX.X%) $XX (XX.X%)$ | xx ( xx.x%) | xx ( xx.x%) |
| 000/ Dalastica in DACI Camanada Daratica | | | |
| 90% Reduction in PASI Compared to Baseline Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | XX (XX.X%) | XX (XX.X%) |
| 1000/ P. 1. ('' PACI C | | | |
| 100% Reduction in PASI Compared to Baseline Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| W. 146 | | , | . , |
| Week 16 75% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in PASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in PASI Compared to Baseline Success | ( | ( 0/) | ( |
| Failure | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| 1 andie | AA ( AA.A/0) | AA ( AA.A/0) | AA ( AA.A/0) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.7.1.1 for the following:

Table 14.2.7.1.2: Dichotomized Percent Reduction(s) in Psoriasis Area and Severity Index (PASI) Compared to Baseline (Per-Protocol Population)



Table 14.2.7.2.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| Week 2 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| 75% Reduction in mPASI Compared to Baseline | 0() | ( , | ( , , , , , , ) |
| Success<br>Failure | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| ranure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline Success Failure | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Week 4 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline Success | (0/) | ( | ( 0/) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.7.2.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| Week 6 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | | |
| 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.7.2.1: Dichotomized Percent Reductions in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Intent-to-Treat Population)


| Week 12 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| 75% Reduction in mPASI Compared to Baseline Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%)<br>xx ( xx.x%) | XX (XX.X%)<br>XX (XX.X%) | xx ( xx.x%)<br>xx ( xx.x%) |
| 1 and | AA ( AA.A/0) | AA ( AA.A/0) | AA ( AA.A/0) |
| 90% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline Success Failure | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Week 16 75% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90% Reduction in mPASI Compared to Baseline | | | 4 |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 100% Reduction in mPASI Compared to Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.7.2.1 for the following:

Table 14.2.7.2.2: Dichotomized Percent Reduction(s) in Modified Psoriasis Area and Severity Index (mPASI) Compared to Baseline (Per-Protocol Population)



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data at Week 16 was not imputed.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| 3SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | xx.x | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| BSA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | x.xxx | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | x.xxx | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data at Week 16 was not imputed.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| SA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.



Table 14.2.8.1: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Intent-to-Treat Population)


| BSA | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline BSA score.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## Repeat Table 14.2.8.1 for the following:

Table 14.2.8.2: Analysis of Secondary Efficacy Endpoint: Percent Change from Baseline in Body Surface Area (BSA) Affected (Per-Protocol Population)


Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| VI-NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | xx | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | xx.x | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |

<sup>&</sup>lt;sup>a</sup>P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| -NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | | X.XXX | |

<sup>&</sup>lt;sup>a</sup>P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| -NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline n Mean | XX | XX | XX |
| SD | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | xx.x | xx.x | XX.X |
| | XX.XX | XX.XX | XX.XX |
| LS SD <sup>a</sup> | ΛΛ.ΛΛ | 74747474 | |

<sup>&</sup>lt;sup>a</sup>P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.9.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Intent-to-Treat Population)


| I-NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | xx | xx | XX |
| Mean | xx.x | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |

<sup>&</sup>lt;sup>a</sup>P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.9.1 for the following:

Table 14.2.9.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score (Per-Protocol Population)



Table 14.2.10.1.1: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline

(Intent-to-Treat Population: Subjects with WI-NRS Score ≥ 6 at Baseline)

| 4 Point Reduction in WI-NRS Compared to Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 2 | (IN-XX) | (IN-XX) | (IN-XX) |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 4 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 6 | | | |
| Success | xx.x% | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 8 | | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% |
| Contrast P-Value vs Vehicle Cream | X.XXX | X.XXX | |
| Week 12 | | | |
| Success | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% |
| Contrast P-Value vs Vehicle Cream | x.xxx | x.xxx | |

Note: P-values and estimates from a logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score.

Restricted to subjects with a baseline WI-NRS Score of 6 or greater.

Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.



Repeat Table 14.2.10.1.1 for the following:

Table 14.2.10.1.2: Analysis of Secondary Endpoint: Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score ≥ 6 at Baseline)



Table 14.2.10.2.1: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score ≥ 6 at Baseline and Achieved a 4 Point Reduction Compared to Baseline

(Intent-to-Treat Population: Subjects with WI-NRS Score ≥ 6 at Baseline)

| 4 Point Reduction in WI-NRS Compared to Baseline<br>Week 2 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx (xx.x%) | xx ( xx.x%) | XX (XX.X%) |
| 1 diluic | AA ( AA.A /0) | AA ( AA.A/0) | AA ( AA.A/0) |
| Week 4 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Week 6 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ` , | , | , |
| Week 12 | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

Restricted to subjects with a baseline WI-NRS Score of 6 or greater.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

## Repeat Table 14.2.10.2.1 for the following:

Table 14.2.10.2.2: Summary of Subjects with a Worst Itch Numerical Rating Scale (WI-NRS) Score  $\geq 6$  at Baseline and Achieved a 4 Point Reduction Compared to Baseline (Per-Protocol Population: Subjects with WI-NRS Score  $\geq 6$  at Baseline)



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| Total PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| otal PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| al PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| al PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| al PSD Score | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.11.1: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Intent-to-Treat Population)


| otal PSD Score<br>Week 16 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD score.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.11.1 for the following:

Table 14.2.11.2: Analysis of Secondary Efficacy Endpoint: Total Psoriasis Symptom Diary (PSD) Score Compared to Baseline (Per-Protocol Population)



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| PSD Responses to Individual Questions <question></question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | xx.xx | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | x.xxx | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| D Responses to Individual Questions | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Question> | | | |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | xx.x | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| D Responses to Individual Questions | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| duestion> | | | |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions Question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Question> | | | |
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Question> | | | |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.



Table 14.2.12.1: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Intent-to-Treat Population)


| SD Responses to Individual Questions<br>Question> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline PSD response.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data for Week 16 was not imputed.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.12.1 for the following:

Table 14.2.12.2: Analysis of Secondary Efficacy Endpoint: Improvement in Psoriasis Symptom Diary (PSD) Responses Compared to Baseline (Per-Protocol Population)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| tch-Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| n-Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| n-Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| -Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score.

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.2.13.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Intent-to-Treat Population)


| h-Related Sleep Loss | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score. Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.13.1 for the following:

Table 14.2.13.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Itch-Related Sleep Loss Score (Per-Protocol Population)



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| DLQI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| QI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| oLQI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| QI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Creama | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.



Table 14.2.14.1: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Intent-to-Treat Population)


| LQI | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| LS Mean <sup>a</sup> | XX.X | XX.X | XX.X |
| LS SD <sup>a</sup> | XX.XX | XX.XX | XX.XX |
| Contrast P-Value vs Vehicle Cream <sup>a</sup> | X.XXX | X.XXX | |

<sup>&</sup>lt;sup>a</sup> P-values and estimates from an ANCOVA with a factor of treatment group and a covariate of baseline DLQI score.

Repeat Table 14.2.14.1 for the following:

Table 14.2.14.2: Analysis of Secondary Efficacy Endpoint: Change from Baseline in Dermatology Life Quality Index (DLQI) Score (Per-Protocol Population)



Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population)


| NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population)


| NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 4 | (2: 122) | (1. 122) | (1, 1111) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.2.15.1: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Intent-to-Treat Population)


| NRS | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 8 | | <u></u> | (= : ====) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Repeat Table 14.2.15.1 for the following: Table 14.2.15.2: Summary of Exploratory Endpoint: Change from Baseline in Fatigue NRS Score (Per-Protocol Population)



Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population)


| Score Type> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population)


| Score Type> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |


Table 14.2.16.1: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Intent-to-Treat Population)


| Score Type> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

Note: Missing data imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Table 14.2.16.1 for the following:

Table 14.2.16.2: Summary of Exploratory Endpoint: Change from Baseline in Work Productivity and Activity Impairment (WPAI) Score (Per-Protocol Population)



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 8 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.17.1: Summary of Whole Body Investigator Global Assessment (IGA)
(Intent-to-Treat Population)


| Whole Body Investigator Global Assessment | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | | |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.17.1 for the following:

Table 14.2.17.2: Summary of Whole Body Investigator Global Assessment (IGA) (Per-Protocol Population)



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | | |
| 0-Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 6 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| ntertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Veek 8 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 12 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.

Note: Missing data through Week 12 imputed using linear interpolation and last observation carried forward where linear interpolation is not computationally possible. Missing data was not imputed for Week 16.



Table 14.2.18.1: Summary of Intertriginous Area Investigator Global Assessment (I-IGA)
(Intent-to-Treat Population)


| Intertriginous Area Investigator Global Assessment <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 16 | | | |
| n | XX | XX | XX |
| 0 – Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Score of Clear or Almost Clear and | | | |
| a 2-Grade Improvement from Baseline <sup>b</sup> | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Collected at baseline for subjects with intertriginous area involvement and collected post-baseline for subjects with a severity of at least mild at baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.18.1 for the following:

Table 14.2.18.2: Summary of Intertriginous Area Investigator Global Assessment (I-IGA) (Per-Protocol Population)

<sup>&</sup>lt;sup>b</sup> Restricted to subjects with a severity of at least mild at baseline.



Table 14.3.0.1.1: Summary of Extent of Exposure (Safety Population)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Number of Doses | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Amount of Drug Applied (g) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Compliant <sup>a</sup> | | | |
| n | XX | XX | XX |
| Yes | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> A subject is considered compliant with the dosing regimen if the subject applied at least 80% of the expected doses during the dosing period and did not miss more than 3 consecutive doses.



Table 14.3.0.2.1: Summary of Pre-Dose Pharmacokinetic Concentrations (PK Population) (Page 1 of xx)

| <parameter> (<units>) Baseline</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | | | |
| SD | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | xx.x |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.0.2.1: Summary of Pre-Dose Pharmacokinetic Concentrations (PK Population) (Page 2 of xx)

| Parameter> ( <units>)<br/>Week 12</units> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.0.2.2: Summary of Additional Pharmacokinetic Concentrations (PK Population)

| <b>D</b> | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| <parameter> (<units>)</units></parameter> | (N=xx) | (N=xx) | (N=xx) |
| 72 hr (3 days) | | | |
| n<br>M | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| 120 hr (5 days) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| 168 hr (7 days) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| 216 hr (9 days) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Baseline | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | , | , | , |
| Minimal edema or minimal papular response | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Subject Local Tolerability Sensation Following Drug Application Baseline | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | xx ( xx.x%) | XX (XX.X%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | AA ( AA.A/0) | AA ( AA.A.70) | AA ( AA.A70) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Week 4 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | , | , | , |
| Minimal edema or minimal papular response | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Subject Local Tolerability Sensation Following<br>Drug Application<br>Week 4 | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Week 8 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | ( | ( | ( |
| Minimal edema or minimal papular response | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx (xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| Subject Local Tolerability Sensation Following<br>Drug Application<br>Week 8 | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Local Tolerability (Safety Population) 

| Investigator Local Tolerability Dermal Response Week 12 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| 0 – No evidence of irritation | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 – Minimal Erythema, Barely Perceptible | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 – Definite Erythema, Readily Visible; | | | |
| Minimal edema or minimal papular response | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Erythema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Definite Edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – Erythema, Edema and Papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 – Vesicular Eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 – Strong Reaction Spreading Beyond Application Site | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Subject Local Tolerability Sensation Following<br>Drug Application<br>Week 12 | | | |
| n | XX | XX | XX |
| 0 – No sensation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Slight warm, tingling sensation; not really bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Definite warm, tingling sensation that is somewhat bothersome | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Hot, tingling/stinging sensation that has caused definite discomfort | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Figure 14.3.1.1: Subject Local Tolerability Sensation Following Drug Application (Safety Population)



Note: 0 (No sensation), 1 (Slight warm, tingling sensation; not really bothersome), 2 (Definite warm, tingling sensation that is somewhat bothersome),

3 (Hot, tingling/stinging sensation that has caused definite discomfort)



Table 14.3.1.2.1: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Injurious Behavior without Suicidal Intent Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population)

| | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| Events during treatment | (N=xx) | (N=xx) | (N=xx) |
| Suicidal Ideation (1-5) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1) Wish to be dead | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2) Non-specific active suicidal thoughts | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3) Active suicidal ideation with any methods (not plan) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| without intent to act | | | |
| 4) Active suicidal ideation with some intent to act, without | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| specific plan | · · · · · · | ` ' | , |
| 5) Active suicidal ideation with specific plan and intent | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| , | | | |
| Suicidal Behavior (6-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6) Preparatory acts or behavior | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7) Aborted attempt | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 8) Interrupted attempt | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 9) Non-fatal suicide attempt | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 10) Completed suicide | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Suicidal Ideation or Behavior (1-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Self-injurious behavior without suicidal intent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.2.2: Number of Patients with Suicide-Related Treatment-Emergent Events Based on the Colombia-Suicide Severity Rating Scale (C-SSRS) During
Treatment
(Safety Population)

| Treatment-emergent (TE) Events TE suicidal ideation (1-5) compared to recent history <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx)<br>xx (xx.x%) | ARQ-151 Cream 0.15%<br>(N=xx)<br>xx (xx.x%) | Vehicle Cream (N=xx) xx (xx.x%) |
|---|---|---|---|
| TE serious suicidal ideation (0-3 to 4-5) compared to recent history <sup>b</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Emergence of serious suicidal ideation (0 to 4-5) compared to recent history <sup>c</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Improvement in suicidal ideation at endpoint compared with baseline <sup>d</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Emergence of suicidal behavior (6-10) compared to all prior history <sup>e</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> N=Number of enrolled patients with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the comparison period is non-missing and <5.

<sup>&</sup>lt;sup>b</sup> N=Number of enrolled patients with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the comparison period is 0-3.

<sup>&</sup>lt;sup>c</sup> N=Number of enrolled patients with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the comparison period is 0.

<sup>&</sup>lt;sup>d</sup> N=Number of enrolled patients whose suicidal ideation score is non-missing and >0 just prior to treatment.

<sup>&</sup>lt;sup>e</sup>N=number of enrolled patients with with at least one post-baseline C-SSRS assessment and who did not have suicidal behavior (6-10) prior to treatment.



Table 14.3.1.3.1: Summary of PHQ-8 Assessments by Treatment Group (Safety Population)

| NIO 0 A | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| PHQ-8 Assessment | (N=xx) | (N=xx) | (N=xx) |
| Baseline | | | |
| n<br>N | XX | ( 0() | ( 0/) |
| None – Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | | |
| n | XX | XX | XX |
| None – Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | | |
| n | XX | XX | XX |
| None – Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | , | , | , , |
| n | XX | XX | XX |
| None – Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population)


| PHQ-8 for (ARQ-151 Cream 0.3%) | | | Week 4 | | |
|---|---|---|---|---|---|
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | $xx \overline{(xx.x\%)}$ |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 8 | | |
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | $xx \overline{(xx.x\%)}$ |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 12 | | |
| <u>Baseline</u> | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).



Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population)


| PHQ-8 for (ARQ-151 Cream 0.15%) | | | Week 4 | | |
|---|---|---|---|---|---|
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 8 | | |
| Baseline | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | | | Week 12 | | |
| <u>Baseline</u> | None | Mild | Moderate | Moderately Severe | Severe |
| None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).



Table 14.3.1.3.2: Shift Summary of PHQ-8 Assessments by Treatment Group (Safety Population)


| PHQ-8 for (Vehicle Cream) Name Mild Medanta N | | |
|---|---|---|
| Baseline None Mild Moderate N | Moderately Severe | Severe |
| None $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Mild $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Moderate $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe xx (xx.x%) xx (xx.x%) xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe $xx (xx.x\%)$ $xx (xx.x\%)$ $xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | |
| Baseline None Mild Moderate M | Moderately Severe | Severe |
| None $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx (xx.x%) |
| Mild $xx (xx.x\%)$ $xx (xx.x\%)$ $xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Moderate $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Severe $xx (xx.x\%)$ $xx (xx.x\%)$ $xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| Baseline None Mild Moderate M | Moderately Severe | Severe |
| None $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Mild $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Moderate $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe $xx (xx.x\%) xx (xx.x\%) xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| Severe $xx (xx.x\%)$ $xx (xx.x\%)$ $xx (xx.x\%)$ | xx ( xx.x%) | xx ( xx.x%) |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).



Table 14.3.1.4.1: Overall Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)

| | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Subjects with any TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of TEAEs | XX | XX | XX |
| subjects with any Related TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related TEAEs | XX | XX | XX |
| subjects with any Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX |
| subjects with any Related Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Serious TEAEs | XX | XX | XX |
| ubjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ubjects who Discontinued Study Drug due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ubjects who Discontinued Study due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity By Subject | | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | |
| Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unrelated | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.4.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Table 14.3.1.4.3: Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug by MedDRA System Organ Class and Preferred Term

(Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | XX (XX.X%) | xx (xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Table 14.3.1.4.4: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | Severity <sup>b</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|---|
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.



Table 14.3.1.4.5: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)


| System Organ Class <sup>a</sup> | | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|---|
| Preferred Term | <u>Relationship</u> | (N=xx) | (N=xx) | (N=xx) |
| Total | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.



Table 14.3.1.4.6: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)

| | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Subjects with any Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX |
| Subjects with any Related Serious TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Related Serious TEAEs | XX | XX | XX |
| Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Subjects who Discontinued Study Drug due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Subjects who Discontinued Study due to TEAE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity By Subject | | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 1 | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | |
| Likely | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset after first dose of study drug. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.3.1.4.7: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.


Table 14.3.1.4.8: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | Severity <sup>b</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|---|
| Total | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| , | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset after first dose of study drug.

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

<sup>&</sup>lt;sup>b</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.



Table 14.3.1.4.9: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)

| System Organ Class <sup>a</sup> | | ARQ-151 Cream 0.3% | ARQ-151 Cream 0.15% | Vehicle Cream |
|---|---|---|---|---|
| Preferred Term | <u>Relationship</u> | (N=xx) | (N=xx) | (N=xx) |
| Total | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| System Organ Class | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA dictionary (Version 21.1). At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: Treatment-emergent adverse events are those with an onset after first dose of study drug.



Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results
(Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results (Safety Population)

| <b>EParameter&gt; (<units>)</units></b> Week 12 | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

Repeat Table 14.3.1.5.1.1: Summary of Chemistry Laboratory Results

For the following tables:

Table 14.3.1.5.1.2: Summary of Hematology Laboratory Results (Safety Population)

Table 14.3.1.5.1.3: Summary of Quantitative Urinalysis Laboratory Results (Safety Population)



# Table 14.3.1.5.2.1: Shift Summary of Chemistry Laboratory Results (Safety Population) (Page 1 of x)

| <test name=""> (<units>)</units></test> | AF | Q-151 Cream 0<br>(N=xx) | 0.3% | ARG | Q-151 Cream 0<br>(N=xx) | 0.15% | | Vehicle Cream<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|
| | | Week 4 | | | Week 4 | | | Week 4 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx( xx.x%) | xx( xx.x%) | xx( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) xx | x( xx.x%) |
| | | | | | | | , , | xx( xx.x%) xx | |
| ANL | xx ( xx.x%) | xx ( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) xx | x( xx.x%) |
| | | Week 12 | | | Week 12 | | | Week 12 | |
| Baseline | BNL | WNL | ANL | BNL | WNL | ANL | BNL | WNL | ANL |
| BNL | xx( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) xx | x( xx.x%) |
| | | | | , , | | | , , | xx( xx.x%) xx | ` ' |
| | | | | | | | | xx ( xx.x%) xx | |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.3.1.5.2.1: Shift Summary of Chemistry Laboratory Results

For the following tables:

Table 14.3.1.5.2.2: Shift Summary of Hematology Laboratory Results (Safety Population)

Table 14.3.1.5.2.3: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population)



Table 14.3.1.6.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.6.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population)

| Parameter> ( <units>)<br/>Week 12</units> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.6.2: Shift Summary of Overall Electrocardiogram (ECG) Assessments (Safety Population)
(Page 1 of x)

| Overall ECG Assessment | _ | ~ | Cream 0.3%<br>=xx) | - | Cream 0.15%<br>=xx) | | e Cream<br>=xx) |
|---|---|---|---|---|---|---|---|
| | _ | We | ek 4 | We | ek 4 | W6 | eek 4 |
| <u>B</u> | Baseline | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal |
| N | Vormal 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| A | Abnormal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | _ | Wee | ek 12 | Wee | ek 12 | We | ek 12 |
| <u>B</u> | Baseline | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal |
| N | Jormal 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| A | Abnormal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 2 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 6 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| <parameter> (<units>)</units></parameter> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream (N=xx) |
|---|---|---|---|
| Week 8 | (IV AA) | (IV AA) | (IV AA) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | xx.x |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.1: Summary of Vital Signs (Safety Population)

| 'arameter> ( <units>)<br/>Week 16</units> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.3.1.7.2: Summary of Change in Body Weight Compared to Baseline (Safety Population)


| Change in Body Weight Compared to Baseline <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 4 | (11-AA) | (IV-AX) | (IV-AA) |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx (xx.x%) | xx ( xx.x%) | XX (XX.X%) |
| Week 6 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |

<sup>&</sup>lt;sup>a</sup> Percentages may sum to over 100% due to the possibility of being included in more than one category. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.3.1.7.2: Summary of Change in Body Weight Compared to Baseline (Safety Population)


| Change in Body Weight Compared to Baseline <sup>a</sup> | ARQ-151 Cream 0.3%<br>(N=xx) | ARQ-151 Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) |
|---|---|---|---|
| Week 16 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Percentages may sum to over 100% due to the possibility of being included in more than one category. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



#### 11. INDEX OF PLANNED LISTINGS

| Listing 16.2.1.1: End of Study Information | 174 |
|---|---|
| Listing 16.2.1.2: Discontinued Subjects | 175 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations | 176 |
| Listing 16.2.2.2: Protocol Deviations | 177 |
| Listing 16.2.3: Analysis Populations | 178 |
| Listing 16.2.4.1: Subject Demographic Information | 179 |
| Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Claude and Preferred Terms | |
| Listing 16.2.4.2.2: Medical/Surgical History | 181 |
| Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DD ATC Level 2 Terms an Preferred Names | |
| Listing 16.2.4.3.2: Prior and Concomitant Medications | 183 |
| Listing 16.2.4.4.1: Unique Therapies and Procedures Coded to MedDRA System Organ Claud Preferred Terms | |
| Listing 16.2.4.4.2: Prior and Concomitant Therapies and Procedures | 185 |
| Listing 16.2.4.5: Physical Examination | 186 |
| Listing 16.2.5.1: Study Visit Compliance | 187 |
| Listing 16.2.5.2: Drug Accountability | 188 |
| Listing 16.2.5.3: Study Drug Application | 189 |
| Listing 16.2.5.4: Dosing Compliance | 190 |
| Listing 16.2.5.5: Dosing Deviations | 191 |
| Listing 16.2.6.1: Investigator Global Assessment (IGA) | 192 |
| Listing 16.2.6.2: Body Surface Area (BSA) Involved with Psoriasis | 193 |
| Listing 16.2.6.3: Psoriasis Area and Severity Index (PASI) | 194 |
| Listing 16.2.6.4: Numeric Rating Scale (NRS) Assessments/Sleep Loss | 195 |
| Listing 16.2.6.5.1: Dermatology Life Quality Index (DLQI) Questionnaire Descriptions | 196 |
| Listing 16.2.6.5.2: Dermatology Life Quality Index (DLQI) Questionnaire | 197 |
| Listing 16.2.6.6.1: Work Productivity and Activity Impairment (WPAI) Questionnaire Descriptions | 198 |
| Listing 16.2.6.6.2: Work Productivity and Activity Impairment (WPAI) Questionnaire | 199 |
| Listing 16.2.6.7: Columbia-Suicide Severity Rating Scale (C-SSRS) | 200 |



| Listing 16.2.6.8.1: Patient Health Questionnaire Depression Scale (PHQ-8) Question Descriptions | 201 |
|---|---|
| Listing 16.2.6.8.2: Patient Health Questionnaire Depression Scale (PHQ-8) | 202 |
| Listing 16.2.6.9.1: Psoriasis Symptom Diary (PSD) Questionnaire Descriptions | 203 |
| Listing 16.2.6.9.2: Psoriasis Symptom Diary (PSD) Questionnaire | 204 |
| Listing 16.2.6.10: Photography Information | 205 |
| Listing 16.2.7.1.1: Investigator Local Tolerability Assessment | 206 |
| Listing 16.2.7.1.2: Subject Local Tolerability Assessment | 207 |
| Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms | 208 |
| Listing 16.2.7.2.2: Treatment-Emergent Adverse Events | 209 |
| Listing 16.2.7.2.3: Serious Adverse Events | 210 |
| Listing 16.2.7.2.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events | 211 |
| Listing 16.2.8.1: Urine Pregnancy Test Results | 212 |
| Listing 16.2.8.2.1: Laboratory Test Results | 213 |
| Listing 16.2.8.2.2: Abnormal Laboratory Results | 214 |
| Listing 16.2.8.3: 12-lead Electrocardiogram Test Results | 215 |
| Listing 16.2.8.4: Vital Signs | 216 |
| Listing 16.2.8.5: Pharmacokinetics Blood Sample Collections | 217 |



### Listing 16.2.1.1: End of Study Information Treatment Group (Page xx of yy)

| S: Subject | | | |
|---|---|---|---|
| A: Age/Sex | F: Date of First Dose of Dr | rug Primary Reason for Study | |
| E: Eval | L: Date of Last Dose of Dru | g Completion/Discontinuation | Date of Completion/Discontinuation |
| S: xxxxxx | F: xxxxxxxxx | ********* ** ********** | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxx | | |
| E: xxxxxxxxx | | | |
| S: xxxxxx | F: xxxxxxxxx | xxxxxxxxx xx xxxxxxxxxxxxx | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxxx | | |
| E: xxxxxxxxx | | | |
| S: xxxxxx | F: xxxxxxxxx | xxxxxxxx xxxx xxxxxxx xxxxx | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxx | | |
| E: xxxxxxxxx | | | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Note to programmer: concatenate 'Describe' text onto Primary Reason where applicable.



# Listing 16.2.1.2: Discontinued Subjects Treatment Group (Page xx of yy)

| S: Subject | | | |
|---|---|---|---|
| A: Age/Sex | F: Date of First Dose of Dru | g Primary Reason for Study | |
| E: Eval | L: Date of Last Dose of Drug | Completion/Discontinuation | Date of Completion/Discontinuation |
| S: xxxxxx | F: xxxxxxxxx | ********* ** ********** | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxxx | | |
| E: xxxxxxxxx | | | |
| S: xxxxxx | F: xxxxxxxxx | xxxxxxxxx xx xxxxxxxxxxxxx | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxx | | |
| E: xxxxxxxx | | | |
| S: xxxxxx | F: xxxxxxxxx | xxxxxxxx xxxx xxxxxxx xxxxx | xxxxxxxxx xxxx |
| A: xxxx | L: xxxxxxxxx | | |
| E: xxxxxxxxx | | | |

\_\_\_\_\_



### Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Criterion<br>Category | Criterion<br>Identifier | Description |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | Х | ******* *** **** * **** ** * ******* ** * |
| | | | xxxxxxxx | х | ******* **** **** * ***** ** * ******** |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxx | х | ******* **** **** * ***** ** * ******** |
| | | | xxxxxxxx | xx | ******** **** ***** **** **** ****** **** |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | х | ******* **** **** * ***** ** * ******** |
| | | | xxxxxxxx | xx | ******* **** **** * **** ** * ******* ** * |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Criterion Category, and Criterion Identifier.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Page 176 of 217



# Listing 16.2.2.2: Protocol Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Protocol Deviation |
|---------|---------|----------|-----------------------------------------------|
| xxxxxx | xxxx | xxxxxxxx | XXXXXXXXX XXXX X XXXXXXX XX XXXXXXXXXX |
| xxxxx | xxxx | xxxxxxxx | XXXXXXXX X XXXXXXX XXXXXXXXX XX XXX<br>XXXXXX |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx xxxx xxxx x xxxxx xx x xxxxxxx |
| xxxxxx | XXXX | xxxxxxxx | XXXXXXXX X XXXXXX XXXXXXXX XXXXXXXX XX |



# Listing 16.2.3: Analysis Populations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Population | Included | Reason(s) Excluded |
|---|---|---|---|---|
| xxxxxx | xxxx | Safety | xx | xxxxxx x xxxxxx xxxxxxxx |
| ^^^^ | AAAA | Intent-to-Treat | XXX | ******* * ****** |
| | | Per-Protocol | XXX | |
| | | Pharmacokinetic | XXX | |
| xxxxxx | xxxx | Safety | xxx | |
| | | Intent-to-Treat | XXX | |
| | | Per-Protocol | XXX | |
| | | Pharmacokinetic | XXX | |
| xxxxx | xxxx | Safety | xxx | |
| | | Intent-to-Treat | XXX | |
| | | Per-Protocol | XX | xxxxxx xxxxxx xxxx |
| | | Pharmacokinetic | XX | xxxxxxxxx xxxxxxx xxx xxxxxxxxx xx xxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, and Population.



### Listing 16.2.4.1: Subject Demographic Information (Page xx of yy)

| Subject | Eval | B: Date of Birth<br>S: Sex | D: Date/Time of<br>Informed Consent<br>A: Age at Consent | R: Race<br>E: Ethnicity | C: Childbearing Potential B: Birth Control Method | P: Did the Subject<br>Consent to Photography?<br>D: Date of<br>Photography Consent |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxx | B: xxxxxxxxxx<br>S: xxxx | D: xxxx-xx-xxTxx:xx:xx<br>A: xx | R: xxxxx xx xxxxxx<br>E: xxx xxxxxxx xx | C: xx<br>B: | P: xxx<br>D: xxxxxxxxx |
| xxxxx | xxxxxxx | B: xxxxxxxxxx<br>S: xxxxxx | D: xxxx-xx-xxTxx:xx<br>A: xx | R: xxxxx<br>E: xxx xxxxxxx xx | C: xxx<br>B: xxxxxxxxx xxxxxxx | P: xx<br>D: |
| xxxxxx | xxxxxxxx | B: xxxxxxxxxx<br>S: xxxxxx | D: xxxx-xx-xxTxx:xx:xx<br>A: xx | R: xxxxx<br>E: xxx xxxxxxx xx | C: xxx<br>B: xxxx xxxxxxxxxxxxx | P: xxx<br>D: xxxxxxxxx |



#### Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Condition/Surgery Verbatim Term |
|---|---|---|
| x xxx xxxxx | xxxx xxx xxxxx | xxxx xxxxxxxxx xx xxxxxx |
| | | xxxxx xxx xxxxxx xx |
| xxxx x xxxxxxxxx | xxxxxx xxxxxxxxxx | xxxx xxxxxx xxxxxxxx xx xxxxxx |
| xxxx xxx xxxxx | xxxx xxx xxxxx | xxxx xxxxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, and Verbatim Term.



### Listing 16.2.4.2.2: Medical/Surgical History Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Condition/Surgery<br>Verbatim Term | P: MedDRA Preferred Term<br>S: MedDRA System Organ Class | S: Onset Date<br>E: End Date |
|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxx xxxxxxx (xxxxxxxx xxxxx) | P: xxxxxx xxxxxxxxx<br>S: xxxxxxxxxx xxxxxxx | S: xxxxxxxxxx<br>E: xxxxxxxxxx |
| | | | xxxxxxx xxxxxxxxx | P: xxxxxxx xxxxxxxx<br>S: xxxxxx xxxxxxxxxxx | S: xxxxxxxxxxx<br>E: xxxxxxxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Medical Condition/Surgery, Start Date, and End Date.



#### Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DD ATC Level 2 Terms and Preferred Names (Page xx of yy)

| ATC Level 2 Term | Preferred Name | Medication Name | <pre>I: Indication R: Route</pre> |
|---|---|---|---|
| | | | I: xxxxxx xxxxxxx |
| XXXXXX XXXXXX XX XXX | xxxxxxxxx | xxxxxxxxx | R: xxxxx |
| | xxxxxx x | xxxxxx | I: xxxxxxx xxxxxxxx xxxxxxx |
| | | | R: xxxx |
| | xxxxxxxx | xxxxxxxx | I: xxxxxxx xxxxxxx xxxx xxxx xxxx |
| | | | R: xxxx |

Note: Preferred Name and ATC Level 2 Term map to the WHO-DD (Version March 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Preferred Name, Medication Name, Indication, and Route.



### Listing 16.2.4.3.2: Prior and Concomitant Medications Treatment Group (Page xx of yy)

M: Medication Name D: Dose P: Preferred Name F: Date of First Dose U: Units A: ATC Level 2 Term S: Start Date (Day) 1 F: Frequency Subject Age/Sex I: Indication E: End Date (Day) 1 Eval R: Route XXXXXX XXXX XXXXXXXXX M: xxxxxxxxxxxx F: xxxxxxxxxx D: xx P: xxxxxxxxxxxxx U: xx S: xxxxxxxxxx A: xxxxxxxxxxxx E: xxxxxxxxxx F: xxxx I: xxxxxxxx R:xxxx M: xxxxxxxxxxx F: xxxxxxxxxx D: xxxxx P: xxxxxxxxxxxx S: xxxxxxxxxx U: xx E: xxxxxxxxxx F: xx A: xxxxxxxxxxxx I: xxxxxxxx R:xxxx M: xxxxxxxxxxxx F: xxxxxxxxxx D: xxx XXXXXX XXXX XXXXXXXXX P: xxxxxxxxxxxx S: xxxxxxxxxx U: xx F: xx A: xxxxxxxxxxxx E: xxxxxxxxxx I: xxxxxxxx R:xxxx

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route. If ongoing, include 'Ongoing' in place of End Date. Concatenate Topical Area Treated onto route where applicable.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose. Note: Preferred Name and ATC Level 2 Term map to the WHO-DD (Version March 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



#### Listing 16.2.4.4.1: Unique Therapies and Procedures Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Procedure/Therapy Verbatim Term |
|---|---|---|
| xxxx xxx xxxxx | xxxx xxx xxxxx | XXXX |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |
| xxxx xxx xxxxx | xxxx xxx xxxxx | XXXX |
| | | ****** ******* ** ***** |
| | | ****** ******* ** **** |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, MedDRA Preferred Term, and Procedure/Therapy Verbatim Term.



#### Listing 16.2.4.4.2: Prior and Concomitant Therapies and Procedures (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | Procedure/Therapy Verbatim Term | I: Indication A: Anatomical Area | P: MedDRA Preferred Term S: MedDRA System Organ Class | S: Start Date<br>E: End Date |
|---|---|---|---|---|
| S: xxxxxx | xxxxx xxxxxxx (xxxxxxx xxxxx) | I: xxxxxxxxx | P: xxxxxx xxxxxxxxx | S: xxxxxxxxxx |
| A: XXXX | | A: xxxx | S: xxxxxxxxxx xxxxxx | E: xxxxxxxxxx |
| : xxxxxxxx | | | | |
| | XXXXXX XXXXXXX XXXXXXX | I: xxxxxxxxx xxxxx | P: xxxxxx xxxxxxxxx | S: xxxxxxxxxxx |
| | | A: | S: xxxxxxxxxx xxxxxxx | E: xxxxxxxxxx |
| S: xxxxxx | xxxxxx xxxxxxxxxxxxx | I: xxxxxxxxx xxxxx | P: xxxxxx xxxxxxxxxx | S: xxxxxxxxxx |
| A: XXXX | | A: xxxx xxx xxxxx | S: xxxxxxxxxx xxxxxx | E: xxxxxxxxxx |
| E: xxxxxxxx | | | | |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Procedure/Therapy, Indication. If ongoing, include 'Ongoing' in place of End Date.



# Listing 16.2.4.5: Physical Examination Treatment Group (Page xx of yy)

| S: Subject A: Age/Sex E: Eval | Visit | Date | Body System Assessed | Finding | Abnormal Finding<br>Specification |
|---|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | xxxxxxxxx | xxxxxxxxx | Heart Lungs Skin (Other than Psoriasis) <other, specify=""></other,> | XXXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | ******* |
| | xxxxxxxxxx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxx<br>xxxxxxxxx | |
| | xxxx xx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxx<br>xxxxxxxx | |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | xxxxxxxxx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxxxx xx<br>xxxxxxxxxx xx | xxxxxx |
| | xxxxxxxxx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxxxxx | |
| | xxxx xx | xxxxxxxxx | Heart<br>Lungs<br>Skin (Other than Psoriasis) | xxxxxxxx<br>xxxxxxxx | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, Body System Assessed.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



### Listing 16.2.5.1: Study Visit Compliance Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Visit Date | Study<br>Day¹ | Within Visit<br>Window | Days Out of<br>Window <sup>2</sup> |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | X | xxx | |
| | | | xxxxxxxx | xxxxxxxxx | Х | XXX | |
| | | | xxxx x | xxxxxxxxx | XX | XXX | XXXX |
| XXXXXX | XXXX | XXXXXXX | XXXXXXXX | xxxxxxxxxx to xxxxxxxxx | X | XXX | |
| | | | XXXXXXX | XXXXXXXXX | X | XXX | |
| | | | XXXX X | XXXXXXXXX | XX | XXX | |
| | | | XXXX X | xxxxxxxxx | XX | XXX | |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xx | XXX | |
| | | | xxxxxxxx | xxxxxxxxx | Х | xxx | |
| | | | xxxx x | xxxxxxxxx | XX | xxx | |

Listing sorted by Subject, Visit, Visit Date.

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - baseline date for dates prior to baseline visit. Otherwise, day is calculated as date - baseline date + 1 for dates on or after baseline visit.

 $<sup>^{2}</sup>$  Populated only for post baseline visits that are planned and out of window. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.5.2: Drug Accountability Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Kit Number | Date<br>Dispensed | Date<br>Returned | Tube ID | Dispensed<br>Weight (g) | Returned<br>Weight (g) |
|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxx | xxxxxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | Х | xx.x | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | Х | XX.X | XX.X |
| | | | XXXXX | XXXXXXXXX | xxxxxxxxx | Х | XX.X | XX.X |
| | | | | | | Х | xx.x | XX.X |
| | | | | | | X | xx.x | XX.X |
| | | | | | | Х | xx.x | XX.X |
| | | | XXXXX | XXXXXXXXX | XXXXXXXXX | Х | xx.x | XX.X |
| | | | | | | Х | xx.x | XX.X |
| | | | | | | Х | xx.x | XX.X |
| | | | | | | X | XX.X | XX.X |
| xxxxx | xxxx | xxxxxxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | x | xx.x | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | Х | XX.X | XX.X |
| | | | | | | Х | XX.X | XX.X |
| | | | XXXXX | XXXXXXXXX | XXXXXXXXX | Х | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |
| | | | | | | X | XX.X | XX.X |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Kit Number, Date Dispensed, Date Returned, and Tube ID.



# Listing 16.2.5.3: Study Drug Application Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date/Time of Study<br>Drug Application | Study Drug<br>Applied in Clinic? | Pre-Dose<br>Weight (g) | Post-Dose<br>Weight (g) | Reason<br>Not Done |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxx | xxxxxTxxxx | xxx | XX.X | XX.X | |
| | | | xxxxx | xxxxxTxxxx | XXX | XX.X | XX.X | |
| | | | xxxxx | xxxxxTxxxx | XXX | xx.x | xx.x | |
| xxxxx | xxxx | xxxxxxx | xxxxx | xxxxxTxxxx | XX | | | xxx xxx xxxxx |
| | | | XXXXX | xxxxxTxxxx | XXX | XX.X | XX.X | |
| | | | XXXXX | xxxxxTxxxx | XXX | XX.X | XX.X | |
| xxxxxx | xxxx | xxxxxxx | xxxxx | xxxxxTxxxx | XXX | xx.x | xx.x | |
| | | | XXXXX | xxxxxTxxxx | XXX | XX.X | XX.X | |
| | | | XXXXX | xxxxTxxxx | XXX | XX.X | XX.X | |
| xxxxx | xxxx | xxxxxxxx | xxxxx | xxxxxTxxxx | XX | | | xxx xxx xxxxx |
| | | | xxxxx | xxxxxTxxxx | XXX | XX.X | XX.X | |
| | | | XXXXX | xxxxxTxxxx | XXX | XX.X | XX.X | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Date/Time of Study Drug Application, Visit.



### Listing 16.2.5.4: Dosing Compliance Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | D: Date of First Dose<br>R: Date of Last Dose | Number of<br>Days of<br>Exposure | Calculated¹<br>Number of<br>Doses | Amount of<br>Study Drug<br>Used (g) | Maximum Number<br>of Missed<br>Consecutive Doses | Percent<br>Compliant | Compliant? <sup>2</sup> |
|---|---|---|---|---|---|---|---|
| S: xxxxx<br>A: xxxx<br>E: xxxxxxxx | D: xxxxxxxxxxx<br>R: xxxxxxxxxxx | xx | xx | xxxx | х | xxx | xxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | D: xxxxxxxxxxx<br>R: xxxxxxxxxxx | xx | xx | xxxx | х | xxx | xx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | D: xxxxxxxxxxx<br>R: xxxxxxxxxxxx | xx | xx | xxxx | | xxxx | xxx |

<sup>&</sup>lt;sup>1</sup> The total number of doses was calculated from the date of first dose and the date of last known dose minus the missed doses plus additional dose deviations.

<sup>&</sup>lt;sup>2</sup> A subject was considered compliant with the dosing regimen if the subject applied at least 80% of the expected doses during the study drug application period and did not miss more than 3 consecutive doses.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.5.5: Dosing Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Date of First Dose | Date of Dosing Deviation | Number of Doses Applied |
|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | ************************************** | х<br>х<br>х |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxxx | x<br>x |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx<br>xxxxxxxxx | x<br>x |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, and Date of Dosing Deviation.



Listing 16.2.6.1: Investigator Global Assessment (IGA)

Treatment Group

(Page xx of yy)

| S: Subject<br>A: Age/Sex<br>A: Eval | Visit | Date of<br>Assessment | Whole Body<br>Investigator Global<br>Assessment Score | Does the Subject have Intertriginous Area involvement? | Intertriginous<br>Investigator Global<br>Assessment Score | Evaluator<br>Initials |
|---|---|---|---|---|---|---|
| : xxxxx<br>: xxxx | SCREENING | xxxxxxxxx | x x xxxxxxx | xxx | x x xxxxxxx | xxx |
| • AAAAAAA | BASELINE | xxxxxxxxx | x x xxxxxxxx | xxx | x x xxxxxxxx | xxx |
| | WEEK 2 | XXXXXXXXX | x x xxxxxxx | XXX | x x xxxxxxx | XXX |
| | WEEK 4 | XXXXXXXXX | x x xxxxxxx | XXX | x x xxxxxxx | XXX |
| | WEEK 6 | xxxxxxxxx | x x xxxxxxxx | XXX | x x xxxxxxxx | XXX |
| | WEEK 8 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |
| | WEEK 12 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |
| | WEEK 16 | xxxxxxxxx | x x xxxxxxxx | XX | | xxx |
| 5: xxxxxx<br>4: xxxx | SCREENING | xxxxxxxxx | x x xxxxxxxx | xx | | x-x |
| • | BASELINE | xxxxxxxxx | x x xxxxxxxx | XX | | x-x |
| | WEEK 2 | XXXXXXXXX | x x xxxxxxx | XX | | x-x |
| | WEEK 4 | XXXXXXXXX | x x xxxxxxx | XX | | x-x |
| | WEEK 6 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |
| | WEEK 8 | xxxxxxxxx | x x xxxxxxxx | XX | | xxx |
| | WEEK 12 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |
| | WEEK 16 | xxxxxxxxx | x x xxxxxxxx | XX | | XXX |

Listing sorted by Subject, Visit, and Date of Assessment.

TOOL.AN.10-01.01 Statistical Analysis Plan Template